Official Title: A Phase 3, Randomized, Double-blind, Multicenter, Placebo-controlled,

Parallel-group Trial Evaluating the Efficacy, Safety, and Tolerability of Centanafadine Sustained-release Tablets in Adults With Attention-

deficit/Hyperactivity Disorder

NCT Number: NCT03605680

**Document Date:** SAP Final Version : 27 April 2020

# **Table of Contents**

| Table of Contents |
|---|
| Statistical Analysis Plan; Final: 27 April 2020 |
| STAT-1.1 Adjusted Mean Change from Baseline in AISRS Line Items at Day 42 - MMRM (Efficacy Sample) |
| STAT-1.2 Adjusted Mean Change from Baseline in ASRS Line Items at Day 42 - MMRM (Efficacy Sample)50 |
| STAT-3.1 MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample) |
| STAT-3.2 MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample) |
| STAT-4.1.1 Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample) |
| STAT-4.1.2 Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample) |
| STAT-4.2 Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, LOCF (Efficacy Sample) |
| STAT-4.3 Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, OC (Efficacy Sample) |
| STAT-4.4 Proc GLM Output for Treatment by Center Interaction at Day 42 in AISRS Total Score, LOCF (Efficacy Sample) |
| STAT-4.5.1 Summary of Mean Change at Day 42 from Baseline in AISRS Total Score By Center - LOCF (Efficacy Sample) |
| STAT-4.5.2 Differences in Unadjusted Mean Changes of AISRS Total Score at Day 42<br>Among Treatment Groups By Center - LOCF (Efficacy Sample) |
| STAT-4.6 Unadjusted Mean Change from Baseline to Double Blind Treatment Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample) |
| STAT-4.7 Unadjusted Mean Change from Baseline to Double Blind Treatment Period by Study Day in AISRS Total Score, OC (Efficacy Sample) |
| STAT-4.8 Non-Parametric Stratified by Center Analysis of Mean Change from Baseline to Double Blind Treatment Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample) |
| STAT-4.9 Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)217 |
| STAT-4.10 Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample) |

| (Efficacy Sample) | 252 |
|---|---|
| STAT-5.2 Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, LOCF (Efficacy Sample) | 266 |
| STAT-5.3 Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, OC (Efficacy Sample) | .272 |
| STAT-6.1.1 Shapiro-Wilk Test for Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample) | 278 |
| STAT-6.1.2 Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample) | 279 |

# Otsuka Pharmaceutical Development & Commercialization, Inc.

**Investigational Medicinal Product** 

Centanafadine (EB-1020)

A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Evaluation the Efficacy, Safety and Tolerability of Centanafadine Sustained-release in Adults with Attention-deficit/Hyperactivity Disorder

Protocol No. 405-201-00013 IND No. 119,361

# Statistical Analysis Plan

**Version: Final** 

Date: April 27, 2020

CONFIDENTIAL - PROPRIETARY INFORMATION

Confidential
May not be used, divulged, published or otherwise disclosed
without the consent of Otsuka Pharmaceutical Development & Commercialization, Inc.

# **Table of Contents**

| Lab | le of Contents | 4 |
|---|---|---|
| 1 | Introduction | 5 |
| 2 | Study Objectives | 5 |
| 3 | Study Design | 5 |
| 4 | Sample Size and Power Justification | <mark>7</mark> |
| 5 | Data Sets for Analysis and Missing Data | <mark>7</mark> |
| 5.1 | Data Sets for Analysis | |
| 5.2 | Handling of Missing Data | 8 |
| 6 | Study Conduct | 9 |
| 6.1 | Subject Disposition, Completion Rate and Reasons for Discontinuation | 9 |
| 6.2 | Treatment Compliance | 9 |
| 6.3 | Protocol Deviation | 10 |
| 7 | Baseline Characteristics | 10 |
| 7.1 | Baseline Definition | 10 |
| 7.2 | Demographic Characteristics | 10 |
| 7.3 | Medical and Psychiatric History | 10 |
| 7.4 | Neuropsychiatric Diagnosis | 11 |
| 7.5 | Baseline Psychiatric Evaluation | 11 |
| 8 | Efficacy Analysis | 11 |
| 8.1 | Primary Efficacy Endpoint | 11 |
| 8.1.1 | Primary Efficacy Analysis | 11 |
| 8.1.2 | Technical Computation Details for Primary Efficacy Analysis | 13 |
| 8.1.3 | Sensitivity Analyses | 14 |
| 8.1.3. | 1 Sensitivity Analyses for Missing at Random (MAR) Assumption | 14 |
| 8.1.3. | 2 Per Protocol Analyses | 15 |
| 8.1.3. | 3 Sensitivity Analyses for Violation of Normality Assumption | 15 |
| 8.1.4 | Subgroup Analyses | 16 |
| 8.2 | Key Secondary Efficacy Endpoint | 16 |
| 8.3 | Other Efficacy Endpoints | |
| 8.4 | Exploratory Efficacy Endpoints | 18 |

| 8.5 | Exploratory Analysis | 18 |
|---|---|---|
| 9 | Safety Analysis | 19 |
| 9.1 | Adverse Events | 19 |
| 9.1.1 | Adverse Events in the Double-Blind Treatment Period | 20 |
| 9.1.2 | Adverse Events in the Single-blind Placebo Run-in Period | 21 |
| 9.2 | Clinical Laboratory Tests | 21 |
| 9.2.1 | Clinical Laboratory Tests in Double-Blind Treatment Period | 21 |
| 9.2.2 | Drug Induced Liver Injury (DILI) | 21 |
| 9.2.3 | Clinical Laboratory Tests in the Single-blind Placebo Run-in Period | 22 |
| 9.3 | Vital Signs | 22 |
| 9.3.1 | Vital Signs in the Double-Blind Treatment Period | 22 |
| 9.3.2 | Vital Signs in the Single-blind Placebo Run-in Period | 22 |
| 9.4 | Electrocardiogram (ECG) Data | 22 |
| 9.4.1 | ECG Data in the Double-Blind Treatment Period | 23 |
| 9.4.2 | ECG Data in the Single-blind Placebo Run-in Period | 23 |
| 9.5 | Physical Examinations | 23 |
| 9.5.1 | Body Weight, Waist Circumference and Body Mass Index (BMI) | 23 |
| 9.6 | Suicidality Data | 24 |
| 9.7 | SMWQ | 24 |
| 9.8 | Medication Handling Irregularities (MHIs) and Events Subject to Addition Monitoring (ESAMs) | |
| 9.9 | Concomitant Medications | 25 |
| 9.10 | Extent of Exposure | 25 |
| 10 | Conventions | 25 |
| 10.1 | Study Visit Windows | 25 |
| 10.2 | Pooling of small centers | 26 |
| 10.3 | Scales: Rules for Scoring and Handling of Missing Data | 27 |
| 10.3.1 | Adult ADHD Investigator Symptom Rating Scale (AISRS) | 27 |
| 10.3.2 | Clinical Global Impression Severity of Illness Scale – Modified for Attention-Deficit Hyperactivity Disorder | 27 |
| 10.3.3 | Clinical Global Impression Change from Baseline | 28 |
| 10.3.4 | Attention-Deficit Hyperactivity Disorder Impact Module – Adult (AIM- | A) 28 |
| 10.3.5 | Adult ADHD Self Report Scale (ASRS) | 28 |

| SA |
|----|

| 10.3 | .6 Study Medication Withdrawal Questionnaire (SMWQ) | 28 |
|------|-----------------------------------------------------|----|
| 10.3 | .7 Columbia-Suicide Severity Rating Scale (C-SSRS) | 29 |
| 11 | References | 30 |
| 12 | Potential Clinical Relevance Criteria from Protocol | 31 |
| 13 | Proposed List of Summary Tables | 34 |

#### 1 Introduction

This statistical analysis plan (SAP) documents the statistical methodology and data analysis algorithms and conventions to be applied for statistical analysis and reporting of efficacy and safety data of study 405-201-00013. All amendments to the protocol are taken into consideration in developing this SAP.

# 2 Study Objectives

Primary: To confirm the efficacy of centanafadine SR tablets administered BID (200 mg or 400 mg TDDs) compared to placebo in the treatment of adults with ADHD

Secondary: To confirm the safety and tolerability of centanafadine SR tablets administered BID (200 mg or 400 mg TDDs) compared to placebo in the treatment of adults with ADHD

# 3 Study Design

This trial is a phase 3, randomized, double-blind, multicenter, placebo-controlled, parallel-group trial to confirm the efficacy, safety, and tolerability of centanafadine SR (200 mg TDD) or 400 mg TDD) compared to placebo for the treatment of adults with ADHD. The trial population will include male and female subjects 18 to 55 years of age (inclusive) with a current diagnosis of ADHD as confirmed by the Adult ADHD Clinical Diagnostic Scale (ACDS) Version 1.2 at screening.

The trial will have 4 periods: (1) screening and washout; (2) 1 week single-blind placebo runin; (3) 6-week double blind treatment; and (4) 7-day follow-up period (follow-up telephone calls at 1, 3, and 5 days after the last dose of IMP, and in-clinic visits 2 and 7 days after the last dose of IMP) for subjects who complete the trial, and decide to enroll in Trial 405-201-00015. For subjects who terminate early, decide to not enroll in Trial 405-201-00015, or who are not eligible to enroll in Trial 405-201-00015, they will be required to participate in the 7-day follow-up period as well as participate in an additional follow-up telephone call 10 days after the last dose of IMP. Subjects randomized to receive a TDD of 200 mg centanafadine SR will start at their target dose at the start of the double-blind treatment period. Subjects randomized to receive a TDD of 400 mg centanafadine SR will start the double-blind treatment period at the TDD of 200 mg centanafadine SR for 7 days, before they are escalated to their target TDD of 400 mg for a total of approximately 42 days of treatment. Subjects will be required to visit the site up to 12 times over the trial. See Figure 3-1 for a schematic of the trial design.

Subjects who complete both the 6-week double-blind treatment period and the 7-day safety follow-up period (follow-up telephone calls at 1, 3, and 5 days after the last dose of IMP, and in-clinic visits 2 and 7 days after the last dose of IMP), and refrain from using prohibited

medications after the IMP is stopped may be eligible to enroll into Trial 405-201-00015, which is a 12-month, observational, open-label trial to evaluate the long-term safety and tolerability of subjects with ADHD who previously participated in Trials 405-201-00013 or 405-201-00014. Subjects who terminate early, decide to not enroll in Trial 405-201-00015, or who are not eligible to enroll in Trial 405-201-00015, will be required to participate in the 7-day follow-up period as well as participate in an additional follow-up telephone call 10 days after the last dose of IMP. For subjects who early terminate or decline participation in the open-label trial, they will be instructed to refrain from utilizing prohibited concomitant medications, including ADHD treatments, until after the follow-up telephone call 10 days after the last dose of IMP.



Figure 3-1 Trial Design Schematic

ASRS = Adult ADHD Self Report Scale; CTN SR = centanafadine sustained release; ET = early termination; P = placebo administration; R = randomization.

During the trial, administration of the investigational medicinal product (IMP) will be double-blinded. In other words, neither the investigator nor the subject will have knowledge of the treatment assignment (e.g., centanafadine SR 200 mg, 400 mg, or placebo). Treatment assignments will be based on a computer-generated randomization code provided by the Otsuka Pharmaceutical Development & Commercialization, Inc (OPDC) Biometrics Department. Sponsor personnel, including those involved in monitoring, data management, and data analysis, will not have access to the treatment code during the trial. The bioanalytical

<sup>&</sup>lt;sup>a</sup>All subjects will be required to participate in the 7-day follow-up period (follow-up telephone calls at 1, 3, and 5 days after the last dose of IMP, and in-clinic follow-up visits at 2 and 7 days after the last dose of IMP). Subjects who terminate early, decide to not enroll in Trial 405-201-00015, or who are not eligible to enroll in Trial 405-201-00015, will be required to participate in an additional follow-up telephone call 10 days after the last dose of IMP.

laboratory will also be sent the randomization code. The randomization will be stratified by trial site and designed to allocate subjects in a 1:1:1 ratio to centanafadine SR 200 mg/day or 400 mg/day or placebo.

# 4 Sample Size and Power Justification

The primary efficacy endpoint is the change from baseline at Day 42 in Adult ADHD Investigator Symptom Rating Scale (AISRS) total score. The trial will compare the placebo arm to the centanafadine dose arms, randomized at a ratio of 1:1:1, with an overall alpha of 0.05 for the primary endpoint.

Based on the results from Phase 2 centanafadine trials, it is reasonable to expect a treatment effect of 5 points with a standard deviation (SD) of 12.5 in the mean change from baseline to Day 42 on AISRS total score. The planned sample size of 405 evaluable subjects (135 in each treatment arm) will yield at least 90% power to detect the treatment effects at a 2-tailed significance level of 0.05.

A sufficient number of subjects will be enrolled and randomized to achieve approximately 405 evaluable subjects in the Double-blind Treatment Phase (i.e., subjects with an AISRS total score at baseline and at least 1 subsequent AISRS total score in the Double-blind Treatment Phase). After allowance of 10% non-evaluable subjects in the Double-blind Treatment Phase, the total number of subjects to be randomized is 450 (150 in each treatment arm). In order to ensure 405 evaluable subjects, the number of non-evaluable subjects will be monitored in a blinded manner on an ongoing basis During the trial. The power and sample size were obtained using the PASS 14 (2015) statistical computing software.

# 5 Data Sets for Analysis and Missing Data

#### 5.1 Data Sets for Analysis

The following analysis samples are defined for this trial:

**Enrolled Sample**: comprises all subjects who signed an informed consent form (ICF) for the trial and enrolled into the single-blind placebo run-in period.

**Randomized Sample**: comprises all subjects who were randomized in the double-blind treatment period. Subjects are considered randomized when they are assigned a treatment group by eSource at the end of single-blind placebo run-in period. A subject receiving IMP outside of the eSource will not be considered randomized, but safety will be reported.

**Safety Sample**: comprises those randomized subjects in the double-blind treatment period who received at least one dose of double-blind IMP as indicated on the dosing record. Subjects will only be excluded from this population if there is documented evidence (i.e., drug

dispensed = drug returned or no IMP dispensed) that the subject did not take IMP. If a subject is dispensed IMP and is lost to follow up, he/she will be considered exposed.

**Efficacy Sample**: the Full Analysis Set (FAS) comprises all subjects in the Safety Sample who have a baseline value and at least one valid post-randomization efficacy evaluation for AISRS total score in the double-blind treatment period.

**Per Protocol (PP) Sample:** comprises those subjects in the Efficacy Sample who complete at least the first 2 weeks of double-blind medication ((last day of IMP - first day of IMP + 1)  $\geq$  14 days) and have at least one post baseline AISRS measurement on or after Day 14 visit during the double-blind treatment period without major protocol violations deemed to compromise the assessment of efficacy. These major protocol violations will be any of the followings:

- 1. Subjects who were not at least 80% or were more than 120% compliant with double-blind IMP or missed 7 or more consecutive days of dosing immediately prior to the Day 42/ET AISRS measurement date during the double-blind treatment period based on subject-reported (eCRF) compliance data
- Subjects who reported concomitant medication use that will impact the primary efficacy endpoint
- 3. Subjects who had major protocol deviation as represented on the protocol deviation eCRF page that will impact the primary efficacy endpoint
- 4. Subjects who took the wrong study treatment

The core dataset for all efficacy analyses is the FAS, which is created based on the intent-to-treat (ITT) principle. However, as will be described below, in order to handle missing data and restrictions imposed by different types of analyses (e.g., change from baseline analysis), other datasets derived from the FAS dataset will be used for the efficacy analyses.

#### 5.2 Handling of Missing Data

The mixed-effect model repeated measure (MMRM) assumes data are missing at random (MAR), which is a reasonable assumption in longitudinal clinical trials in MDD<sup>1</sup>. However, the possibility of "missing not at random" (MNAR) data can never be ruled out. As sensitivity analyses, selection model<sup>2</sup>, pattern-mixture model<sup>3,4,5,6</sup>, and/or shared parameter model<sup>7</sup> will be used to explore data missing mechanisms of MNAR and investigate the response profile of dropout patients by last dropout reason under MNAR mechanism for the following 3 scenarios: 1) Dropout reasons due to either AE or LOE as MNAR, 2) Dropout reasons due to either AE or LOE or subject withdrew consent as MNAR, 3) All dropouts as MNAR using

both 1) Delta adjustment imputation method which is to departure from MAR assumption by progressively increasing the delta until conclusion from the primary analysis is overturned, and 2) Placebo based imputation methods in which missing data for both placebo and drug group are imputed based on the imputation model derived from placebo data. If drug improved outcomes prior to dropout, this benefit is carried into subsequent imputed values, but will diminish over time in accordance with the correlation structure. Details are provided in Section 8.1.3 Sensitivity Analysis.

The observed-cases (OC) data set will consist of actual observations recorded at each visit during the double-blind treatment period and no missing data will be imputed. MMRM, Wu-Bailey, and pattern-mixture model will be performed on the OC dataset.

The last-observation-carried-forward (LOCF) data set will include data recorded at a scheduled double-blind treatment period visit or, if no observation is recorded at that visit, data carried forward from the previous scheduled double-blind treatment period visit.

Baseline data (e.g., the last visit of the single-blind placebo run-in period) will not be carried forward to impute missing values for the LOCF data set. The analysis of covariance (ANCOVA) analysis will be performed for the change from baseline to the end of the double-blind treatment period (Day 42, LOCF) in AISRS total score as sensitivity analysis. The ANCOVA\_LOCF model includes treatment and study center as main effects, and baseline value as a covariate.

ANCOVA analysis with OC data will also be conducted on change from baseline for AISRS total score, as well as all continuous change from baseline efficacy endpoints.

For Clinical Global Impression (CGI) Change from Baseline and categorical response/remission variables, OC analyses will be performed in addition to LOCF analyses. Study center will not be included in the models for OC analyses.

# 6 Study Conduct

# 6.1 Subject Disposition, Completion Rate and Reasons for Discontinuation

Subject disposition will be summarized for the Randomized Sample by treatment group, and by center.

Subject completion rate and reasons for discontinuation will be summarized for the Randomized Sample by treatment group for the double-blind treatment period.

#### **6.2 Treatment Compliance**

For each subject, compliance in taking IMP is calculated by dividing the number of tablets taken by the total number of tablets the patients were scheduled to take during the double-blind

treatment period. Compliance is calculated on double-blind IMP for the double-blind treatment period. For lost-to-follow up patients, the last IMP end date record will be used as the treatment end date.

Summary of Treatment compliance will be provided based on both eCRF data and AiCure captured data, respectively.

#### 6.3 Protocol Deviation

Protocol deviations are summarized by center and type of deviation for randomized subjects by treatment group. Listing of protocol deviation will list the treatment phases during which the deviations occurred. In addition, protocol deviations affected by the COVID-19 will be summarized. Listing of subjects with protocol deviations affected by the COVID-19 will also be provided.

#### 7 Baseline Characteristics

#### 7.1 Baseline Definition

Baseline for the single-blind placebo run-in period refers to last available measurement prior to the start of administration of placebo in the single-blind placebo run-in period.

For analyses of the double-blind treatment period data, the baseline is defined as the last available measurement prior to the first dose of double-blind Investigational Medicinal Product (IMP) in the double-blind treatment period.

# 7.2 Demographic Characteristics

For the Randomized Sample, demographic characteristics will be summarized by treatment group. Age, race, ethnicity, height, weight, waist circumference, and body mass index (BMI) will be tabulated by gender and overall using the baseline assessments for the single-blind placebo run-in period.

Mean, range and standard deviation will be used to describe continuous variables such as age. Frequency distributions will be tabulated for categorical variables such as race.

# 7.3 Medical and Psychiatric History

A summary of medical and psychiatric history will be presented for the Randomized Sample by treatment group and overall.

A summary of the Adult ADHD Clinical Diagnostic Scale (ACDS) at screening will also be presented for the Randomized Sample (by treatment group and overall). The number and

percentage of patients with each response to items A23-A41 from Section A (Childhood ADHD Symptoms Summary), B22-B39 from Section B (Adult ADHD Symptoms Summary), and C1-C5 will be presented.

#### 7.4 Neuropsychiatric Diagnosis

A summary of MINI International Neuropsychiatric Interview (M.I.N.I.) will be presented for the Randomized Sample by treatment group and overall. Summarized will be the number and percentage of patients who meet each diagnosis criteria, and number and percentage of patients with each primary diagnosis.

#### 7.5 Baseline Psychiatric Evaluation

For the Randomized Sample, baseline for the single-blind placebo run-in period and baseline for the double-blind treatment period psychiatric scale evaluation will be summarized by treatment group and overall. The mean, median, range and standard deviation will be used to summarize the assessments of: AISRS total score, ASRS and CGI - Severity of Illness Score (CGI-S).

# 8 Efficacy Analysis

All efficacy analyses pertaining to the double-blind treatment period will be performed on the Efficacy Sample, and patients will be included in the treatment group as randomized.

For analysis of the double-blind treatment period data, the baseline for the double-blind treatment period defined in Section 7.1 will be used. Statistical comparisons are based on 2-sided, 0.05 significance levels.

# 8.1 Primary Efficacy Endpoint

The primary efficacy endpoint is the change from the baseline of the double-blind treatment period to Day 42 in AISRS total score.

# 8.1.1 Primary Efficacy Analysis

The objective of the primary efficacy analysis is to compare the efficacy between centanafadine (SR 200 mg TDD or SR 400 mg TDD) and placebo.

The primary estimand defining the treatment effect of interest in the trial uses the hypothetical strategy specified in the draft ICH E9 (R1) Addendum. The objective of the primary analysis is to evaluate the efficacy of centanafadine SR 400mg TDD in adult subjects with ADHD

versus placebo. The estimand, or target of estimation, following the hypothetical strategy is the pharmacological effect seen, had no withdrawals occurred. This hypothetical estimand is justifiable in this case, since the focus is on the pharmacological effect of the drug additional to non-specific effects. Subjects who withdraw from a symptomatic IMP treatment either could have lost their treatment effect, had the subjects not taken any other symptomatic medication after withdrawal, or could have their treatment effect been masked, had the subjects taken other symptomatic medication after withdrawal. This means that any observations taken after subjects stop IMP will most likely not contribute relevant information about the pharmacological effect of the drug. Due to this strategy, the last collected efficacy assessment after premature trial discontinuation will be done only once at the ET Visit. Every effort will be made to complete all of the ET evaluations prior to administering any additional medications for the treatment of ADHD or other prohibited medications. In the case of terminal or lost to follow-up events, no ET evaluations would be expected, and only scheduled assessments performed before such an event has occurred.

The primary estimand for this trial is defined by the following components:

- Target Population: Efficacy Sample
- Endpoint: Change from baseline to Day 42 in the AISRS total score
- Intercurrent Events: Premature treatment discontinuation
- Measure of Intervention Effect: Difference in endpoint means between centanafadine (SR 200 mg TDD or SR 400 mg TDD) and placebo.

In this hypothetical strategy, the event of withdrawing IMP is considered missing at random (MAR), and the primary endpoint of the trial could be considered as a combination of the responses of on-treatment completers at Day 42 and the imputation of the endpoint to Day 42 following the trend in each treatment group using the MMRM method for subjects who withdraw IMP during the trial. All data collected during the trial treatment period will be used for statistical analysis. For the primary efficacy analysis, the treatment effect will be estimated using the MMRM method described below. Under the MAR assumption, MMRM provides an unbiased estimate of treatment effect for the treatment period. Analyses with missing values imputed by multiple imputation under MNAR and other methods will be performed as sensitivity analyses. The primary analysis will be performed on Efficacy Sample which includes all randomized subjects who took at least 1 dose of IMP in the double-blind treatment period and who have both a baseline for the double-blind treatment period. The primary efficacy analysis will be performed by fitting a MMRM analysis with an unstructured (UN) variance covariance structure in which the change from baseline for the double-blind

treatment period in AISRS total score at the scheduled double-blind treatment period visits will be the dependent variable based on the OC data set. The model will include fixed class effect terms for treatment, study center, visit day, and an interaction term of treatment by visit day. The model will also include the interaction term of baseline values for the double-blind treatment period of AISRS Total score by visit day as covariates. The primary comparison between centanafadine (400 mg TDD group or 200 mg TDD group) and placebo at Day 42 in the double-blind treatment period will be estimated as the difference between Least Squares (LS) means utilizing the computing software SAS procedure PROC MIXED.

In case there is a convergence problem with MMRM model with the unstructured (UN) variance covariance matrix, the following structures other than unstructured will be used in order of 1) heterogeneous toeplitz (TOEPH), 2) heterogeneous autoregressive of order 1 (ARH1), and 3) heterogeneous compound symmetry (CSH) and the first (co)variance structure converging to the best fit will be used as the primary analysis. If a structured covariance has to be used, the empirical "sandwich" estimator of the standard error of the fixed effects parameters will be used in order to deal with possible model misspecification of the covariance matrix.

Small centers will be defined as centers that do not have at least one evaluable subject (evaluable with regard to the primary efficacy variable) in each treatment arm in the double-blind treatment period. All small centers will be pooled to form "pseudo centers" for the purpose of analysis according to the following algorithm. Small centers will be ordered from the largest to the smallest based on the number of evaluable subjects (i.e., subjects who have baseline and at least one post-baseline value for the primary endpoint in the double-blind treatment period). The process will start by pooling the largest of the small centers with the smallest of the small centers until a non-small center is formed. This process will be repeated using the centers left out of the previous pass. In case of ties in center size, the center with the smallest center code will be selected. If any centers are left out at the end of this process, they will be pooled with the smallest pseudo centers, or if no pseudo centers exist, they will be pooled with the smallest non-small center.

# 8.1.2 Technical Computation Details for Primary Efficacy Analysis

The SAS code for the PROC MIXED procedure to carry out the above MMRM analysis with an unstructured variance covariance structure is illustrated as follows:

```
proc mixed;
  class treatment center visit subjid;
  model change=treatment center visit treatment*visit baseline*visit / s cl
ddfm=kenwardroger;
  repeated visit /type=un subject=subjid r rcorr;
```

lsmeans treatment\*visit / pdiff cl alpha=0.05 slice=visit; run;

where baseline is the last AISRS Total score prior to the first dose of double-blind IMP in the double-blind treatment period.

#### 8.1.3 Sensitivity Analyses

### 8.1.3.1 Sensitivity Analyses for Missing at Random (MAR) Assumption

Traditionally the dropout mechanisms are divided into three types (Little, 1995): (1) Missing Completely at Random (MCAR), in which the probability of dropout doesn't depend on the observed data and the missing data; (2) Missing at Random (MAR), in which the probability of dropout depends on the observed data, and (3) Missing Not at Random (MNAR), where the probability of dropout depends on the missing data and possibly the observed data.

Most of MNAR methods (Diggle P, Kenward MG, 1994) have treated all observations with dropout as if they fall within the same dropout type. In practice, we would find that different dropout reasons may be related to the outcomes in different ways, for example, detailed dropout reasons for this study are: adverse events (AE), lack of efficacy (LOE), lost to follow-up, protocol deviation, sponsor discontinued study, subject met (protocol specified) withdrawal criteria, subject was withdrawn from participation by the investigator, and subject withdrew consent to participate. Dropout due to an AE and LOE may lead to MNAR dropout. Subject withdrew consent may also lead to MNAR dropout. However, it is debatable whether a dropout caused by subjects withdrew consent is MAR or MNAR. Except AE, LOE, and subject withdrew consent, all the other dropout reasons may be assumed as either MCAR or MAR dropout. Dropout due to COVID-19 will also be assumed as MAR.

As sensitivity analyses for missing at random (MAR) assumption, analyses for missing not at random (MNAR) will be carried out. Pattern Mixture Models (PMM) based on Multiple Imputation (MI) with mixed missing data mechanisms will be used to investigate the response profile of dropout patients by last dropout reason under MNAR mechanism for the following three scenarios:

- 1) Dropout reasons due to either AE or LOE as MNAR
- 2) Dropout reasons due to either AE or LOE or subject withdrew consent as MNAR
- 3) All dropouts as MNAR

#### **Delta Adjustment Imputation Methods**

This MNAR sensitivity analysis is to departure from MAR assumption by progressively increasing the delta until conclusion from the primary analysis is overturned. The delta is 0%, 10%, 20%, 30%, ..., 100% of the expected treatment difference of 5 points and/or the observed

treatment difference between centanafadine and Placebo from the primary analysis of MMRM model until conclusion of the primary analysis is overturned. When delta=0 it is MAR. When delta > 0 it is MNAR.

- 1) Using Monte Carlo Markov Chain (MCMC) methodology from PROC MI to impute the intermittent missing data to a monotone missing pattern;
- 2) Using a standard MAR-based multiple imputation approach from PROC MI to impute the monotone missingness data
- 3) For patients in the treated group and with a dropout reason of AE or LOE or subject withdrew consent, a delta will be added for all the values after the dropout time.
- 4) Using MMRM model in the primary analysis to analyze the completed data using PROC MIXED on the multiple imputed data
- 5) Obtaining the overall results using PROC MIANALYZE.

#### **Placebo Based Imputation Methods**

Similar to "Standard" multiple imputations, except parameters for imputation model obtained from only the placebo (control) group. Missing data for both placebo and drug group are imputed based on the imputation model derived from placebo data. If drug improved outcomes prior to dropout, this benefit is carried into subsequent imputed values, but will diminish over time in accordance with the correlation structure.

In addition, model based MNAR methods such as the shared parameter model (Wu and Baily, 1989) and random coefficient pattern mixture model (Hedeker D, Gibbons RD, 1997) will be also performed.

#### **LOCF and OC Analyses**

Change from baseline of the double-blind treatment period for the AISRS total score will be evaluated using ANCOVA with baseline of the double-blind treatment period value as covariate and treatment and, in LOCF analyses, study center as main effects. For the OC analyses, study center will not be included in the model.

# 8.1.3.2 Per Protocol Analyses

Per Protocol analysis will be performed using the Per Protocol Sample.

# 8.1.3.3 Sensitivity Analyses for Violation of Normality Assumption

The primary endpoint MMRM analysis is a maximum likelihood method that relies on normality assumption. Residual analyses will be carried out to examine model assumption.

In the case of gross violations of the normality assumptions, nonparametric van Elteren test<sup>8</sup> (van Elteren, 1960) will be performed to compare treatment effect at Week 14 on both LOCF

dataset and Multiple Imputation (MI) data. The van Elteren test is a generalized CMH procedure useful for stratified continuous data in non-normal setting. It belongs to a general family of Mantel-Haenszel mean score tests. The test is performed via SAS procedure PROC FREQ, by including CMH2 and SCORES=MODRIDIT options in the TABLE statement. The stratification factor is trial center.

In addition, other methods that are robust to distributional assumption will also be performed to provide different views on the primary efficacy result, these include generalized estimating equations (GEE), weighted GEE (WGEE), and MI-robust regression<sup>9</sup>.

For MI-van Elteren test and MI-robust regression, imputation datasets will be generated with SAS MI procedure, each dataset will be analyzed, then an overall estimate is derived with SAS MIANALYZE procedure.

# 8.1.4 Subgroup Analyses

Subgroup analyses of change from baseline of the double-blind treatment period in AISRS total score to every scheduled visit in the double-blind treatment period will be performed by the following factors:

- Sex (Based on the biological status)
- Race (White and All Other Races)

All subgroup analyses will be conducted using the same MMRM analysis as for the primary efficacy analysis except that the fixed class effect term for trial center will not be included in the model.

Interaction effects of treatment-by-subgroup will be assessed at Day 42 for the subgroups identified in the previous paragraph. MMRM analyses will be performed by adding addition of terms for subgroup-by-day and treatment-by-subgroup-by-day. These treatment-by-subgroup interaction analyses will be presented in statistical documentation.

## 8.2 Key Secondary Efficacy Endpoint

The key secondary efficacy endpoint is the change from baseline of the double-blind treatment period to Day 42 using the CGI-S. This key secondary efficacy endpoint will be analyzed by fitting the same MMRM model described in the primary analysis.

To control the overall experiment-wise type I error at 0.05 level, A fixed sequence testing approach will be applied. The statistical test will be performed in the following order:

1) Change from baseline to Day 42 in the double-blind treatment period in AISRS total score between centanafadine 400 mg TDD and placebo;

- 2) Change from baseline to Day 42 in the double-blind treatment period in AISRS total score between centanafadine 200 mg TDD and placebo;
- 3) Change from baseline to Day 42 in CGI-S score between centanafadine 400 mg TDD and placebo;
- 4) Change from baseline to Day 42 in CGI-S score between centanafadine 200 mg TDD and placebo.

The testing procedure will stop at the first comparison where the p-value is  $\geq 0.05$ . None of the subsequent comparisons will be performed.

#### 8.3 Other Efficacy Endpoints

Other efficacy analyses are listed below. All other efficacy variables will be evaluated at a nominal 0.05 level (2-sided) without adjusting for multiplicity.

- 1) Change from baseline in AISRS total score for every scheduled visit during the doubleblind treatment period other than the Day 42 visit;
- 2) Change from baseline for the Inattentive subscale and Hyperactive-Impulsive subscale of the AISRS for scheduled visits during the double-blind treatment period, separately at every visit
- 3) Change from baseline in CGI-S for every scheduled visit during the double-blind treatment period other than the Day 42 visit
- 4) CGI Change from Baseline will be collected at each scheduled visit
- 5) Percentage of responders at each post-baseline visit during the double-blind treatment period, where a responder is defined as a subject with a CGI Change from Baseline score of 1 or 2 OR a ≥ 30% improvement in ADHD symptoms compared with baseline as measured by the AISRS total score
- 6) Response rate at each post-baseline visit during the double-blind treatment period, where response is defined as
  - a) a CGI Change from Baseline score of 1 or 2 OR a  $\geq$  20% improvement in ADHD symptoms compared with baseline as measured by the AISRS total score.
  - b) a CGI Change from Baseline score of 1 or 2 OR a  $\geq$  40% improvement in ADHD symptoms compared with baseline as measured by the AISRS total score.
- 7) Remission rate for every scheduled visit during the double-blind treatment period, where remission is defined as AISRS total score  $\leq 18$ .

Variable (1) through variable (3) will be evaluated using the same MMRM model described in the primary analysis. Variable (4) will be evaluated by the Cochran Mantel Haenszel (CMH) Row Mean Score Differ Test controlling, in LOCF analysis, for trial center. Variable (5) through variable (7) will be evaluated by the CMH General Association Test controlling, in LOCF analysis, for study center. An OC analysis will also be conducted for variables (4)

through (7) but will not control for trial center. Separate summary and statistical test for response rate based only on the AISRS improvement and only on the CGI Change from Baseline score will be presented for (5) and (6).

#### 8.4 Exploratory Efficacy Endpoints

The exploratory efficacy endpoints are listed below. The exploratory efficacy endpoints, when applicable, will be evaluated at a nominal 0.05 level (2-sided) without adjusting for multiplicity.

- Change from baseline for Question 1 (Global Quality of Life) and Questions 9Aa –
   9Ai and 9Ba 9Bi (Impact of Symptoms) of AIM-A at scheduled visits during the double-blind treatment period, separately at every visit
- 2) Proportion of subjects in each response for the following questions of AIM-A at scheduled visits during the double-blind treatment period, separately at every visit
  - a. Questions 2-4 (Global Quality of Life)
  - b. Questions 5a-5j (Living with ADHD)
  - c. Questions 6a-6k (General Well-Being)
  - d. Questions 7a-7j (Work, Home and School Performance and Daily Functioning)
  - e. Questions 8a-8h (Relationships and Communication)
  - f. Economic impact (5 items)
  - g. Questions 17-23 (Demographics/Medication Status)
- 3) Change from baseline in the total score of (18 item) ADHD Symptoms score of the ASRS and subscale scores for ASRS at scheduled visits during the double-blind treatment period, separately at every visit

Variables (1) and (3) will be evaluated using the same MMRM model described in the primary analysis. Variable (2) will be summarized by descriptive statistics and no statistical comparisons between centanafadine and placebo will be performed.

#### 8.5 Exploratory Analysis

Exploratory efficacy analyses will be presented in Statistical Documentation.

Treatment-by-center interaction will be assessed at Day 42 by including the treatment-by-center-by-visit interaction in the model. Results for study centers will be displayed from largest center to smallest center.

Line Item score will be performed for AISRS and ASRS on Change from baseline of the double-blind treatment period to Day 42 using the MMRM model for AISRS and ASRS, where Cohen's D Effect Size<sup>10</sup> is the difference between the two means divided by their standard deviation [as defined by Cohen's D and reviewed on pages 4-6 from the Sage book "Effect Size for ANOVA Designs" (Vol 129) by Cortina and Nouri]. For MMRM (using SAS PROC MIXED), or ANCOVA (Using SAS PROC GLM), LSMean difference of treatment effects for the between centanafadine and placebo groups, and the standard error of the difference (Stderr) will be obtained with an Estimate statement. Let n<sub>1</sub> and n<sub>2</sub> denote the respective sample sizes of the two groups to compare, Effect Size =  $d = (LSMean_1 - LSMean_1)$ 

LSMean<sub>2</sub>) / 
$$\sigma$$
, where  $\sigma = \frac{\text{Stderr}}{\sqrt{\frac{1}{n_1} + \frac{1}{n_2}}}$ .

#### 9 Safety Analysis

Standard safety variables to be analyzed include AEs, clinical laboratory tests, vital signs, electrocardiograms (ECGs), body weight, waist circumference, and BMI. In addition, data from the following safety scales will be evaluated: C-SSRS and Study Medication Withdrawal Questionnaire (SMWQ).

Analyses of the double-blind treatment period safety data will be performed on the Safety Sample unless indicated otherwise.

The Safety Sample will also be analyzed for the single-blind placebo lead-in period safety data, as applicable, by treatment groups the subjects eventually being assigned in the doubleblind treatment period.

#### 9.1 **Adverse Events**

All adverse events (AEs) will be coded by system organ class (SOC) and Medical Dictionary for Regulatory Activities (MedDRA) Preferred Term (PT). The incidence of the following events will be summarized:

- Treatment-emergent AEs (TEAEs) a)
- b) TEAEs by severity
- TEAEs potentially causally related to the IMP c)
- d) TEAEs with an outcome of death
- e) Serious TEAEs
- f) TEAEs leading to discontinuation of the IMP

- g) Treatment-emergent Adverse Events of Special Interest (AESI)
- h) Abuse-related TEAEs and TEAEs involving MHIs (Medication handling irregularities)

AEs will be classified by Primary SOC and PT according to the MedDRA. AEs that are gender-specific, e.g., ovarian cancer, will have their incidence rates evaluated for the specific gender.

Incidence of TEAEs will be summarized by double-blind treatment group for the double-blind treatment period. Incidence of TEAEs by SOC and MedDRA PT will be summarized for sex and race.

#### Adverse Events of Special Interest

Newly acquired skin eruptions that are non-traumatic will be considered AESIs. These may include but are not limited to eruptions such as skin rashes, skin irritations, skin reactions, or acneiform lesions. This does not include localized contact irritation at ECG lead sites due to application or removal of lead adhesive.

Refer to the separate rash workup plan for complete details, including reporting forms, and extra measures that must be performed to characterize any skin AESI of a newly acquired skin eruption that is non-traumatic. The trial site will have a local designated dermatologist available for immediate consultation during the trial for these AESIs.

#### 9.1.1 Adverse Events in the Double-Blind Treatment Period

TEAEs in the double-blind treatment period are defined as AEs with an onset date on or after the start of double-blind treatment. In more detail, TEAEs are all adverse events which started after start of double-blind IMP; or if the event was continuous from end of the single-blind placebo run-in period and was worsening, serious, study drug related, or resulted in death, discontinuation, interruption or reduction of study therapy. Adverse Events occurring up to 30 days after the last day of double-blind dosing will be included in the summary tables. The incidence of AEs in the double-blind treatment period will be tabulated by treatment group and overall using the Safety Sample. Incidence of TEAE during the double-blind treatment period of at least 5% in either centanafadine group and also greater than placebo by SOC and MedDRA PT will be provided.

Unless otherwise specified, in general, analysis of safety data will be performed on observed case and for last visit.

#### 9.1.2 Adverse Events in the Single-blind Placebo Run-in Period

Adverse Events in the single-blind placebo run-in period will be summarized for patients in the Safety Sample. AEs occurring up to 30 days after the last day of IMP in this period, but prior to the start of the double-blind treatment period, will be included in these summary tables. The incidence of adverse events in the single-blind placebo run-in period will be tabulated by the double-blind treatment patients receive in the double-blind treatment period.

#### 9.2 Clinical Laboratory Tests

Summary statistics for routine clinical laboratory measurements will be provided. For The double-blind treatment period laboratory tests, change from baseline for the double-blind treatment period will be summarized by treatment group. Potentially clinically relevant results in laboratory tests will also be summarized.

#### 9.2.1 Clinical Laboratory Tests in Double-Blind Treatment Period

Potentially clinically relevant laboratory measurement test results in the double-blind treatment period will be identified for the Safety Sample and will be summarized by treatment group and listed. Criteria for identifying laboratory values of potential clinical relevance are provided in Appendix 2.

# 9.2.2 Drug Induced Liver Injury (DILI)

Total bilirubin level should be checked for any subject with increased ALT or AST levels  $\geq$  three times the upper normal limits (ULN) or baseline.

| • | Reporting all DILI as SAE to the FDA based on Hy's Law: |
|---|---------------------------------------------------------|
| | $\square$ AST or ALT $\geq$ 3 x ULN or baseline and |

$$\Box$$
 T\_Bili  $\geq 2 \times ULN$  or baseline

A separate incidence table will be provided for DILI cases, and the corresponding listing will be provided for Safety Sample during the double-blind treatment period and the single-blind placebo run-in period.

## 9.2.3 Clinical Laboratory Tests in the Single-blind Placebo Run-in Period

Potentially clinically relevant laboratory measurement test results in the Single-blind Placebo Run-in Period will be summarized for the Safety Sample by treatment group and overall as well as listed by subject and by laboratory test.

#### 9.3 Vital Signs

Summary statistics for vital signs will be provided. For the double-blind treatment period vital signs, change from baseline for the double-blind treatment period will be summarized for the Safety Sample by treatment group. Potentially clinically relevant results in vital signs will also be summarized. Similar summaries will be provided for the Safety Sample during the Single-blind Placebo Run-in Period.

#### 9.3.1 Vital Signs in the Double-Blind Treatment Period

Potentially clinically relevant vital signs measurements identified in the double-blind treatment period for the Safety Sample will be summarized by treatment group. Criteria for identifying vital signs of potential clinical relevance are provided in Appendix 1. All potentially clinically relevant events or changes will be listed and included in summary tables.

#### 9.3.2 Vital Signs in the Single-blind Placebo Run-in Period

Potentially clinically relevant vital signs measurements identified in the Single-blind Placebo Run-in Period for the Safety Sample will be summarized by treatment group.

# 9.4 Electrocardiogram (ECG) Data

Summary statistics and incidence of potentially clinically relevant changes will be provided for ECG parameters.

For the analysis of QT and QTc, data from three consecutive complexes (representing three consecutive heart beats) will be measured to determine average values. The following QT corrections will be used for reporting purposes in the clinical study report:

- 1) QTcB is the length of the QT interval corrected for heart rate by the Bazett formula:  $QTcB=QT/(RR)^{0.5}$  and
- 2) QTcF is the length of the QT interval corrected for heart rate by the Fridericia formula:  $QTcF=QT/(RR)^{0.33}$
- 3) QTcN is the length of the QT interval corrected for heart rate by the FDA Neuropharm Division formula: QTcN=QT/(RR)<sup>0.37</sup>

#### 9.4.1 ECG Data in the Double-Blind Treatment Period

Potentially clinically relevant changes in the 12-lead ECG identified in the double-blind treatment period for the Safety Sample will be listed and summarized by treatment group. Criteria for identifying ECG measurements of potential clinical relevance are provided in Appendix 3.

Categorical changes in ECG parameters during the double-blind treatment period will be summarized based on the following criteria:

| Categorical Change Criteria in QT/QTc Parameters | | |
|---|---|---|
| Classification | Category | Criteria |
| QT | New Onset (> 450 Msec) | New onset (>450 msec) in QT means a subject who attains a value > 450 msec during treatment period but not at baseline. |
| QTc * | New Onset (> 450 Msec) | 0 Msec) New onset (> 450 msec) in QTc means a subject who attains a value > 450 msec during treatment period but not at baseline. |
| | New Onset (> 450 Msec)<br>And > 10% Increase | New onset (> 450 msec) and > 10% increase in QTc means a subject who attains a value > 450 msec and > 10% increase during treatment period but not at baseline |
| | New Onset (> 500 Msec) | New onset (> 500 msec) in QTc means a subject who attains a value > 500 msec during treatment period but not at baseline. |
| | Increase 30 - 60 Msec | Increase from baseline value $> 30$ and $\le 60$ msec in QTc |
| | Increase > 60 Msec | Increase from baseline value > 60 msec in QTc |

<sup>\*</sup> QTc categorical change criteria apply to QTcB, QTcF and QTcN.

## 9.4.2 ECG Data in the Single-blind Placebo Run-in Period

Potentially clinically relevant changes in the 12-lead ECG identified in the Single-blind Placebo Run-in Period for the Safety Sample will be listed and summarized by treatment group.

### 9.5 Physical Examinations

By-patient listings will be provided for physical examination.

# 9.5.1 Body Weight, Waist Circumference and Body Mass Index (BMI)

Analyses of body weight, waist circumference and BMI will be performed for the Safety Sample. The mean change from baseline of the double-blind treatment period to Day 42 (OC) and last visit in the double-blind treatment period in body weight will be tabulated and analyzed using ANCOVA. The ANCOVA models for both the OC and last visit analyses will

include the baseline of the double-blind treatment period body weight and the treatment group.

Percentages of patients showing significant weight gain ( $\geq 7$  % increase in weight), as well as percentages of patients showing significant weight loss ( $\geq 7$  % decrease in weight) baseline of the double-blind treatment period to Day 42 (OC and LOCF) will be analyzed using Cochran-Mantel-Haenszel (CMH) General Association Test.

Body mass index is defined as weight in kilograms divided by the square of height in meters.

### 9.6 Suicidality Data

Suicidality will be monitored during the study using the C-SSRS and will be summarized as number and percentage of subjects reporting any suicidal behavior, ideation, behavior by type (4 types), ideation by type (5 types) and treatment emergent suicidal behavior and ideation. Summary will be provided for the single-blind placebo run-in period and the double-blind treatment period for the Safety Sample.

Suicidality is defined as report of at least one occurrence of any type of suicidal ideation or at least one occurrence of any type of suicidal behavior during assessment period (count each person only once).

Treatment emergent suicidal behavior and ideation is summarized by four types: Emergence of suicidal ideation, Emergence of serious suicidal ideation, Worsening of suicidal ideation, Emergence of suicidal behavior.

Emergence of suicidal behavior/ideation is defined as report of any type of suicidal behavior/ideation during treatment when there was no baseline suicidal behavior/ideation.

Emergence of serious suicidal ideation is defined as observation of suicidal ideation severity rating of 4 or 5 during treatment when there was no baseline suicidal ideation.

Worsening of suicidal ideation is defined as a suicidal ideation severity rating that is more severe than it was at baseline.

For the double-blind treatment period analyses, the last available measurement prior to the first dose of double-blind IMP is being used as "Baseline".

#### **9.7 SMWQ**

Medication withdrawal symptoms assessed by SMWQ total scores at the scheduled visits during the double-blind treatment period and follow-up period will be summarized for the Safety Sample by treatment group and overall. The number of patients, mean, median, range and standard deviation will be presented.

# 9.8 Medication Handling Irregularities (MHIs) and Events Subject to Additional Monitoring (ESAMs)

MHIs and ESAMs will be summarized for the Safety Sample by treatment group and overall. By-patient listings will be provided.

#### 9.9 Concomitant Medications

Number and proportion of patients taking concomitant medications prior to the single-blind placebo run-in period, during the single-blind placebo run-in period, during the double-blind treatment period, and after study therapy are tabulated by drug classification using the World Health Organization (WHO) drug dictionary. For the double-blind treatment period Randomized Sample, data will be presented by treatment group and overall.

#### 9.10 Extent of Exposure

The start date of double-blind IMP - centanafadine or placebo - will be the first day of double-blind dosing. The number and percentage of subjects who receive double-blind IMP, will be presented by week and by treatment group. Each dosing week will be based on the actual week; i.e., Day 1-7 in Week 1, Day 8-14 in Week 2, etc. This summary will be performed on the Safety Sample.

The mean daily dosage will be summarized by week and treatment group using descriptive statistics. The mean daily dosage per subject per week will be determined for each week of the study. This will be calculated by dividing the sum of individual total doses by the number of days in the week interval. The summary will contain for each treatment group the number of patients receiving double-blind IMP, and the mean and range of the mean daily dose for each week.

#### 10 Conventions

#### 10.1 Study Visit Windows

Study visit windows will be used to map visits using study day intervals. This visit window convention applies to tables and listings for all efficacy and safety scales (AISRS, CGI-S, AIM-A, ASRS and CGI Change from Baseline). This derived study window variable will be named as DAY and will be footnoted. In listings it will be listed along with the eCRF study visit.

Table 10-1 shows classifications for study day intervals in the double-blind treatment period. The variable "target day" is defined using the number of days since the start of double-blind

dosing in the double-blind treatment period. The first day of double-blind dosing is defined as "Day 1".

If more than one observation falls within a particular study day interval, then the last observation within that interval is used. Evaluations occurring more than three days after the last double-blind dosing date and evaluations occurring during the follow-up period will not be mapped into study visit windows and will be excluded from the double-blind treatment period analysis.

Table 10-1: Study Day and Visit Windows in the Double-Blind Treatment Period

| Day | Target Day <sup>a</sup> | Study Day Interval <sup>a</sup> |
|-----|-------------------------|---------------------------------|
| 7 | 7 | 2-10 |
| 14 | 14 | 11-17 |
| 21 | 21 | 18-24 |
| 28 | 28 | 25-31 |
| 35 | 35 | 32-38 |
| 42 | 42 | 39-49 b |

<sup>&</sup>lt;sup>a</sup> Relative to the first day of double-blind IMP in the double-blind treatment period.

#### 10.2 Pooling of small centers

Primary efficacy analysis will be performed on the Efficacy Sample which comprises those subjects in the Randomized Sample who have a baseline value for the double-blind treatment period and at least one post-randomization value for AISRS total score in the double-blind treatment period. Small centers will be defined as centers that do not have at least one evaluable subject (evaluable with regard to the primary efficacy variable) in each treatment arm in the double-blind treatment period. All small centers will be pooled to form "pseudo centers" for the purpose of analysis according to the following algorithm. Small centers will be ordered from the largest to the smallest based on the number of evaluable subjects (i.e., subjects who have a baseline value for the double-blind treatment period value and at least one post-randomization value for AISRS total score in the double-blind treatment period). The process will start by pooling the largest of the small centers with the smallest of the small centers until a non-small center is formed. This process will be repeated using the centers left out of the previous pass. In case of ties in center size, the center with the smallest center code will be selected. If any centers are left out at the end of this process, they will be pooled with

b Evaluations occurring more than three days after the last double-blind dosing date and evaluations occurring during the follow-up period will be excluded from the double-blind treatment period analyses.

the smallest pseudo centers, or if no pseudo centers exist, they will be pooled with the smallest non-small center.

#### 10.3 Scales: Rules for Scoring and Handling of Missing Data

#### 10.3.1 Adult ADHD Investigator Symptom Rating Scale (AISRS)

The AISRS is utilized as the primary efficacy assessment of a subject's level of ADHD symptoms. It is a modified version of the ADHD Rating Scale that reflects the impact and severity of ADHD among adults and will be administered at each scheduled visit in the screening period, the single-blind placebo run-in period, the double-blind treatment period, and at 2 and 7 days after the last dose of IMP in the follow-up period. It is a clinician-administered scale that measures the 18 symptoms of adult ADHD using a Likert scale: 0 (none); 1 (mild); 2 (moderate); and 3 (severe) and uses a semi-structured interview methodology with suggested prompts for each item to improve interrater reliability. The scale's 18 items directly correspond to the 18 DSM-5 symptoms of ADHD where 9 inattentive items alternate with 9 hyperactive impulsive items. The maximum total score for the scale is 54 points, with 27 points for each subscale. The total score is the sum of both the Inattentive and Hyperactive Impulsive subscales.

The AISRS inattentive subscale score and hyperactive-impulsive subscale score, as well as the AISRS total score is set to be missing if more than one item of a subscale is missing for inattentive subscale or hyperactive-impulsive subscale, separately. If one item is missing for a given subscale (inattentive or hyperactive-impulsive), then the subscale score is derived as the mean of scores from the 8 non-missing items multiplied by 9. All imputed scores are rounded to the first decimal place. The 9 inattentive items consist of the 9 odd numbered items and the 9 hyperactive impulsive items consist of the 9 even numbered items.

# 10.3.2 Clinical Global Impression Severity of Illness Scale – Modified for Attention-Deficit Hyperactivity Disorder

The CGI-S modified is an observer-rated scale that will be used to measure symptom severity. To perform this assessment, the investigator or rater will respond to the following question: "Considering your total clinical experience with adult ADHD, how mentally ill is the patient at this time?" Response choices include: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients. CGI-S is assessed at each scheduled visit in the double-blind treatment period.

#### 10.3.3 Clinical Global Impression Change from Baseline

The CGI Change from Baseline is an observer-rated scale that will be used to measure the subject's total improvement compared to before trial drug treatment was initiated. The rater or investigator will rate the subject's total improvement relative to baseline. Response choices include: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. CGI Change from Baseline is assessed at each scheduled visit in the double-blind treatment period except for the Day -1 visit.

# 10.3.4 Attention-Deficit Hyperactivity Disorder Impact Module – Adult (AIM-A)

The AIM-A is a subject self-report questionnaire which assesses quality of life in adults with ADHD. The questionnaire has 4 global quality of life items, 5 economic impact items, and 5 multi-item scales that assess the following key concepts: Living with ADHD, General Well-Being, Work, Home and School Performance and Daily Functioning. Additionally, Relationships and Communication, and Impact of Symptoms are also included.

#### 10.3.5 Adult ADHD Self Report Scale (ASRS)

The ASRS is a self-report questionnaire developed by the WHO. The subject will answer 18 questions about the frequency of recent ADHD symptoms that are consistent with the DSM-IV criteria. The ASRS is assessed at the scheduled visits during the screening period, the single-blind placebo run-in period, and at Days -1, 28 and 42/ET during the double-blind treatment period.

The total score of (18 item) ADHD Symptoms score of the ASRS is set to be missing if more than one item of a subscale is missing for inattentive subscale or hyperactive-impulsive subscale, separately. If one item is missing for a given subscale (inattentive or hyperactive-impulsive), then the subscale score is derived as the mean of scores from the 8 non-missing items multiplied by 9. All imputed scores are rounded to the first decimal place. The 9 inattentive items consist of items 1-4 and 7-11 and the 9 hyperactive impulsive items consist of items 5-6 and 12-18.

# 10.3.6 Study Medication Withdrawal Questionnaire (SMWQ)

The SMWQ is a questionnaire to assess withdrawal symptoms. The SMWQ is a modification of the Amphetamine Withdrawal Questionnaire in which the terms "amphetamines and methamphetamine" are replaced with the term "the study medication." The SMWQ is assessed at Day 35 and Day 42/ET in the double-blind treatment period and at 1, 2, 3, 5, 7, and 10 days after the last dose of IMP in the follow-up period.

#### 10.3.7 Columbia-Suicide Severity Rating Scale (C-SSRS)

Suicidality will be monitored during the trial using the C-SSRS. The C-SSRS is a semi-structured interview that captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The interview includes definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behavior has occurred. The interview and rating for the C-SSRS must be completed by a licensed clinician who has been successfully trained to rate this scale by the sponsor or a designee and is medically responsible for the subject. Documentation of trial training should be maintained in the investigational site's files.

The C-SSRS has a "Screening/Baseline" version, which will be completed at screening and a "Since Last Visit" version that will be completed at all other visits (including the ET visit, if applicable). There are a maximum of 19 items to be completed: 7 required, 10 potential additional items if there is a positive response to a required item, and 2 items for suicide/suicide behavior present during the interview. The C-SSRS uses dichotomous scales (i.e., yes or no), Likert scales, and text or narrative to further describe the thoughts or behaviors.

The C-SSRS is assessed at each scheduled visit in the screening period, the single-blind placebo run-in period, the double-blind treatment period, and at 2 and 7 days after the last dose of IMP in the follow-up period.

#### 11 References

- Siddiqui O, Hung JHM, O'Neill R. MMRM vs. LOCF: A comprehensive comparison based on simulation study and 25 NDA datasets. J Biopharmaceutical Stats. 2009; 19(2):227-46.
- Diggle P, Kenward MG. Informative drop-out in longitudinal data analysis. Applied Statistics. 1994; 43:49-93.
- Little RJA. Pattern-mixture models for multivariate incomplete data. J Am Stat Assoc. 1993; 88:125-34.
- <sup>4</sup> Little RJA. Modeling the drop-out mechanism in repeated measures studies. J Am Stat Assoc. 1995; 90:1112-21.
- Hedeker D, Gibbons RD. Application of random effects pattern-mixture models for missing data in longitudinal studies. Psychological Methods. 1997; 2:64-78.
- Ali MW, Siddiqui O. Multiple imputation compared with some information dropout procedures in the estimation and comparison of rates of change in longitudinal clinical trials with dropouts. J Biopharmaceutical Stats. 2000;10(2):165-81.
- Wu MC, Bailey KR. Estimation and comparison of changes in the presence of informative right censoring: Conditional linear model. Biometrics. 1989; 45:939-55.
- van Elteren, PH. On the combination of independent two sample tests of Wilcoxon. Bull Int Stat Inst. 1960; 37:351-61.
- Mehrotra D, Li X, Liu J, Lu K. Analysis of Longitudinal Clinical Trials with Missing Data Using Multiple Imputation in Conjunction with Robust Regression. Biometrics 2012; 68:1250-1259.
- Cortina, J. M., & Nouri, H. (2000). Effect size for ANOVA designs. Thousand Oaks, Calif.: Sage Publications.

#### 12 Potential Clinical Relevance Criteria from Protocol

# Appendix 1 Criteria for Identifying Vital Signs of Potential Clinical Relevance

| Variable | Criterion Value <sup>a</sup> | Change Relative to Baseline <sup>a</sup> |
|---|---|---|
| Heart Rate <sup>b</sup> | > 100 bpm<br>< 50 bpm | ≥ 10 bpm increase<br>≥ 10 bpm decrease |
| Systolic Blood Pressure <sup>b</sup> | ≥ 140 mmHg<br>< 90 mmHg | ≥ 20 mmHg increase<br>≥ 20 mmHg decrease |
| Diastolic Blood Pressure <sup>b</sup> | $\geq 90 \text{ mmHg}$ $< 60 \text{ mmHg}$ | ≥ 10 mmHg increase<br>≥ 10 mmHg decrease |
| Orthostatic Hypotension | ≥ 30 mmHg decrease in systolic blood<br>pressure or a ≥ 20 mmHg<br>in diastolic blood pressure after at least<br>3 minutes of standing compared to the<br>previous supine blood pressure. | Not Applicable (baseline status not considered) |
| Orthostatic Tachycardia | ≥ 25 bpm increase in heart rate from supine to standing | Not Applicable (baseline status not considered) |
| Weight | - | ≥ 7% increase<br>≥ 7% decrease |

<sup>&</sup>lt;sup>a</sup> In order to be identified as potentially clinically relevant, an on-treatment value must meet the "Criterion Value" and also represent a change from the subject's baseline value of at least the magnitude shown in the "Change Relative to Baseline" column.

<sup>&</sup>lt;sup>b</sup> As defined in "Supplementary Suggestions for Preparing an Integrated Summary of Safety Information in an Original NDA Submission and for Organizing Information in Periodic Safety Updates," FDA Division of Neuropharmacological Drug Products draft (2/27/87).

Appendix 2 Criteria for Identifying Laboratory Values of Potential Clinical Relevance

| Laboratory Tests | Criteria |
|---|---|
| Chemistry | |
| AST (SGOT) | $\geq$ 3 x upper limit of normal (ULN) |
| ALT (SGPT) | $\geq 3 \times ULN$ |
| Alkaline phosphatase | $\geq$ 3 x ULN |
| BUN | $\geq 30 \text{ mg/dL}$ |
| Creatinine | $\geq 2.0 \text{ mg/dL}$ |
| Uric Acid | |
| Men | $\geq 10.5 \text{ mg/dL}$ |
| Women | $\geq 8.5 \text{ mg/dL}$ |
| Bilirubin (total) | $\geq 2.0 \text{ mg/dL}$ |
| Creatine Phosphokinase (CPK) | > 3 x ULN |
| Hematology | |
| Hematocrit | |
| Men | $\leq$ 37 % and decrease of $\geq$ 3 percentage points from Baseline |
| Women | $\leq$ 32 % and decrease of $\geq$ 3 percentage points from Baseline |
| Hemoglobin | |
| Men | $\leq 11.5 \text{ g/dL}$ |
| Women | $\leq 9.5 \text{ g/dL}$ |
| White blood count | $\leq 2,800/ \text{ mm}^3 \text{ or } \geq 16,000/ \text{ mm}^3$ |
| Eosinophils | ≥ 10% |
| Neutrophils | ≤ 15% |
| Absolute neutrophil count | $\leq 1,500/ \text{ mm}^3$ |
| Platelet count | $\leq 75,000/ \text{ mm}^3 \text{ or } \geq 700,000/ \text{ mm}^3$ |
| Urinalysis | |
| Protein | Increase of $\geq 2$ units |
| Glucose | Increase of $\geq 2$ units |
| Additional Criteria | |
| Chloride | $\leq$ 90 mEq/L or $\geq$ 118 mEq/L |
| Potassium | $\leq 2.5 \text{ mEq/L or} \geq 6.5 \text{ mEq/L}$ |
| Sodium | $\leq 126 \text{ mEq/L or} \geq 156 \text{ mEq/L}$ |
| Calcium | $\leq 8.2 \text{ mg/dL or} \geq 12 \text{ mg/dL}$ |
| Glucose | |
| Fasting | $\geq 100 \text{ mg/dL}$ |
| Non-Fasting | $\geq$ 200 mg/dL |
| Total Cholesterol, Fasting | $\geq 240 \text{ mg/dL}$ |
| LDL Cholesterol, Fasting | $\geq 160 \text{ mg/dL}$ |
| HDL Cholesterol, Fasting | Č |
| Men | < 40 mg/dL |
| Women | < 50 mg/dL |
| Triglycerides, Fasting | $\geq 150 \text{ mg/dL}$ |

# Appendix 3 Relevance

# Criteria for Identifying ECG Measurements of Potential Clinical

| Variable | Criterion Value <sup>a</sup> | Change Relative to Baseline <sup>a</sup> |
|---|---|---|
| Rate | | |
| Tachycardia | ≥ 120 bpm | increase of $\geq 15$ bpm |
| Bradycardia | ≤ 50 bpm | decrease of $\geq 15$ bpm |
| Rhythm | | |
| Sinus tachycardia <sup>b</sup> | ≥ 120 bpm | increase of ≥ 15 bpm |
| Sinus bradycardia <sup>c</sup> | ≤ 50 bpm | decrease of ≥ 15 bpm |
| Supraventricular premature beat | all | not present → present |
| Ventricular premature beat | all | not present → present |
| Supraventricular tachycardia | all | not present → present |
| Ventricular tachycardia | all | not present → present |
| Atrial fibrillation | all | not present $\rightarrow$ present |
| Atrial flutter | all | not present $\rightarrow$ present |
| Conduction | | |
| 1° atrioventricular block | $PR \ge 200 \text{ msec}$ | increase of $\geq 50$ msec |
| 2° atrioventricular block | all | not present $\rightarrow$ present |
| 3° atrioventricular block | all | not present $\rightarrow$ present |
| Left bundle-branch block | all | not present $\rightarrow$ present |
| Right bundle-branch block | all | not present $\rightarrow$ present |
| Pre-excitation syndrome | all | not present $\rightarrow$ present |
| Other intraventricular conduction block <sup>d</sup> | QRS $\geq$ 120 msec | increase of $\geq 20$ msec |
| Infarction | | |
| Acute or subacute | all | not present $\rightarrow$ present |
| Old | all | not present $\rightarrow$ present |
| | | ≥ 12 weeks post study entry |
| ST/T Morphological | | _ |
| Myocardial Ischemia | all | not present → present |
| Symmetrical T-wave inversion | all | not present $\rightarrow$ present |
| Increase in QTc | QTcF > 450 msec | |
| | (men)<br>QTcF > 470 msec | |
| | (women) | |

<sup>&</sup>lt;sup>a</sup> In order to be identified as potentially clinically relevant, an on-treatment value must meet the "Criterion Value" and also represent a change from the subject's baseline value of at least the magnitude shown in the "Change Relative to Baseline" column.

<sup>&</sup>lt;sup>b</sup> No current diagnosis of supraventricular tachycardia, ventricular tachycardia, atrial fibrillation, atrial flutter, or other rhythm abnormality.

<sup>&</sup>lt;sup>c</sup> No current diagnosis of atrial fibrillation, atrial flutter, or other rhythm abnormality.

<sup>&</sup>lt;sup>d</sup> No current diagnosis of left bundle branch block or right bundle branch block.
## 13 Proposed List of Summary Tables

- CT-1.1 Subject Disposition
- CT-1.2 Subject Disposition by Center
- CT-1.3 Subject Completion Rates by Week During the Double-Blind Treatment Period (Randomized Sample)
- CT-1.4.1 Subject Enrollment by Country (Randomized Sample)
- CT-1.4.2 Subject Enrollment by Country by Age Group (Randomized Sample)
- CT-2 Reasons for Discontinuation in the Double-Blind Treatment Period (Randomized Sample)
- CT-3.1 Demographic Characteristics (Randomized Sample)
- CT-3.2.1 Medical History (Randomized Sample)
- CT-3.2.2 Psychiatric History (Randomized Sample)
- CT-3.2.3 Summary of Adult ADHD Clinical Diagnostic Scale (ACDS) (Randomized Sample)
- CT-3.3 MINI International Neuropsychiatric Interview (M.I.N.I.) (Randomized Sample)
- CT-3.4.1 Baseline Psychiatric Scale Evaluations for the Single-Blind Placebo Run-in Period (Randomized Sample)
- CT-3.4.2 Baseline Psychiatric Scale Evaluations for the Double-Blind Treatment Period (Randomized Sample)
- CT-4.1 Concomitant Medications: Medications Taken Prior to Start of Double-Blind Treatment (Safety Sample)
- CT-4.2 Concomitant Medications: Medications Taken During the Double-Blind Treatment Period (Safety Sample)
- CT-4.3 Concomitant Medications: Medications Taken Post Study Period (Safety Sample)
- CT-5.1 Summary of Efficacy Results at Day 42 in the Double-Blind Treatment Period (Efficacy Sample)
- CT-5.2.1.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MMRM, UN (Efficacy Sample)
- CT-5.2.1.2 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MMRM, UN (Per Protocol Sample)
- CT-5.2.2 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MMRM, TOEPH Empirical (Efficacy Sample)
- CT-5.2.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MMRM, ARH1 Empirical (Efficacy Sample)
- CT-5.2.4 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MMRM, CSH Empirical (Efficacy Sample)
- CT-5.2.5 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MMRM, DDFM=SATTERTHWAITE (Efficacy Sample)
- CT-5.2.6.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score LOCF (Efficacy Sample)
- CT-5.2.6.2 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score OC (Efficacy Sample)
- CT-5.2.7 Summary of Mean Change from Baseline to End of the Single-Blind Run-in Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score OC (Efficacy Sample)

- CT-5.2.8 Summary of Mean Change from Baseline to End of the Follow-up Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score OC (Efficacy Sample)
- CT-5.3.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in AISRS Inattentive Subscale MMRM, UN (Efficacy Sample)
- CT-5.3.2 Summary of Mean Change Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in AISRS Inattentive Subscale LOCF (Efficacy Sample)
- CT-5.3.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day AISRS Inattentive Subscale OC (Efficacy Sample)
- CT-5.3.4 Summary of Mean Change from Baseline to End of Single-Blind Placebo Run-in Period in AISRS Inattentive Subscale OC (Efficacy Sample)
- CT-5.3.5 Summary of Mean Change from Baseline to End of the Follow-up Period in AISRS Inattentive Subscale OC (Efficacy Sample)
- CT-5.3.6 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in AISRS Hyperactive-Impulsive Subscale MMRM, UN (Efficacy Sample)
- CT-5.3.7 Summary of Mean Change Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in AISRS Hyperactive-Impulsive Subscale LOCF (Efficacy Sample)
- CT-5.3.8 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day AISRS Hyperactive-Impulsive Subscale OC (Efficacy Sample)
- CT-5.3.9 Summary of Mean Change from Baseline to End of Single-Blind Placebo Run-in Period in AISRS Hyperactive-Impulsive Subscale OC (Efficacy Sample)
- CT-5.3.10 Summary of Mean Change from Baseline to End of the Follow-up Period in AISRS Hyperactive-Impulsive Subscale - OC (Efficacy Sample)
- CT-5.4.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Clinical Global Impression Severity of Illness Modified for ADHD (CGI-S) Scale MMRM, UN (Efficacy Sample)
- CT-5.4.2 Summary of Mean Change Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Clinical Global Impression Severity of Illness Modified for ADHD (CGI-S) Scale LOCF (Efficacy Sample)
- CT-5.4.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Clinical Global Impression Severity of Illness Modified for ADHD (CGI-S) Scale OC (Efficacy Sample)
- CT-5.5.1 Summary of Mean Clinical Global Impression Change from Baseline Scale by Study Day in the Double-Blind Treatment Period LOCF (Efficacy Sample)
- CT-5.5.2 Summary of Mean Clinical Global Impression Improvement Change from Baseline Scale by Study Day in the Double-Blind Treatment Period OC (Efficacy Sample)
- CT-5.6.1 Summary of Proportion of Responders to Treatment During the Double-Blind Treatment Period Relative to the End of the Single-Blind Run-in Period LOCF (Efficacy Sample)
- CT-5.6.2 Summary of Proportion of Responders to Treatment During the Double-Blind Treatment Period Relative to the End of the Single-Blind Run-in Period OC (Efficacy Sample)
- CT-5.6.3 Summary of Proportion of Subjects with an Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score or a CGI Change from Baseline Response During the Double-Blind Treatment Period LOCF (Efficacy Sample)
- CT-5.6.4 Summary of Proportion of Subjects with an Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score or a CGI Change from Baseline Response During the Double-Blind Treatment Period OC (Efficacy Sample)
- CT-5.6.5 Summary of Proportion of Subjects with an Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score Remission During the Double-Blind Treatment Period LOCF (Efficacy Sample)
- CT-5.6.6 Summary of Proportion of Subjects with an Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score Remission During the Double-Blind Treatment Period OC (Efficacy Sample)

- CT-5.7.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Attention-Deficit Hyperactivity Disorder Impact Module Adult (AIM-A) Scale MMRM, UN (Efficacy Sample)
- CT-5.7.2 Summary of Mean Change Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Attention-Deficit Hyperactivity Disorder Impact Module Adult (AIM-A) Scale LOCF (Efficacy Sample)
- CT-5.7.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Attention-Deficit Hyperactivity Disorder Impact Module Adult (AIM-A) Scale OC (Efficacy Sample)
- CT-5.7.4 Summary of Mean Change from Baseline to End of Single-Blind Placebo Run-in Period in Attention-Deficit Hyperactivity Disorder Impact Module - Adult (AIM-A) Scale - OC (Efficacy Sample)
- CT-5.7.5 Summary of Proportion of Subjects in Each Category During the Single-Blind Run-in Period and Double-Blind Treatment Period by Study Day in Attention-Deficit Hyperactivity Disorder Impact Module Adult (AIM-A) Scale OC (Efficacy Sample)
- CT-5.8.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Self Report Scale (ASRS) Scale MMRM, UN (Efficacy Sample)
- CT-5.8.2 Summary of Mean Change Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Self Report Scale (ASRS) Scale LOCF (Efficacy Sample)
- CT-5.8.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Self Report Scale (ASRS) Scale OC (Efficacy Sample)
- CT-5.8.4 Summary of Mean Change from Baseline to End of Single-Blind Placebo Run-in Period in Adult ADHD Self Report Scale (ASRS) Scale OC (Efficacy Sample)
- CT-5.9.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in ASRS Inattentive Subscale MMRM, UN (Efficacy Sample)
- CT-5.9.2 Summary of Mean Change Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in ASRS Inattentive Subscale LOCF (Efficacy Sample)
- CT-5.9.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in ASRS Inattentive Subscale OC (Efficacy Sample)
- CT-5.9.4 Summary of Mean Change from Baseline to End of Single-Blind Placebo Run-in Period in ASRS Inattentive Subscale OC (Efficacy Sample)
- CT-5.9.5 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in ASRS Hyperactive-Impulsive Subscale MMRM, UN (Efficacy Sample)
- CT-5.9.6 Summary of Mean Change Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in ASRS Hyperactive-Impulsive Subscale LOCF (Efficacy Sample)
- CT-5.9.7 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in ASRS Hyperactive-Impulsive Subscale OC (Efficacy Sample)
- CT-5.9.8 Summary of Mean Change from Baseline to End of Single-Blind Placebo Run-in Period in ASRS Hyperactive-Impulsive Subscale OC (Efficacy Sample)
- CT-5.10.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MI, VAN ELTEREN TEST (Efficacy Sample)
- CT-5.10.2 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score GEE (Efficacy Sample)
- CT-5.10.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score WGEE (Efficacy Sample)
- CT-5.11.1 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 1) in AISRS Total Score Assume All Dropouts as MNAR (Efficacy Sample)

- CT-5.11.2 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 2) in AISRS Total Score Assume All Dropouts as MNAR (Efficacy Sample)
- CT-5.11.3 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 1) in AISRS Total Score Dropout due to AE or LOE or Withdrew Consent as MNAR (Efficacy Sample)
- CT-5.11.4 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 2) in AISRS Total Score Dropout due to AE or LOE or Withdrew Consent as MNAR (Efficacy Sample)
- CT-5.11.5 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 1) in AISRS Total Score Dropouts due to AE or Lack of Efficacy (LOE) as MNAR (Efficacy Sample)
- CT-5.11.6 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 2) in AISRS Total Score Dropouts due to AE or Lack of Efficacy (LOE) as MNAR (Efficacy Sample)
- CT-5.11.7 Sensitivity Analysis of MNAR using Placebo Based Imputation in AISRS Total Score (Efficacy Sample)
- CT-5.11.8 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 1) in CGI-S Score Assume All Dropouts as MNAR (Efficacy Sample)
- CT-5.11.9 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 2) in CGI-S Score Assume All Dropouts as MNAR (Efficacy Sample)
- CT-5.11.10 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 1) in CGI-S Score Dropout due to AE or LOE or Withdrew Consent as MNAR (Efficacy Sample)
- CT-5.11.11 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 2) in CGI-S Score Dropout due to AE or LOE or Withdrew Consent as MNAR (Efficacy Sample)
- CT-5.11.12 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 1) in SDS Mean Score Dropouts due to AE or Lack of Efficacy (LOE) as MNAR (Efficacy Sample)
- CT-5.11.13 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 2) in CGI-S Score Dropouts due to AE or Lack of Efficacy (LOE) as MNAR (Efficacy Sample)
- CT-5.11.14 Sensitivity Analysis of MNAR using Placebo Based Imputation in CGI-S Score (Efficacy Sample)
- CT-5.11.15 Sensitivity Analysis of MNAR Using Model Based Methods: Shared Parameter Model and Random Coefficient Pattern Mixture Model –OC (Efficacy Sample)
- CT-6.1.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS)Total Score in the Subgroup of Females MMRM (Efficacy Sample)
- CT-6.1.2 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score in the Subgroup of Males MMRM (Efficacy Sample)
- CT-6.2.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score in the Subgroup of Whites MMRM (Efficacy Sample)
- CT-6.2.2 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score in the Subgroup of All Other Races MMRM (Efficacy Sample)
- CT-7.1 Extent of Exposure to Study Medication During the Double-Blind Treatment Period (Safety Sample)
- CT-7.2 Number and Percentage of Subjects Receiving Study Medication and Mean and Range of Average Daily Dose in the Double-Blind Treatment Period (Safety Sample)
- CT-8.1.1 Adverse Events During the Double-Blind Treatment Period (All Causalities) (Safety Sample)
- CT-8.1.2 Adverse Events During the Single-Blind Placebo Run-in Period (All Causalities) (Safety Sample)
- CT-8.2.1.1 Incidence of TEAEs During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.1.2 Incidence of TEAEs During the Double-Blind Treatment Period by System Organ Class, MedDRA Preferred Term and Severity (Safety Sample)

- CT-8.2.1.3 Incidence of TEAE During the Double-Blind Treatment Period of at Least 5% in Any Centanafadine Group and Greater Than Placebo by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.1.4 Incidence of TEAEs During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term, by Sex (Safety Sample)
- CT-8.2.1.5 Incidence of TEAEs During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term, by Race (Safety Sample)
- CT-8.2.1.6 Incidence of Non-Serious TEAEs During the Double-Blind Treatment Period of at Least 5% in Any Centanafadine Group and Greater Than Placebo by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.1.7 Incidence of TEAE During the Double-Blind Treatment Period of at Least 2% in Any Centanafadine Group and Greater Than Placebo by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.1.8 Incidence and Occurrence (Number of Events) of Serious TEAEs by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.1.9 Incidence and Occurrence (Number of Events) of Potentially Drug-Related Serious TEAEs by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.1.10 Incidence and Occurrence (Number of Events) of Non-Serious TEAEs by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.2 Incidence of AEs During the Single-Blind Placebo Run-in Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.3.1 Incidence of Potentially Drug-Related TEAEs During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.3.2 Incidence of Potentially Drug-Related TEAEs During the Double-Blind Treatment Period by System Organ Class, MedDRA Preferred Term and Severity (Safety Sample)
- CT-8.4.1.1 Incidence of Deaths Due to TEAEs During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.4.1.2 Incidence of Deaths Due to TEAEs During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term and Severity (Safety Sample)
- CT-8.4.2 Incidence of Deaths Due to AEs During the Single-Blind Placebo Run-in Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.5.1.1 Incidence of Serious TEAEs During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.5.1.2 Incidence of Serious TEAEs During the Double-Blind Treatment Period by System Organ Class, MedDRA Preferred Term and Severity (Safety Sample)
- CT-8.5.2.1 Incidence of Serious AEs During the Single-Blind Placebo Run-in Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.6.1 Incidence of TEAEs Resulting in Discontinuation of Study Medication During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.6.2 Incidence of TEAEs Resulting in Discontinuation of Study Medication During the Double-Blind Treatment Period by System Organ Class, MedDRA Preferred Term and Severity (Safety Sample)
- CT-8.7.1 Incidence of Treatment-Emergent Adverse Events of Special Interests (AESIs) During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.7.2 Incidence of Treatment-Emergent Adverse Events of Special Interests (AESIs) During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term and Severity (Safety Sample)
- CT-8.7.3 Listing of Treatment-Emergent Adverse Events of Special Interests (AESIs) During the Double-Blind Treatment Period (Safety Sample)
- CT-8.8.1 Incidence of Treatment-Emergent Abuse Potential-Related Adverse Events During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term (Safety Sample)

- SAP 405-201-00013
- CT-8.8.2 Incidence of Treatment-Emergent Abuse Potential-Related Adverse Events During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term and Severity (Safety Sample)
- CT-8.8.3 Listing of Treatment-Emergent Abuse Potential-Related Adverse Events During the Double-Blind Treatment Period (Safety Sample)
- CT-9.1.1 Listing of Deaths During the Double-Blind Treatment Period
- CT-9.1.2 Listing of Deaths During the Single-Blind Placebo Run-in Period
- CT-9.2.1 Listing of Serious Adverse Events During the Double-Blind Treatment Period
- CT-9.2.2 Listing of Serious Adverse Events During the Single-Blind Placebo Run-in Period
- CT-9.3 Listing of Discontinuations of Study Medication Due to Adverse Events During the Double-Blind Treatment Period
- CT-9.4 Listing of Adverse Events for Subjects Discontinued from Study Due to Adverse Events During the Double-Blind Treatment Period
- CT-10.1 Criteria for Laboratory Test Values with Potential Clinical Relevance
- CT-10.2.1.1 Listing of Laboratory Test Values with Potential Clinical Relevance During the Double-Blind Treatment Period by Subject (Safety Sample)
- CT-10.2.1.2 Listing of Laboratory Test Values with Potential Clinical Relevance During the Double-Blind Treatment Period by Test (Safety Sample)
- CT-10.2.2 Incidence of Laboratory Test Values with Potential Clinical Relevance During the Double-Blind Treatment Period (Safety Sample)
- CT-10.2.3.1 Mean Change from Baseline of the Double-Blind Treatment Period in Clinical Laboratory Test Results Serum Chemistry (Safety Sample)
- CT-10.2.3.2 Mean Change from Baseline of the Double-Blind Treatment Period in Clinical Laboratory Test Results Hematology (Safety Sample)
- CT-10.2.3.3 Mean Change from Baseline of the Double-Blind Treatment Period in Clinical Laboratory Test Results Urinalysis (Safety Sample)
- CT-10.3.1.1 Listing of Laboratory Test Values with Potential Clinical Relevance During the Single-Blind Placebo Run-in Period by Subject (Safety Sample)
- CT-10.3.1.2 Listing of Laboratory Test Values with Potential Clinical Relevance During the Single-Blind Placebo Run-in Period by Test (Safety Sample)
- CT-10.3.2 Incidence of Laboratory Test Values with Potential Clinical Relevance During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-10.3.3.1 Mean Change from Baseline of the Single-Blind Placebo Run-in Period in Clinical Laboratory Test Results During the Single-Blind Placebo Run-in Period Serum Chemistry (Safety Sample)
- CT-10.3.3.2 Mean Change from Baseline of the Single-Blind Placebo Run-in Period in Clinical Laboratory Test Results During the Single-Blind Placebo Run-in Period Hematology (Safety Sample)
- CT-10.3.3.3 Mean Change from Baseline of the Single-Blind Placebo Run-in Period in Clinical Laboratory Test Results During the Single-Blind Placebo Run-in Period Urinalysis (Safety Sample)
- CT-10.4.1 Incidence of Potentially Liver Injury Related Laboratory Test Abnormalities During the Double-Blind Treatment Period (Safety Sample)
- CT-10.4.2 Incidence of Potentially Liver Injury Related Laboratory Test Abnormalities During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-10.5.1 Listing of Potentially Liver Injury Related Laboratory Test Abnormalities During the Double-Blind Treatment Period (Safety Sample)
- CT-10.5.2 Listing of Potentially Liver Injury Related Laboratory Test Abnormalities During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-11.1 Criteria for Potentially Clinically Relevant Abnormalities in Vital Signs
- CT-11.2.1 Listing of Potentially Clinically Relevant Abnormalities in Vital Signs During the Double-Blind Treatment Period (Safety Sample)

- CT-11.2.2 Incidence of Potentially Clinically Relevant Abnormalities in Vital Signs During the Double-Blind Treatment Period (Safety Sample)
- CT-11.2.3 Mean Change from Baseline of the Double-Blind Treatment Period in Vital Signs During the Double-Blind Treatment Period (Safety Sample)
- CT-11.3.1 Listing of Potentially Clinically Relevant Abnormalities in Vital Signs During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-11.3.2 Incidence of Potentially Clinically Relevant Abnormalities in Vital Signs During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-11.3.3 Mean Change from Baseline of the Single-Blind Placebo Run-in Period in Vital Signs During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-12.1 Criteria for Potentially Clinically Relevant Abnormalities in ECG Evaluations
- CT-12.2.1 Listing of Potentially Clinically Relevant Abnormalities in ECG Evaluations During the Double-Blind Treatment Period (Safety Sample)
- CT-12.2.2 Incidence of Potentially Clinically Relevant Changes in ECG Evaluations During the Double-Blind Treatment Period (Safety Sample)
- CT-12.2.3 Mean Change from Baseline of the Double-Blind Treatment Period in Electrocardiogram Results During the Double-Blind Treatment Period (Safety Sample)
- CT-12.3.1 Listing of Categorical Changes in QT/QTc During the Double-Blind Treatment Period (Safety Sample)
- CT-12.3.2 Incidence of Categorical Changes in QT/QTc During the Double-Blind Treatment Period (Safety Sample)
- CT-12.4.1 Listing of Potentially Clinically Relevant Abnormalities in ECG Evaluations During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-12.4.2 Incidence of Potentially Clinically Relevant Changes in ECG Evaluations During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-12.4.3 Mean Change from Baseline of the Single-Blind Placebo Run-in Period in Electrocardiogram Results During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-12.5.1 Listing of Categorical Changes in QT/QTc During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-12.5.2 Incidence of Categorical Changes in QT/QTc During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-13.1.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Body Weight (kg) (Safety Sample)
- CT-13.1.2 Summary of Proportion of Patients with Potentially Clinically Relevant Weight Gain or Weight Loss During the Double-Blind Treatment Period (Safety Sample)
- CT-13.2 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Waist Circumference (cm) (Safety Sample)
- CT-13.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in BMI (kg/m2) (Safety Sample)
- CT-14.1.1 Columbia-Suicide Severity Rating Scale(C-SSRS) During the Double-Blind Treatment Period, Suicidality (Safety Sample)
- CT-14.1.2 Columbia-Suicide Severity Rating Scale(C-SSRS) During the Double-Blind Treatment Period, Suicidal Behavior by Type (Safety Sample)
- CT-14.1.3 Columbia-Suicide Severity Rating Scale(C-SSRS) During the Double-Blind Treatment Period, Suicidal Ideation by Type (Safety Sample)
- CT-14.1.4 Columbia-Suicide Severity Rating Scale(C-SSRS) During the Double-Blind Treatment Period, Treatment Emergent Suicidal Behavior and Ideation (Safety Sample)
- CT-14.1.5 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Suicidal Ideation During the Double-Blind Treatment Period (Safety Sample)

- CT-14.1.6 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Suicidal Behavior During the Double-Blind Treatment Period (Safety Sample)
- CT-14.1.7 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Serious Suicidal Ideation During the Double-Blind Treatment Period (Safety Sample)
- CT-14.1.8 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Worsening Suicidal Ideation During the Double-Blind Treatment Period (Safety Sample)
- CT-14.2.1 Columbia-Suicide Severity Rating Scale (C-SSRS) During the Single-Blind Placebo Run-in Period, Suicidality (Safety Sample)
- CT-14.2.2 Columbia-Suicide Severity Rating Scale (C-SSRS) During the Single-Blind Placebo Run-in Period, Suicidal Behavior by Type (Safety Sample)
- CT-14.2.3 Columbia-Suicide Severity Rating Scale (C-SSRS) During the Single-Blind Placebo Run-in Period, Suicidal Ideation by Type (Safety Sample)
- CT-14.2.4 Columbia-Suicide Severity Rating Scale (C-SSRS) During the Single-Blind Placebo Run-in Period, Treatment Emergent Suicidal Behavior and Ideation (Safety Sample)
- CT-14.2.5 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Suicidal Ideation During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-14.2.6 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Suicidal Behavior During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-14.2.7 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Serious Suicidal Ideation During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-14.2.8 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Worsening Suicidal Ideation During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-15 Summary of Mean Study Medication Withdrawal Questionnaire (SMWQ) Total Score During the Double-Blind Treatment Period and Follow-up Period by Study Day (Safety Sample)
- CT-16 Summary of Medication Handling Irregularity (Safety Sample)
- CT-17.1 Summary of ESAMs Reported as Abuse Potential AEs During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-17.2 Summary of Non-Adverse Events Reported as Findings (ESAM) During the Double-Blind Treatment Period (Safety Sample)
- CT-17.3 Summary of ESAMs Reported as Abuse Potential AEs During the Single-Blind Placebo Run-in Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-17.4 Summary of Non-Adverse Events Reported as Findings (ESAM) During the Single-Blind Placebo Run-in Period (Safety Sample)



## This page is a manifestation of an electronically captured signature

### SIGNATURE PAGE

Document Name: 405-201-00013\_Statistical\_Analysis\_Plan

Document Number: 0001300268

**Document Version: 6.0** 

| Signed by | Meaning of Signature | Server Date (dd-MMM- yyyyy hh:min) - UTC timezone |
|---|---|---|
| | Clinical Approval | 27-Apr-2020<br>19:49:24 |
| | Biostatistics Approval | 27-Apr-2020<br>22:34:44 |

CENTANAFADINE 1 OF 5
PROTOCOL 405-201-00013

 ${\tt STAT-1.1} \\ {\tt Adjusted Mean Change from Baseline in AISRS Line Items at Day 42 - MMRM} \\ ({\tt Efficacy Sample})$ 

CTN SR 200MG CTN SR 400MG PLACEBO COHEN's D AISRS MEAN LSMean MEAN LSMean TREATMENT MEAN LSMean TREATMENT EFFECT N Base Change¹ N Base Change¹ N Base Change¹ COMPARISON EFFECT 1 P-VALUE1 SIZE Line Items EB-1020 200mg VS MAKE CARELESS MISTAKES 147 2.23 -0.61 147 2.17 -0.61 144 2.27 -0.32 -0.29 0.0080 -0.31 PLACEBO EB-1020 400mg VS -0.29 0.0064 -0.32 PLACEBO EB-1020 200mg VS FIDGET OR SQUIRM WITH 147 2.37 -0.49 147 2.33 -0.50 144 2.28 -0.23 -0.26 0.0120 -0.30 YOUR HANDS OR FEET PLACEBO EB-1020 400mg VS -0.27 0.0084 -0.31 PLACEBO EB-1020 200mg VS 147 2.74 -0.76 147 2.67 -0.69 144 2.58 -0.40 -0.36 0.0014 -0.38 DIFFICULTY KEEPING YOUR ATTENTION PLACEBO EB-1020 400mg VS -0.28 0.0094 -0.31 PLACEBO LEAVE YOUR SEAT 147 1.77 -0.56 147 1.79 -0.62 144 1.78 -0.46 EB-1020 200mg VS -0.10 0.3832 -0.10 PLACEBO EB-1020 400mg VS -0.16 0.1456 -0.17PLACEBO DIFFICULTY 147 2.37 -0.80 147 2.42 -0.60 144 2.41 -0.48 EB-1020 200mg VS -0.32 0.0033 -0.35 CONCENTRATING ON PLACEBO

<sup>&</sup>lt;sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE 2 OF 5

 ${\tt STAT-1.1} \\ {\tt Adjusted Mean Change from Baseline in AISRS Line Items at Day 42 - MMRM} \\ ({\tt Efficacy Sample})$ 

CTN SR 200MG CTN SR 400MG COHEN's D ESTIMATED AISRS MEAN LSMean MEAN LSMean MEAN LSMean MEAN LSMean TREATMENT TREATMENT EFFECT Line Items N Base Change¹ N Base Change¹ N Base Change¹ COMPARISON EFFECT P-VALUE¹ SIZE EFFECT DIFFICULTY EB-1020 400mg VS -0.12 0.2531 -0.13 CONCENTRATING ON PLACEBO FEEL RESTLESS OR 147 2.18 -0.47 147 2.20 -0.54 144 2.10 -0.36 EB-1020 200mg VS -0.10 0.3769 -0.10 FIDGETY PLACEBO EB-1020 400mg VS -0.18 0.1134 -0.19 PLACEBO 147 2.58 -0.69 147 2.52 -0.54 144 2.51 -0.35 TROUBLE WRAPPING UP EB-1020 200mg VS -0.34 0.0040 -0.34 THE FINAL DETAILS PLACEBO EB-1020 400mg VS -0.19 0.1020 -0.19 PLACEBO -0.08 DIFFICULTY UNWINDING 147 1.84 -0.47 147 1.96 -0.40 144 1.86 -0.39 EB-1020 200mg VS 0.4738 -0.08 AND RELAXING PLACEBO EB-1020 400mg VS -0.02 0.8874 -0.02 PLACEBO DIFFICULTY GETTING 147 2.50 -0.60 147 2.49 -0.64 144 2.47 -0.38 EB-1020 200mg VS -0.21 0.0691 -0.21 THINGS IN ORDER PLACEBO

EB-1020 400mg VS

PLACEBO

-0.26

0.0256

-0.26

<sup>&</sup>lt;sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE 3 OF 5

 ${\tt STAT-1.1} \\ {\tt Adjusted Mean Change from Baseline in AISRS Line Items at Day 42 - MMRM} \\ ({\tt Efficacy Sample})$ 

CTN SR 200MG CTN SR 400MG COHEN's D ESTIMATED AISRS MEAN LSMean MEAN LSMean MEAN LSMean TREATMENT TREATMENT EFFECT N Base Change¹ N Base Change¹ N Base Change¹ COMPARISON Line Items EFFECT 1 P-VALUE1 SIZE OVERLY ACTIVE AND 147 2.05 -0.55 147 2.08 -0.55 144 1.93 -0.38 EB-1020 200mg VS -0.17 0.1608 -0.16 COMPELLED TO DO THINGS PLACEBO EB-1020 400mg VS -0.17 0.1541 -0.17 PLACEBO AVOID OR DELAY 147 2.63 -0.71 147 2.52 -0.55 144 2.65 -0.45 EB-1020 200mg VS -0.26 0.0348 -0.25 GETTING STARTED PLACEBO EB-1020 400mg VS -0.10 0.3848 -0.10 PLACEBO TALKING TOO MUCH 147 1.89 -0.62 147 1.75 -0.50 144 1.80 -0.34 EB-1020 200mg VS -0.27 0.0148 -0.29 PLACEBO EB-1020 400mg VS -0.15 0.1649 -0.16 PLACEBO MISPLACE OR HAVE 147 2.23 -0.54 147 2.16 -0.49 144 2.35 -0.47 EB-1020 200mg VS -0.07 0.5480 -0.07 DIFFICULTY FINDING PLACEBO -0.02 0.8648 EB-1020 400mg VS -0.02 PLACEBO FINISHING THE 147 1.89 -0.64 147 1.93 -0.65 144 2.00 -0.53 EB-1020 200mg VS -0.11 0.3294 -0.11 SENTENCES OF THE PLACEBO PEOPLE

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE 4 OF 5

 ${\tt STAT-1.1} \\ {\tt Adjusted Mean Change from Baseline in AISRS Line Items at Day 42 - MMRM} \\ ({\tt Efficacy Sample})$ 

CTN SR 200MG CTN SR 400MG COHEN's D ESTIMATED MEAN LSMean MEAN LSMean MEAN LSMean TREATMENT AISRS TREATMENT EFFECT AISRS MEAN LSMean MEAN LSMean MEAN LSMean TREATMENT TREATMENT EFFECT
Line Items N Base Change¹ N Base Change¹ N Base Change¹ COMPARISON EFFECT ¹ P-VALUE¹ SIZE FINISHING THE EB-1020 400mg VS -0.12 0.2683 -0.13 SENTENCES OF THE PLACEBO PEOPLE BEING DISTRACTED BY 147 2.59 -0.56 147 2.58 -0.55 144 2.59 -0.30 EB-1020 200mg VS -0.26 0.0229 -0.27 ACTIVITY OR NOISE PLACEBO EB-1020 400mg VS -0.24 0.0311 -0.25 PLACEBO 147 1.91 -0.39 147 1.99 -0.55 144 1.88 -0.39 -0.01 0.9533 DIFFICULTY WAITING EB-1020 200mg VS -0.01 YOUR TURN PLACEBO EB-1020 400mg VS -0.16 0.1284 -0.18 PLACEBO PROBLEMS REMEMBERING 147 2.13 -0.54 147 2.18 -0.77 144 2.26 -0.63 EB-1020 200mg VS 0.09 0.4350 0.09 PLACEBO -0.14 EB-1020 400mg VS 0.2301 -0.14 PLACEBO INTERRUPT OTHERS WHEN 147 1.69 -0.62 147 1.82 -0.58 144 1.80 -0.54 -0.08 0.4580 EB-1020 200mg VS -0.09 THEY ARE BUSY PLACEBO EB-1020 400mg VS -0.04 0.7183 -0.04 PLACEBO

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE 5 OF 5 PROTOCOL 405-201-00013

# $$\tt STAT-1.1$$ Adjusted Mean Change from Baseline in AISRS Line Items at Day 42 - MMRM (Efficacy Sample)

| AISRS<br>Line Items | CTN SR 200MG<br>MEAN LSMean<br>N Base Change <sup>1</sup> | CTN SR 400MG<br>MEAN LSMean<br>N Base Change <sup>1</sup> | PLACEBO MEAN LSMean TREATN N Base Change¹ COMPAF | | EFFECT |
|---|---|---|---|---|---|
| AISRS TOTAL SCORE | 147 39.60 -10.1 | 147 39.56 -9.73 | 144 39.53 -6.98 EB-102 | 20 200mg VS -3.15 | 0.0193 -0.28 |
| (DEKIVED) | | | | 20 400mg VS -2.74 | 0.0392 -0.24 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE 1 OF 5

# $\begin{array}{c} {\rm STAT-1.2} \\ {\rm Adjusted\ Mean\ Change\ from\ Baseline\ in\ ASRS\ Line\ Items\ at\ Day\ 42\ -\ MMRM} \\ {\rm (Efficacy\ Sample)} \end{array}$

CTN SR 200MG CTN SR 400MG PLACEBO COHEN's D ESTIMATED ASRS MEAN LSMean MEAN LSMean TREATMENT MEAN LSMean TREATMENT EFFECT N Base Change¹ N Base Change¹ N Base Change¹ COMPARISON EFFECT 1 P-VALUE1 SIZE Line Items EB-1020 200mg VS ASRS-TROUBLE TO WRAP 118 3.10 -0.55 127 3.05 -0.57 131 2.97 -0.26 -0.29 0.0210 -0.29 DETAILS OF PROJECT PLACEBO EB-1020 400mg VS -0.31 0.0129 -0.31 PLACEBO ASRS-DIFFICULTY 118 3.25 -0.59 127 3.08 -0.66 131 3.03 -0.38 EB-1020 200mg VS -0.22 0.0855 -0.22 GETTING THINGS IN PLACEBO ORDER EB-1020 400mg VS -0.28 0.0196 -0.29 PLACEBO ASRS-PROBLEM 118 2.86 -0.62 127 2.80 -0.78 131 2.79 -0.41 EB-1020 200mg VS -0.21 0.1187 -0.20 REMEMBERING PLACEBO APPTS/OBLIGATNS EB-1020 400mg VS -0.37 0.0050 -0.35PLACEBO -0.30 118 3.36 -0.66 127 3.31 -0.66 131 3.31 -0.36 EB-1020 200mg VS 0.0188 -0.30 ASRS-AVOID/DELAY GETTNG STARTD ON PLACEBO THGHTS EB-1020 400mg VS -0.30 0.0159 -0.30 PLACEBO

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE 2 OF 5

 $\begin{array}{c} {\rm STAT-1.2} \\ {\rm Adjusted~Mean~Change~from~Baseline~in~ASRS~Line~Items~at~Day~42~-MMRM} \\ {\rm (Efficacy~Sample)} \end{array}$ 

| ASRS<br>Line Items | | TN SR<br>MEAN<br>Base | 200MG<br>LSMean<br>Change <sup>1</sup> | | IN SR<br>MEAN<br>Base | 400MG<br>LSMean<br>Change <sup>1</sup> | N | PLAC<br>MEAN<br>Base | | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE¹ | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ASRS-FIDGET/SQUIRM<br>WITH HANDS/FEET | 118 | 3.11 | -0.56 | 127 | 3.18 | -0.56 | 131 | 3.10 | -0.31 | EB-1020 200mg VS<br>PLACEBO | -0.26 | 0.0490 | -0.25 |
| | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.25 | 0.0497 | -0.25 |
| ASRS-FEEL OVERLY<br>ACTIVE TO DO THINGS | 118 | 2.58 | -0.56 | 127 | 2.76 | -0.72 | 131 | 2.66 | -0.35 | EB-1020 200mg VS<br>PLACEBO | -0.20 | 0.1266 | -0.19 |
| | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.37 | 0.0047 | -0.35 |
| ASRS-MAKE CARELESS | 118 | 2.98 | -0.65 | 127 | 2.72 | -0.67 | 131 | 2.97 | -0.38 | EB-1020 200mg VS<br>PLACEBO | -0.26 | 0.0357 | -0.27 |
| | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.29 | 0.0216 | -0.29 |
| ASRS-DIFFICULTY KEEPING ATTENTION | 118 | 3.45 | -0.61 | 127 | 3.36 | -0.66 | 131 | 3.32 | -0.37 | EB-1020 200mg VS<br>PLACEBO | -0.24 | 0.0717 | -0.23 |
| | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.29 | 0.0235 | -0.28 |
| ASRS-DIFFICULTY KEEPING CONCENTRATION | 118 | 3.02 | -0.80 | 127 | 3.09 | -0.80 | 131 | 3.12 | -0.47 | EB-1020 200mg VS<br>PLACEBO | -0.33 | 0.0129 | -0.32 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE 3 OF 5

 $\begin{array}{c} {\rm STAT-1.2} \\ {\rm Adjusted\ Mean\ Change\ from\ Baseline\ in\ ASRS\ Line\ Items\ at\ Day\ 42\ -\ MMRM} \\ {\rm (Efficacy\ Sample)} \end{array}$ 

CTN SR 200MG CTN SR 400MG COHEN's D ESTIMATED ASRS MEAN LSMean MEAN LSMean MEAN LSMean TREATMENT TREATMENT EFFECT Line Items N Base Change¹ N Base Change¹ N Base Change¹ COMPARISON EFFECT P-VALUE¹ SIZE EFFECT ASRS-DIFFICULTY EB-1020 400mg VS -0.33 0.0107 -0.32 KEEPING CONCENTRATION PLACEBO ASRS-MISPLACE/DIFFICUL 118 3.05 -0.63 127 2.98 -0.69 131 3.07 -0.50 EB-1020 200mg VS -0.13 0.3334 -0.12 TY FINDING THINGS PLACEBO EB-1020 400mg VS -0.19 0.1470 -0.18 PLACEBO ASRS-DISTRACTED BY 118 3.25 -0.63 127 3.28 -0.61 131 3.30 -0.28 EB-1020 200mg VS -0.35 0.0130 -0.32 ACTIVITY OR NOISE PLACEBO EB-1020 400mg VS -0.32 0.0184 -0.29 PLACEBO ASRS-LEAVE SEAT IN 118 2.26 -0.59 127 2.14 -0.70 131 2.02 -0.32 EB-1020 200mg VS -0.27 0.0307 -0.28 MEETNGS/ORDR SITUATNS PLACEBO EB-1020 400mg VS -0.39 0.0015 -0.40 PLACEBO ASRS-FEELING RESTLESS 118 2.97 -0.56 127 3.02 -0.68 131 2.98 -0.34 EB-1020 200mg VS -0.22 0.0909 -0.22 OR FIDGETY PLACEBO EB-1020 400mg VS -0.34 0.0093 -0.33 PLACEBO

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE 4 OF 5

 $\begin{array}{c} {\rm STAT-1.2} \\ {\rm Adjusted\ Mean\ Change\ from\ Baseline\ in\ ASRS\ Line\ Items\ at\ Day\ 42\ -\ MMRM} \\ {\rm (Efficacy\ Sample)} \end{array}$ 

CTN SR 200MG CTN SR 400MG COHEN's D ESTIMATED MEAN LSMean MEAN LSMean TREATMENT ASRS MEAN LSMean TREATMENT EFFECT MEAN LSMean MEAN LSMean MEAN LSMean TREATMENT TREATMENT EFFECT

N Base Change¹ N Base Change¹ N Base Change¹ COMPARISON EFFECT ¹ P-VALUE¹ SIZE Line Items EB-1020 200mg VS ASRS-DIFF UNWINDING 118 2.60 -0.55 127 2.91 -0.55 131 2.76 -0.32 -0.23 0.0946 -0.21 AND RELAXING PLACEBO EB-1020 400mg VS -0.23 0.0835 -0.22 PLACEBO ASRS-FIND YOURSELF 118 2.64 -0.70 127 2.59 -0.68 131 2.66 -0.38 EB-1020 200mg VS -0.32 0.0170 -0.30 TALKING TOO MUCH PLACEBO EB-1020 400mg VS -0.29 0.0251 -0.28 PLACEBO ASRS-FINISH SENTENCES 118 2.70 -0.78 127 2.66 -0.78 131 2.73 -0.50 EB-1020 200mg VS -0.28 0.0417 -0.26 OF PEOPLE PLACEBO EB-1020 400mg VS -0.28 0.0405 -0.26 PLACEBO ASRS-DIFFCULTY 118 2.57 -0.60 127 2.65 -0.82 131 2.44 -0.40 EB-1020 200mg VS -0.20 0.1576 -0.18 WAITING YOUR TURN PLACEBO -0.42 0.0028 EB-1020 400mg VS -0.38 PLACEBO ASRS-INTERRUPT OTHERS 118 2.46 -0.82 127 2.48 -0.81 131 2.46 -0.62 EB-1020 200mg VS -0.20 0.1216 -0.20 WHEN THEY ARE BUSY PLACEBO

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO


# $\begin{array}{c} {\rm STAT-1.2} \\ {\rm Adjusted~Mean~Change~from~Baseline~in~ASRS~Line~Items~at~Day~42~-MMRM} \\ {\rm (Efficacy~Sample)} \end{array}$

| ASRS<br>Line Items | CTN SR 200MG<br>MEAN LSMean<br>N Base Change | CTN SR 400MG<br>MEAN LSMean<br>N Base Change | PLACEBO<br>MEAN LSMean<br>N Base Change <sup>1</sup> | TREATMENT<br>COMPARISON | ESTIMATED TREATMENT EFFECT 1 P-VALUE | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|
| ASRS-INTERRUPT OTHERS WHEN THEY ARE BUSY | | | | EB-1020 400mg VS<br>PLACEBO | -0.19 0.1325 | -0.19 |
| ASRS TOTAL SCORE OF<br>18 ITEMS (DERIVED) | 118 52.22 -11.3 | 127 52.06 -12.0 | 131 51.67 -6.70 | EB-1020 200mg VS<br>PLACEBO<br>EB-1020 400mg VS<br>PLACEBO | -4.60 0.0062<br>-5.28 0.0014 | |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE 1 OF 28 PROTOCOL 405-201-00013

STAT-3.1

MMRM Output for Test on Treatment by Sex Interaction at Day 42

(Efficacy Sample)

\_\_\_\_\_

### The Mixed Procedure

#### Model Information

Data Set WORK.INDATA
Dependent Variable CHG
Covariance Structure Unstructured
Subject Effect SUBJID
Estimation Method REML
Residual Variance Method Fixed Effects SE Method
Degrees of Freedom Method Kenward-Roger

### Class Level Information

| Class | Levels | Values |
|------------------------------|--------------|---------------------------|
| AVISITN<br>TRTPN<br>POOLCNTR | 6<br>3<br>38 | 7 14 21 28 35 42<br>1 2 3 |

CENTANAFADINE
2 OF 28

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Class Level Information

Class Levels Values
SUBJID 438

CENTANAFADINE 3 OF 28 PROTOCOL 405-201-00013

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure



CENTANAFADINE 4 OF 28 PROTOCOL 405-201-00013

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure



CENTANAFADINE 5 OF 28 PROTOCOL 405-201-00013

STAT-3.1

MMRM Output for Test on Treatment by Sex Interaction at Day 42

(Efficacy Sample)

......

The Mixed Procedure



CENTANAFADINE 6 OF 28 PROTOCOL 405-201-00013

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

......

The Mixed Procedure



CENTANAFADINE 7 OF 28 PROTOCOL 405-201-00013

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42  $(\tt Efficacy\ Sample)$ 

......

The Mixed Procedure



| CENTANAFADINE | 8 OF 28 |
|------------------------|---------|

 $$\operatorname{STAT-3.1}$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42  $$\left(\operatorname{Efficacy\ Sample}\right)$$ 

......

The Mixed Procedure

Class Level Information

Class Levels Values

SEX

Dimensions

2 F M

Covariance Parameters 21
Columns in X 128
Columns in Z 0
Subjects 438
Max Obs per Subject 6

Number of Observations

Number of Observations Read 2292 Number of Observations Used 2292 Number of Observations Not Used 0

CENTANAFADINE 9 OF 28 PROTOCOL 405-201-00013

STAT-3.1

MMRM Output for Test on Treatment by Sex Interaction at Day 42  $\,$  (Efficacy Sample)

......

The Mixed Procedure

Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 16471.93771301 | |
| 1 | 2 | 14206.06433817 | 0.00014910 |
| 2 | 1 | 14205.26506836 | 0.00000141 |
| 3 | 1 | 14205.25788280 | 0.00000000 |

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | 52.3976 |
| UN(2,1) | SUBJID | 40.2284 |
| UN(2,2) | SUBJID | 72.6755 |
| UN(3,1) | SUBJID | 38.1964 |
| UN(3,2) | SUBJID | 62.4528 |
| UN(3,3) | SUBJID | 81.8612 |
| UN(4,1) | SUBJID | 37.6894 |
| UN(4,2) | SUBJID | 63.0768 |

CENTANAFADINE 10 OF 28 PROTOCOL 405-201-00013

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

### The Mixed Procedure

#### Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(4,3) | SUBJID | 77.7325 |
| UN (4,4) | SUBJID | 105.92 |
| UN(5,1) | SUBJID | 38.4856 |
| UN(5,2) | SUBJID | 63.7432 |
| UN(5,3) | SUBJID | 81.2609 |
| UN(5,4) | SUBJID | 96.6536 |
| UN(5,5) | SUBJID | 111.49 |
| UN(6,1) | SUBJID | 38.7755 |
| UN(6,2) | SUBJID | 64.7203 |
| UN(6,3) | SUBJID | 79.0855 |
| UN(6,4) | SUBJID | 96.9247 |
| UN(6,5) | SUBJID | 99.9728 |
| UN(6,6) | SUBJID | 118.03 |

### Fit Statistics

| -2 Res Log Likelihood | 14205.3 |
|--------------------------|---------|
| AIC (Smaller is Better) | 14247.3 |
| AICC (Smaller is Better) | 14247.7 |
| BIC (Smaller is Better) | 14333.0 |

CENTANAFADINE 11 OF 28 PROTOCOL 405-201-00013

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 20 2266.68 <.0001

Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|-------------------|-----------|-----------|---------|--------|
| POOLCNTR | 37 | 393 | 2.24 | <.0001 |
| AVISITN | 5 | 377 | 2.31 | 0.0434 |
| TRTPN | 2 | 396 | 3.03 | 0.0495 |
| AVISITN*TRTPN | 10 | 558 | 1.63 | 0.0954 |
| SEX | 1 | 412 | 0.02 | 0.8821 |
| AVISITN*SEX | 5 | 376 | 1.58 | 0.1649 |
| TRTPN*SEX | 2 | 408 | 0.17 | 0.8404 |
| AVISITN*TRTPN*SEX | 10 | 558 | 0.54 | 0.8603 |
| BASE*AVISITN | 6 | 402 | 2.38 | 0.0287 |

CENTANAFADINE 12 OF 28 PROTOCOL 405-201-00013

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42  $(\tt Efficacy\ Sample)$ 

The Mixed Procedure

Coefficients for 1 vs. 3 BY SEX AT DAY 42

| Effect | Pooled<br>Center<br>Number | Sex | Analysis<br>Visit<br>(N) | Row1 |
|---|---|---|---|---|
| Intercept | | | | |
| POOLCNTR | | | | |

CENTANAFADINE 13 OF 28 PROTOCOL 405-201-00013

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Coefficients for 1 vs. 3 BY SEX AT DAY 42

| Eff | ect | Pooled<br>Center<br>Number | Sex | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| 200 | T CHEED | | | | | |
| | LCNTR | | | | | |
| | LCNTR | | | | | |
| | LCNTR | | | | | |
| POO | LCNTR | | | | | |
| | LCNTR | | | | | |
| | - | | | | | |

CENTANAFADINE 14 OF 28 PROTOCOL 405-201-00013

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

\_\_\_\_\_

Parameter Code=AISRSTOT ------

### The Mixed Procedure

Coefficients for 1 vs. 3 BY SEX AT DAY 42

| | Pooled | | Analysis | Planned | |
|---------------|--------|-----|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | Sex | (N) | (N) | Row1 |
| POOLCNTR | | | | | |
| AVISITN | | | 7 | | |
| AVISITN | | | 14 | | |
| AVISITN | | | 21 | | |
| AVISITN | | | 28 | | |
| AVISITN | | | 35 | | |
| AVISITN | | | 42 | | |
| TRTPN | | | | 1 | |
| TRTPN | | | | 2 | |
| TRTPN | | | | 3 | |
| AVISITN*TRTPN | | | 7 | 1 | |
| AVISITN*TRTPN | | | 7 | 2 | |
| AVISITN*TRTPN | | | 7 | 3 | |
| AVISITN*TRTPN | | | 14 | 1 | |
| AVISITN*TRTPN | | | 14 | 2 | |
| AVISITN*TRTPN | | | 14 | 3 | |
| AVISITN*TRTPN | | | 21 | 1 | |
| AVISITN*TRTPN | | | 21 | 2 | |
| AVISITN*TRTPN | | | 21 | 3 | |


CENTANAFADINE 15 OF 28

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

Parameter Code=AISRSTOT ------

The Mixed Procedure

Coefficients for 1 vs. 3 BY SEX AT DAY 42

| | Pooled | | Analysis | Planned | |
|---------------|--------|-----|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | Sex | (N) | (N) | Row1 |
| AVISITN*TRTPN | | | 28 | 1 | |
| AVISITN*TRTPN | | | 28 | 2 | |
| AVISITN*TRTPN | | | 28 | 3 | |
| AVISITN*TRTPN | | | 35 | 1 | |
| AVISITN*TRTPN | | | 35 | 2 | |
| AVISITN*TRTPN | | | 35 | 3 | |
| AVISITN*TRTPN | | | 42 | 1 | |
| AVISITN*TRTPN | | | 42 | 2 | |
| AVISITN*TRTPN | | | 42 | 3 | |
| SEX | | F | | | |
| SEX | | M | | | |
| AVISITN*SEX | | F | 7 | | |
| AVISITN*SEX | | M | 7 | | |
| AVISITN*SEX | | F | 14 | | |
| AVISITN*SEX | | M | 14 | | |
| AVISITN*SEX | | F | 21 | | |
| AVISITN*SEX | | M | 21 | | |
| AVISITN*SEX | | F | 28 | | |
| AVISITN*SEX | | M | 28 | | |

CENTANAFADINE 16 OF 28 PROTOCOL 405-201-00013

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

Parameter Code=AISRSTOT ------

### The Mixed Procedure

Coefficients for 1 vs. 3 BY SEX AT DAY 42

| | Pooled | | Analysis | Planned | |
|-------------------|--------|-----|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | Sex | (N) | (N) | Row1 |
| AVISITN*SEX | | F | 35 | | |
| AVISITN*SEX | | M | 35 | | |
| AVISITN*SEX | | F | 42 | | |
| AVISITN*SEX | | M | 42 | | |
| TRTPN*SEX | | F | | 1 | 1 |
| TRTPN*SEX | | M | | 1 | -1 |
| TRTPN*SEX | | F | | 2 | |
| TRTPN*SEX | | M | | 2 | |
| TRTPN*SEX | | F | | 3 | -1 |
| TRTPN*SEX | | M | | 3 | 1 |
| AVISITN*TRTPN*SEX | | F | 7 | 1 | |
| AVISITN*TRTPN*SEX | | M | 7 | 1 | |
| AVISITN*TRTPN*SEX | | F | 7 | 2 | |
| AVISITN*TRTPN*SEX | | M | 7 | 2 | |
| AVISITN*TRTPN*SEX | | F | 7 | 3 | |
| AVISITN*TRTPN*SEX | | M | 7 | 3 | |
| AVISITN*TRTPN*SEX | | F | 14 | 1 | |
| AVISITN*TRTPN*SEX | | M | 14 | 1 | |
| AVISITN*TRTPN*SEX | | F | 14 | 2 | |

CENTANAFADINE 17 OF 28 PROTOCOL 405-201-00013

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

-----

Parameter Code=AISRSTOT ------

#### The Mixed Procedure

Coefficients for 1 vs. 3 BY SEX AT DAY 42

| | Pooled | | Analysis | Planned | |
|-------------------|--------|-----|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | Sex | (N) | (N) | Row1 |
| AVISITN*TRTPN*SEX | | M | 14 | 2 | |
| AVISITN*TRTPN*SEX | | F | 14 | 3 | |
| AVISITN*TRTPN*SEX | | M | 14 | 3 | |
| AVISITN*TRTPN*SEX | | F | 21 | 1 | |
| AVISITN*TRTPN*SEX | | M | 21 | 1 | |
| AVISITN*TRTPN*SEX | | F | 21 | 2 | |
| AVISITN*TRTPN*SEX | | M | 21 | 2 | |
| AVISITN*TRTPN*SEX | | F | 21 | 3 | |
| AVISITN*TRTPN*SEX | | M | 21 | 3 | |
| AVISITN*TRTPN*SEX | | F | 28 | 1 | |
| AVISITN*TRTPN*SEX | | M | 28 | 1 | |
| AVISITN*TRTPN*SEX | | F | 28 | 2 | |
| AVISITN*TRTPN*SEX | | M | 28 | 2 | |
| AVISITN*TRTPN*SEX | | F | 28 | 3 | |
| AVISITN*TRTPN*SEX | | M | 28 | 3 | |
| AVISITN*TRTPN*SEX | | F | 35 | 1 | |
| AVISITN*TRTPN*SEX | | M | 35 | 1 | |
| AVISITN*TRTPN*SEX | | F | 35 | 2 | |
| AVISITN*TRTPN*SEX | | M | 35 | 2 | |
CENTANAFADINE 18 OF 28 PROTOCOL 405-201-00013

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

Parameter Code=AISRSTOT ------

#### The Mixed Procedure

Coefficients for 1 vs. 3 BY SEX AT DAY 42

| | Pooled<br>Center | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|
| Effect | Number | Sex | (N) | (N) | Row1 |
| AVISITN*TRTPN*SEX | | F | 35 | 3 | |
| AVISITN*TRTPN*SEX | | M | 35 | 3 | |
| AVISITN*TRTPN*SEX | | F | 42 | 1 | 1 |
| AVISITN*TRTPN*SEX | | M | 42 | 1 | -1 |
| AVISITN*TRTPN*SEX | | F | 42 | 2 | |
| AVISITN*TRTPN*SEX | | M | 42 | 2 | |
| AVISITN*TRTPN*SEX | | F | 42 | 3 | -1 |
| AVISITN*TRTPN*SEX | | M | 42 | 3 | 1 |
| BASE*AVISITN | | | 7 | | |
| BASE*AVISITN | | | 14 | | |
| BASE*AVISITN | | | 21 | | |
| BASE*AVISITN | | | 28 | | |
| BASE*AVISITN | | | 35 | | |
| BASE*AVISITN | | | 42 | | |

CENTANAFADINE 19 OF 28 PROTOCOL 405-201-00013

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Coefficients for 2 vs. 3 BY SEX AT DAY 42

| | Pooled | | Analysis | Planned | |
|-----------|--------|-----|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | Sex | (N) | (N) | Row1 |
| T | | | | | |
| Intercept | | | | | |
| POOLCNTR | | | | | |

CENTANAFADINE 20 OF 28 PROTOCOL 405-201-00013

 $$\operatorname{\mathtt{STAT-3.1}}$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42

(Efficacy Sample)

The Mixed Procedure

Coefficients for 2 vs. 3 BY SEX AT DAY 42

| Effect | Pooled<br>Center<br>Number | Sex | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|
| POOLCNTR<br>POOLCNTR | | | | | |
| POOLCNTR<br>POOLCNTR | | | | | |
| POOLCNTR<br>POOLCNTR | | | | | |
| POOLCNTR | | | | | |
| POOLCNTR<br>POOLCNTR | | | | | |
| POOLCNTR | | | | | |
| POOLCNTR<br>POOLCNTR | | | | | |
| POOLCNTR<br>POOLCNTR | | | | | |
| POOLCNTR | | | | | |
| POOLCNTR<br>POOLCNTR | | | | | |
| POOLCNTR<br>POOLCNTR | | | | | |
| FOOLCNIK | | | | | |

CENTANAFADINE 21 OF 28 PROTOCOL 405-201-00013

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

Parameter Code=AISRSTOT ------

# The Mixed Procedure

Coefficients for 2 vs. 3 BY SEX AT DAY 42

| | Pooled<br>Center | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|
| Effect | Number | Sex | (N) | (N) | Row1 |
| POOLCNTR | | | | | |
| AVISITN | | | 7 | | |
| AVISITN | | | 14 | | |
| AVISITN | | | 21 | | |
| AVISITN | | | 28 | | |
| AVISITN | | | 35 | | |
| AVISITN | | | 42 | | |
| TRTPN | | | | 1 | |
| TRTPN | | | | 2 | |
| TRTPN | | | | 3 | |
| AVISITN*TRTPN | | | 7 | 1 | |
| AVISITN*TRTPN | | | 7 | 2 | |
| AVISITN*TRTPN | | | 7 | 3 | |
| AVISITN*TRTPN | | | 14 | 1 | |
| AVISITN*TRTPN | | | 14 | 2 | |
| AVISITN*TRTPN | | | 14 | 3 | |
| AVISITN*TRTPN | | | 21 | 1 | |
| AVISITN*TRTPN | | | 21 | 2 | |
| AVISITN*TRTPN | | | 21 | 3 | |


CENTANAFADINE 22 OF 28

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

Parameter Code=AISRSTOT ------

The Mixed Procedure

Coefficients for 2 vs. 3 BY SEX AT DAY 42

| Pooled | | Analysis | Planned | |
|---|---|---|---|---|
| Center | | Visit | Treatment | |
| Number | Sex | (N) | (N) | Row1 |
| | | 28 | 1 | |
| | | 28 | 2 | |
| | | 28 | 3 | |
| | | 35 | 1 | |
| | | 35 | 2 | |
| | | 35 | 3 | |
| | | 42 | 1 | |
| | | 42 | 2 | |
| | | 42 | 3 | |
| | F | | | |
| | M | | | |
| | F | 7 | | |
| | M | 7 | | |
| | F | 14 | | |
| | M | 14 | | |
| | F | 21 | | |
| | M | 21 | | |
| | F | 28 | | |
| | M | 28 | | |
| | Center | Center<br>Number Sex | Center Visit Number Sex (N) 28 28 28 28 35 35 35 42 42 42 7 42 42 42 42 F M F 7 M 7 F 14 M 14 F 21 M 21 F 28 | Center Number Sex (N) (N) (N) 28 1 28 2 28 3 35 1 35 2 35 3 42 1 42 2 42 3 F M F 7 M 7 F 14 M 14 F 21 M 21 F 28 |

CENTANAFADINE 23 OF 28


# STAT-3.1 MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

# The Mixed Procedure

Coefficients for 2 vs. 3 BY SEX AT DAY 42

| | Pooled<br>Center | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|
| Effect | Number | Sex | (N) | (N) | Row1 |
| AVISITN*SEX | | F | 35 | | |
| AVISITN*SEX | | M | 35 | | |
| AVISITN*SEX | | F | 42 | | |
| AVISITN*SEX | | M | 42 | | |
| TRTPN*SEX | | F | | 1 | |
| TRTPN*SEX | | M | | 1 | |
| TRTPN*SEX | | F | | 2 | 1 |
| TRTPN*SEX | | M | | 2 | -1 |
| TRTPN*SEX | | F | | 3 | -1 |
| TRTPN*SEX | | M | | 3 | 1 |
| AVISITN*TRTPN*SEX | | F | 7 | 1 | |
| AVISITN*TRTPN*SEX | | M | 7 | 1 | |
| AVISITN*TRTPN*SEX | | F | 7 | 2 | |
| AVISITN*TRTPN*SEX | | M | 7 | 2 | |
| AVISITN*TRTPN*SEX | | F | 7 | 3 | |
| AVISITN*TRTPN*SEX | | M | 7 | 3 | |
| AVISITN*TRTPN*SEX | | F | 14 | 1 | |
| AVISITN*TRTPN*SEX | | M | 14 | 1 | |
| AVISITN*TRTPN*SEX | | F | 14 | 2 | |

CENTANAFADINE 24 OF 28 PROTOCOL 405-201-00013

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

-----

Parameter Code=AISRSTOT ------

#### The Mixed Procedure

Coefficients for 2 vs. 3 BY SEX AT DAY 42

| Pooled | | Analysis | Planned | |
|---|---|---|---|---|
| Center | | Visit | Treatment | |
| Number | Sex | (N) | (N) | Row1 |
| | M | 14 | | |
| | F | 14 | | |
| | M | 14 | 3 | |
| | F | 21 | 1 | |
| | M | 21 | 1 | |
| | F | 21 | 2 | |
| | M | 21 | 2 | |
| | F | 21 | 3 | |
| | M | 21 | 3 | |
| | F | 28 | 1 | |
| | M | 28 | 1 | |
| | F | 28 | 2 | |
| | M | 28 | 2 | |
| | F | 28 | | |
| | M | 28 | 3 | |
| | F | 35 | 1 | |
| | M | 35 | 1 | |
| | F | 35 | 2 | |
| | M | 35 | 2 | |
| | Center | Center<br>Number Sex M F M | Center Visit Number Sex (N) M 14 F 14 M 14 F 21 M 21 F 21 M 21 F 21 M 21 F 22 M 22 F 22 M 28 F 28 M 28 F 28 M 28 F 28 M 28 F 28 M 28 F 35 M 35 F 35 | Center Number Sex (N) (N) (N) M 14 2 F 14 3 M 14 3 F 21 1 M 21 1 F 21 2 M 21 2 F 21 3 M 21 2 F 21 3 M 21 2 F 22 5 M 22 5 F 22 8 1 M 28 2 F 28 3 M 28 2 F 28 3 M 28 3 F 35 1 M 35 1 F 35 2 |

CENTANAFADINE 25 OF 28 PROTOCOL 405-201-00013

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

-----

#### The Mixed Procedure

Coefficients for 2 vs. 3 BY SEX AT DAY 42

| | Pooled | | Analysis | Planned | |
|-------------------|--------|-----|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | Sex | (N) | (N) | Row1 |
| AVISITN*TRTPN*SEX | | F | 35 | 3 | |
| AVISITN*TRTPN*SEX | | M | 35 | 3 | |
| AVISITN*TRTPN*SEX | | F | 42 | 1 | |
| AVISITN*TRTPN*SEX | | M | 42 | 1 | |
| AVISITN*TRTPN*SEX | | F | 42 | 2 | 1 |
| AVISITN*TRTPN*SEX | | M | 42 | 2 | -1 |
| AVISITN*TRTPN*SEX | | F | 42 | 3 | -1 |
| AVISITN*TRTPN*SEX | | M | 42 | 3 | 1 |
| BASE*AVISITN | | | 7 | | |
| BASE*AVISITN | | | 14 | | |
| BASE*AVISITN | | | 21 | | |
| BASE*AVISITN | | | 28 | | |
| BASE*AVISITN | | | 35 | | |
| BASE*AVISITN | | | 42 | | |

CENTANAFADINE 26 OF 28 PROTOCOL 405-201-00013

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 $(\tt Efficacy\ Sample)$

------

# The Mixed Procedure

# Estimates

| | | Standard | | | |
|--------------------------|----------|----------|-----|---------|---------|
| Label | Estimate | Error | DF | t Value | Pr > t |
| 1 vs. 3 BY SEX AT DAY 42 | 0.008634 | 2.7164 | 405 | 0.00 | 0.9975 |
| 2 vs. 3 BY SEX AT DAY 42 | 1.0223 | 2.7042 | 403 | 0.38 | 0.7056 |

# Least Squares Means

| | | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN*SEX | F | 7 | 1 | -5.5125 | 0.9145 | 398 | -6.03 | <.0001 | 0.05 | -7.3104 | -3.7146 |
| AVISITN*TRTPN*SEX | M | 7 | 1 | -5.4466 | 0.9030 | 402 | -6.03 | <.0001 | 0.05 | -7.2219 | -3.6713 |
| AVISITN*TRTPN*SEX | F | 7 | 2 | -3.7780 | 0.9336 | 400 | -4.05 | <.0001 | 0.05 | -5.6133 | -1.9427 |
| AVISITN*TRTPN*SEX | M | 7 | 2 | -4.3169 | 0.9075 | 402 | -4.76 | <.0001 | 0.05 | -6.1010 | -2.5329 |
| AVISITN*TRTPN*SEX | F | 7 | 3 | -5.2355 | 0.9157 | 396 | -5.72 | <.0001 | 0.05 | -7.0357 | -3.4352 |
| AVISITN*TRTPN*SEX | M | 7 | 3 | -3.0663 | 0.9328 | 400 | -3.29 | 0.0011 | 0.05 | -4.9001 | -1.2324 |
| AVISITN*TRTPN*SEX | F | 14 | 1 | -7.9530 | 1.0866 | 431 | -7.32 | <.0001 | 0.05 | -10.0887 | -5.8173 |
| AVISITN*TRTPN*SEX | M | 14 | 1 | -6.9443 | 1.0453 | 415 | -6.64 | <.0001 | 0.05 | -8.9991 | -4.8895 |
| AVISITN*TRTPN*SEX | F | 14 | 2 | -6.6749 | 1.0980 | 431 | -6.08 | <.0001 | 0.05 | -8.8330 | -4.5169 |
| AVISITN*TRTPN*SEX | M | 14 | 2 | -6.7586 | 1.0477 | 416 | -6.45 | <.0001 | 0.05 | -8.8180 | -4.6993 |

CENTANAFADINE 27 OF 28


# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

### The Mixed Procedure

# Least Squares Means

| | | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Visit | Treatment | | Standard | | | | | | |
| Effect | Sex | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN*SEX | F | 14 | 3 | -7.0864 | 1.0693 | 422 | -6.63 | <.0001 | 0.05 | -9.1883 | -4.9846 |
| AVISITN*TRTPN*SEX | M | 14 | 3 | -5.8234 | 1.0854 | 422 | -5.37 | <.0001 | 0.05 | -7.9569 | -3.6899 |
| AVISITN*TRTPN*SEX | F | 21 | 1 | -8.8044 | 1.1479 | 418 | -7.67 | <.0001 | 0.05 | -11.0608 | -6.5480 |
| AVISITN*TRTPN*SEX | M | 21 | 1 | -8.1444 | 1.1330 | 432 | -7.19 | <.0001 | 0.05 | -10.3713 | -5.9176 |
| AVISITN*TRTPN*SEX | F | 21 | 2 | -8.2616 | 1.1716 | 434 | -7.05 | <.0001 | 0.05 | -10.5644 | -5.9589 |
| AVISITN*TRTPN*SEX | M | 21 | 2 | -8.3214 | 1.1086 | 410 | -7.51 | <.0001 | 0.05 | -10.5007 | -6.1422 |
| AVISITN*TRTPN*SEX | F | 21 | 3 | -6.5243 | 1.1292 | 415 | -5.78 | <.0001 | 0.05 | -8.7439 | -4.3047 |
| AVISITN*TRTPN*SEX | M | 21 | 3 | -6.5280 | 1.1518 | 416 | -5.67 | <.0001 | 0.05 | -8.7920 | -4.2640 |
| AVISITN*TRTPN*SEX | F | 28 | 1 | -9.7129 | 1.3221 | 429 | -7.35 | <.0001 | 0.05 | -12.3114 | -7.1143 |
| AVISITN*TRTPN*SEX | M | 28 | 1 | -9.5818 | 1.2976 | 433 | -7.38 | <.0001 | 0.05 | -12.1321 | -7.0315 |
| AVISITN*TRTPN*SEX | F | 28 | 2 | -8.5617 | 1.3340 | 435 | -6.42 | <.0001 | 0.05 | -11.1835 | -5.9398 |
| AVISITN*TRTPN*SEX | M | 28 | 2 | -10.5997 | 1.2679 | 423 | -8.36 | <.0001 | 0.05 | -13.0919 | -8.1075 |
| AVISITN*TRTPN*SEX | F | 28 | 3 | -5.7966 | 1.2745 | 413 | -4.55 | <.0001 | 0.05 | -8.3020 | -3.2913 |
| AVISITN*TRTPN*SEX | M | 28 | 3 | -6.8225 | 1.3154 | 423 | -5.19 | <.0001 | 0.05 | -9.4081 | -4.2369 |
| AVISITN*TRTPN*SEX | F | 35 | 1 | -10.3738 | 1.3557 | 421 | -7.65 | <.0001 | 0.05 | -13.0386 | -7.7090 |
| AVISITN*TRTPN*SEX | M | 35 | 1 | -10.1739 | 1.3368 | 429 | -7.61 | <.0001 | 0.05 | -12.8014 | -7.5463 |
| AVISITN*TRTPN*SEX | F | 35 | 2 | -10.6335 | 1.3813 | 440 | -7.70 | <.0001 | 0.05 | -13.3484 | -7.9187 |
| AVISITN*TRTPN*SEX | M | 35 | 2 | -10.7772 | 1.3026 | 417 | -8.27 | <.0001 | 0.05 | -13.3378 | -8.2166 |
| AVISITN*TRTPN*SEX | F | 35 | 3 | -7.3509 | 1.3131 | 412 | -5.60 | <.0001 | 0.05 | -9.9321 | -4.7697 |


CENTANAFADINE 28 OF 28

STAT-3.1

MMRM Output for Test on Treatment by Sex Interaction at Day 42

(Efficacy Sample)

------

The Mixed Procedure

Least Squares Means

| | | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN*SEX | М | 35 | 3 | -7.0325 | 1.3507 | 417 | -5.21 | <.0001 | 0.05 | -9.6875 | -4.3774 |
| AVISITN*TRTPN*SEX | F | 42 | 1 | -10.3674 | 1.4025 | 421 | -7.39 | <.0001 | 0.05 | -13.1242 | -7.6106 |
| AVISITN*TRTPN*SEX | M | 42 | 1 | -9.9078 | 1.3872 | 433 | -7.14 | <.0001 | 0.05 | -12.6343 | -7.1814 |
| AVISITN*TRTPN*SEX | F | 42 | 2 | -9.4500 | 1.4201 | 434 | -6.65 | <.0001 | 0.05 | -12.2411 | -6.6589 |
| AVISITN*TRTPN*SEX | M | 42 | 2 | -10.0041 | 1.3380 | 410 | -7.48 | <.0001 | 0.05 | -12.6344 | -7.3738 |
| AVISITN*TRTPN*SEX | F | 42 | 3 | -7.2141 | 1.3547 | 411 | -5.33 | <.0001 | 0.05 | -9.8771 | -4.5510 |
| AVISITN*TRTPN*SEX | M | 42 | 3 | -6.7459 | 1.3983 | 419 | -4.82 | <.0001 | 0.05 | -9.4945 | -3.9972 |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction at Day 42

(Efficacy Sample)

\_\_\_\_\_

# The Mixed Procedure

#### Model Information

Data Set WORK.INDATA Dependent Variable CHG Covariance Structure Unstructured Subject Effect SUBJID Estimation Method REML Residual Variance Method None Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger

#### Class Level Information

| Class | Levels | Values |
|------------------------------|--------------|---------------------------|
| AVISITN<br>TRTPN<br>POOLCNTR | 6<br>3<br>38 | 7 14 21 28 35 42<br>1 2 3 |

CENTANAFADINE
2 OF 28

 $$\operatorname{STAT-3.2}$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

......

The Mixed Procedure

Class Level Information

Class Levels Values

SUBJID 438




 $$\operatorname{STAT-3.2}$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

......

The Mixed Procedure



CENTANAFADINE
4 OF 28

 $$\operatorname{STAT-3.2}$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

......

The Mixed Procedure




 $$\operatorname{STAT-3.2}$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

......

The Mixed Procedure




 $$\operatorname{STAT-3.2}$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

......

The Mixed Procedure




 $$\operatorname{STAT-3.2}$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

......

The Mixed Procedure



| CENTANAFADINE | 8 OF 28 |
|------------------------|---------|

STAT-3.2

MMRM Output for Test on Treatment by Race Interaction at Day 42  $$({\tt Efficacy\ Sample})$$ 

The Mixed Procedure

Class Level Information

Class Levels Values

RACEGRP 2 All Other Races White

Dimensions

Covariance Parameters 21
Columns in X 128
Columns in Z 0
Subjects 438
Max Obs per Subject 6

Number of Observations

Number of Observations Read 2292
Number of Observations Used 2292
Number of Observations Not Used 0


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction at Day 42  $\,$  (Efficacy Sample)

......

The Mixed Procedure

Iteration History

| Criterion | -2 Res Log Like | Evaluations | Iteration |
|------------|-------------------|-------------|-----------|
| | 16457.56446856 | 1 | 0 |
| 0.00015243 | 14194.15343914 | 2 | 1 |
| 0.00000121 | 14193.34064068 | 1 | 2 |
| 0.0000000 | 1/11/93 33///7925 | 1 | 3 |

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|--------------------|------------------|--------------------|
| UN(1,1)<br>UN(2,1) | SUBJID<br>SUBJID | 52.6274<br>40.2457 |
| UN(2,2)<br>UN(3,1) | SUBJID<br>SUBJID | 72.4424 |
| UN(3,2) | SUBJID | 62.1116 |
| UN(3,3)<br>UN(4,1) | SUBJID<br>SUBJID | 81.4367<br>37.1824 |
| UN (4,1) | SUBJID | 62.6074 |


CENTANAFADINE 10 OF 28

 $$\operatorname{STAT-3.2}$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

# The Mixed Procedure

#### Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(4,3) | SUBJID | 77.2494 |
| UN(4,4) | SUBJID | 105.45 |
| UN(5,1) | SUBJID | 38.0335 |
| UN(5,2) | SUBJID | 63.1832 |
| UN(5,3) | SUBJID | 80.6593 |
| UN(5,4) | SUBJID | 95.9188 |
| UN(5,5) | SUBJID | 110.56 |
| UN(6,1) | SUBJID | 38.5893 |
| UN(6,2) | SUBJID | 64.3249 |
| UN(6,3) | SUBJID | 78.5308 |
| UN(6,4) | SUBJID | 96.2386 |
| UN(6,5) | SUBJID | 99.4627 |
| UN(6,6) | SUBJID | 117.27 |

# Fit Statistics

| -2 Res Log Likelihood | 14193.3 |
|--------------------------|---------|
| AIC (Smaller is Better) | 14235.3 |
| AICC (Smaller is Better) | 14235.8 |
| BIC (Smaller is Better) | 14321.1 |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction at Day 42  $\,$  (Efficacy Sample)

The Mixed Procedure

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 20 2264.23 <.0001

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------------------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| POOLCNTR | 37 | 393 | 2.25 | <.0001 |
| AVISITN | 5 | 377 | 1.96 | 0.0837 |
| TRTPN | 2 | 402 | 2.69 | 0.0690 |
| AVISITN*TRTPN | 10 | 559 | 1.68 | 0.0821 |
| RACEGRP | 1 | 415 | 1.14 | 0.2857 |
| AVISITN*RACEGRP | 5 | 376 | 1.25 | 0.2836 |
| TRTPN*RACEGRP | 2 | 410 | 0.44 | 0.6436 |
| AVISIT*TRTPN*RACEGRP | 10 | 559 | 1.01 | 0.4349 |
| BASE*AVISITN | 6 | 402 | 2.39 | 0.0280 |


 $$\tt STAT-3.2$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Coefficients for 1 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|-----------|--------|---------|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| Intercept | | | | | |
| POOLCNTR | | | | | |


 $$\operatorname{STAT-3.2}$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

......

The Mixed Procedure

Coefficients for 1 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|-----------|--------|---------|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| POOLCNTR | | | | | |
| 100101111 | | | | | |


CENTANAFADINE 14 OF 28

 $$\operatorname{STAT-3.2}$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

......

#### The Mixed Procedure

# Coefficients for 1 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|---------------|--------|---------|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| POOLCNTR | | | | | |
| AVISITN | | | 7 | | |
| AVISITN | | | 14 | | |
| AVISITN | | | 21 | | |
| AVISITN | | | 28 | | |
| AVISITN | | | 35 | | |
| AVISITN | | | 42 | | |
| TRTPN | | | | 1 | |
| TRTPN | | | | 2 | |
| TRTPN | | | | 3 | |
| AVISITN*TRTPN | | | 7 | 1 | |
| AVISITN*TRTPN | | | 7 | 2 | |
| AVISITN*TRTPN | | | 7 | 3 | |
| AVISITN*TRTPN | | | 14 | 1 | |
| AVISITN*TRTPN | | | 14 | 2 | |
| AVISITN*TRTPN | | | 14 | 3 | |
| AVISITN*TRTPN | | | 21 | 1 | |
| AVISITN*TRTPN | | | 21 | 2 | |
| AVISITN*TRTPN | | | 21 | 3 | |

CENTANAFADINE 15 OF 28 PROTOCOL 405-201-00013

 $$\operatorname{STAT-3.2}$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

......

Parameter Code=AISRSTOT -----

#### The Mixed Procedure

# Coefficients for 1 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|-----------------|--------|-----------------|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| AVISITN*TRTPN | | | 28 | 1 | |
| AVISITN*TRTPN | | | 28 | 2 | |
| AVISITN*TRTPN | | | 28 | 3 | |
| AVISITN*TRTPN | | | 35 | 1 | |
| AVISITN*TRTPN | | | 35 | 2 | |
| AVISITN*TRTPN | | | 35 | 3 | |
| AVISITN*TRTPN | | | 42 | 1 | |
| AVISITN*TRTPN | | | 42 | 2 | |
| AVISITN*TRTPN | | | 42 | 3 | |
| RACEGRP | | All Other Races | | | |
| RACEGRP | | White | | | |
| AVISITN*RACEGRP | | All Other Races | 7 | | |
| AVISITN*RACEGRP | | White | 7 | | |
| AVISITN*RACEGRP | | All Other Races | 14 | | |
| AVISITN*RACEGRP | | White | 14 | | |
| AVISITN*RACEGRP | | All Other Races | 21 | | |
| AVISITN*RACEGRP | | White | 21 | | |
| AVISITN*RACEGRP | | All Other Races | 28 | | |
| AVISITN*RACEGRP | | White | 28 | | |


# $$\operatorname{\mathtt{STAT-3.2}}$$ MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

\_\_\_\_\_

Parameter Code=AISRSTOT ------

# The Mixed Procedure

# Coefficients for 1 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | | Analysis | Planned | |
|---|---|---|---|---|---|---|
| | Center | | | Visit | Treatment | |
| Effect | Number | RACEGRP | | (N) | (N) | Row1 |
| AVISITN*RACEGRP | | All Other Ra | | 35 | | |
| AVISITN*RACEGRP | | White | | 35 | | |
| AVISITN*RACEGRP | | All Other Ra | ces | 42 | | |
| AVISITN*RACEGRP | | White | | 42 | | |
| TRTPN*RACEGRP | | All Other Ra | ces | | 1 | 1 |
| TRTPN*RACEGRP | | White | | | 1 | -1 |
| TRTPN*RACEGRP | | All Other Ra | ces | | 2 | |
| TRTPN*RACEGRP | | White | | | 2 | |
| TRTPN*RACEGRP | | All Other Ra | ces | | 3 | -1 |
| TRTPN*RACEGRP | | White | | | 3 | 1 |
| AVISIT*TRTPN*RACEGRP | | All Other Ra | ces | 7 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | | 7 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Ra | ces | 7 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | | 7 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Ra | ces | 7 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | | 7 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Ra | ces | 14 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | | 14 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Ra | ces | 14 | 2 | |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction at Day 42  $$({\tt Efficacy\ Sample})$$ 

The Mixed Procedure

Coefficients for 1 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|---|---|---|---|---|---|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| AVISIT*TRTPN*RACEGRP | | White | 14 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 14 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 14 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 21 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 21 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 21 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 21 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 21 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 21 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 28 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 28 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 28 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 28 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 28 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 28 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 35 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 35 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 35 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 35 | 2 | |


 $$\operatorname{STAT-3.2}$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Coefficients for 1 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|---|---|---|---|---|---|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 35 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 35 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 42 | 1 | 1 |
| AVISIT*TRTPN*RACEGRP | | White | 42 | 1 | -1 |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 42 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 42 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 42 | 3 | -1 |
| AVISIT*TRTPN*RACEGRP | | White | 42 | 3 | 1 |
| BASE*AVISITN | | | 7 | | |
| BASE*AVISITN | | | 14 | | |
| BASE*AVISITN | | | 21 | | |
| BASE*AVISITN | | | 28 | | |
| BASE*AVISITN | | | 35 | | |
| BASE*AVISITN | | | 42 | | |


 $$\operatorname{\mathtt{STAT-3.2}}$$  MMRM Output for Test on Treatment by Race Interaction at Day 42

(Efficacy Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for 2 vs. 3 BY RACEGRP AT DAY 42

| | | Pooled | | Analysis | Planned | |
|----|------------|--------|---------|----------|-----------|------|
| | | Center | | Visit | Treatment | |
| Εf | fect | Number | RACEGRP | (N) | (N) | Row1 |
| Tr | ntercept . | | | | | |
| | OOLCNTR | | | | | |
| | OOLCNTR | | | | | |
| | OOLCNTR | | | | | |
| PC | OOLCNTR | | | | | |
| | OOLCNTR | | | | | |
| | OOLCNTR | | | | | |
| PC | OTCNIV | | | | | |


 $$\operatorname{STAT-3.2}$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

......

The Mixed Procedure

Coefficients for 2 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|----------|------------------|---------|--------------|---------------|------|
| Effect | Center<br>Number | RACEGRP | Visit<br>(N) | Treatment (N) | Row1 |
| POOLCNTR | | | | | |


CENTANAFADINE 21 OF 28

 $$\operatorname{STAT-3.2}$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

......

Parameter Code=AISRSTOT ------

# The Mixed Procedure

# Coefficients for 2 vs. 3 BY RACEGRP AT DAY 42

| Pooled Analysis P | |
|---------------------------|----------|
| Center Visit T | reatment |
| Effect Number RACEGRP (N) | N) Row1 |
| POOLCNTR | |
| AVISITN 7 | |
| AVISITN 14 | |
| AVISITN 21 | |
| AVISITN 28 | |
| AVISITN 35 | |
| AVISITN 42 | |
| TRTPN 1 | |
| TRTPN 2 | |
| TRTPN 3 | |
| AVISITN*TRTPN 7 1 | |
| AVISITN*TRTPN 7 2 | |
| AVISITN*TRTPN 7 3 | |
| AVISITN*TRTPN 14 1 | |
| AVISITN*TRTPN 14 2 | |
| AVISITN*TRTPN 14 3 | |
| AVISITN*TRTPN 21 1 | |
| AVISITN*TRTPN 21 2 | |
| AVISITN*TRTPN 21 3 | |

CENTANAFADINE 22 OF 28 PROTOCOL 405-201-00013

STAT-3.2

MMRM Output for Test on Treatment by Race Interaction at Day 42  $$({\tt Efficacy\ Sample})$$ 

-----

The Mixed Procedure

Coefficients for 2 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|-----------------|--------|-----------------|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| | | | 00 | | |
| AVISITN*TRTPN | | | 28 | 1 | |
| AVISITN*TRTPN | | | 28 | 2 | |
| AVISITN*TRTPN | | | 28 | 3 | |
| AVISITN*TRTPN | | | 35 | 1 | |
| AVISITN*TRTPN | | | 35 | 2 | |
| AVISITN*TRTPN | | | 35 | 3 | |
| AVISITN*TRTPN | | | 42 | 1 | |
| AVISITN*TRTPN | | | 42 | 2 | |
| AVISITN*TRTPN | | | 42 | 3 | |
| RACEGRP | | All Other Races | | | |
| RACEGRP | | White | | | |
| AVISITN*RACEGRP | | All Other Races | 7 | | |
| AVISITN*RACEGRP | | White | 7 | | |
| AVISITN*RACEGRP | | All Other Races | 14 | | |
| AVISITN*RACEGRP | | White | 14 | | |
| AVISITN*RACEGRP | | All Other Races | 21 | | |
| AVISITN*RACEGRP | | White | 21 | | |
| AVISITN*RACEGRP | | All Other Races | 28 | | |
| AVISITN*RACEGRP | | White | 28 | | |

CENTANAFADINE 23 OF 28 PROTOCOL 405-201-00013

STAT-3.2

MMRM Output for Test on Treatment by Race Interaction at Day 42  $$({\tt Efficacy\ Sample})$$ 

The Mixed Procedure

Coefficients for 2 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|---|---|---|---|---|---|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| AVISITN*RACEGRP | | All Other Races | 35 | | |
| AVISITN*RACEGRP | | White | 35 | | |
| AVISITN*RACEGRP | | All Other Races | 42 | | |
| AVISITN*RACEGRP | | White | 42 | | |
| TRTPN*RACEGRP | | All Other Races | | 1 | |
| TRTPN*RACEGRP | | White | | 1 | |
| TRTPN*RACEGRP | | All Other Races | | 2 | 1 |
| TRTPN*RACEGRP | | White | | 2 | -1 |
| TRTPN*RACEGRP | | All Other Races | | 3 | -1 |
| TRTPN*RACEGRP | | White | | 3 | 1 |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 7 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 7 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 7 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 7 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 7 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 7 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 14 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 14 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 14 | 2 | |

CENTANAFADINE 24 OF 28


 $$\operatorname{STAT-3.2}$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

Parameter Code=AISRSTOT ------

The Mixed Procedure

Coefficients for 2 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|---|---|---|---|---|---|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| AVISIT*TRTPN*RACEGRP | | White | 14 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 14 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 14 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 21 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 21 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 21 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 21 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 21 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 21 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 28 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 28 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 28 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 28 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 28 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 28 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 35 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 35 | 2 | |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction at Day 42  $$({\tt Efficacy\ Sample})$$ 

Parameter Code=AISRSTOT ------

The Mixed Procedure

Coefficients for 2 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|---|---|---|---|---|---|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 35 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 35 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 42 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 42 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 42 | 2 | 1 |
| AVISIT*TRTPN*RACEGRP | | White | 42 | 2 | -1 |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 42 | 3 | -1 |
| AVISIT*TRTPN*RACEGRP | | White | 42 | 3 | 1 |
| BASE*AVISITN | | | 7 | | |
| BASE*AVISITN | | | 14 | | |
| BASE*AVISITN | | | 21 | | |
| BASE*AVISITN | | | 28 | | |
| BASE*AVISITN | | | 35 | | |
| BASE*AVISITN | | | 42 | | |

# STAT-3.2 MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

# The Mixed Procedure

#### Estimates

| | | | | | | | | | Standard | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Lab | pel | | | | | | | Estimate | Error | DF | t Value | Pr > t |
| 1 v | 7S. | 3 | вч | RACEGRP | AT | DAY | 42 | -4.2107 | 3.6531 | 413 | -1.15 | 0.2497 |
| 2 v | 7S. | 3 | BY | RACEGRP | AΤ | DAY | 42 | -4.6414 | 3.5664 | 405 | -1.30 | 0.1939 |

# Least Squares Means

| | | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | RACEGRP | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISIT*TRTPN*RACEGRP | All Other Races | 7 | 1 | -5.4070 | 1.4741 | 402 | -3.67 | 0.0003 | 0.05 | -8.3049 | -2.5092 |
| AVISIT*TRTPN*RACEGRP | White | 7 | 1 | -5.5130 | 0.7191 | 401 | -7.67 | <.0001 | 0.05 | -6.9267 | -4.0993 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 7 | 2 | -5.5362 | 1.4286 | 409 | -3.88 | 0.0001 | 0.05 | -8.3446 | -2.7278 |
| AVISIT*TRTPN*RACEGRP | White | 7 | 2 | -3.6971 | 0.7401 | 399 | -5.00 | <.0001 | 0.05 | -5.1521 | -2.2421 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 7 | 3 | -4.4167 | 1.6472 | 402 | -2.68 | 0.0076 | 0.05 | -7.6548 | -1.1786 |
| AVISIT*TRTPN*RACEGRP | White | 7 | 3 | -4.1607 | 0.7267 | 399 | -5.73 | <.0001 | 0.05 | -5.5893 | -2.7320 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 14 | 1 | -9.1406 | 1.7282 | 425 | -5.29 | <.0001 | 0.05 | -12.5375 | -5.7437 |
| AVISIT*TRTPN*RACEGRP | White | 14 | 1 | -7.0447 | 0.8377 | 421 | -8.41 | <.0001 | 0.05 | -8.6913 | -5.3981 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 14 | 2 | -7.7555 | 1.6612 | 425 | -4.67 | <.0001 | 0.05 | -11.0208 | -4.4903 |
| AVISIT*TRTPN*RACEGRP | White | 14 | 2 | -6.4603 | 0.8573 | 427 | -7.54 | <.0001 | 0.05 | -8.1453 | -4.7753 |

CENTANAFADINE 27 OF 28 PROTOCOL 405-201-00013

# $$\tt STAT-3.2$$ MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

------

Parameter Code=AISRSTOT ------

# The Mixed Procedure

# Least Squares Means

| | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | Treatment | | Standard | | | | | | |
| RACEGRP | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| All Other Races | 14 | 3 | -6.8926 | 1.8839 | 401 | -3.66 | 0.0003 | 0.05 | -10.5961 | -3.1891 |
| White | 14 | 3 | -6.4045 | 0.8426 | 433 | -7.60 | <.0001 | 0.05 | -8.0607 | -4.7484 |
| All Other Races | 21 | 1 | -9.1324 | 1.8815 | 447 | -4.85 | <.0001 | 0.05 | -12.8302 | -5.4346 |
| White | 21 | 1 | -8.3083 | 0.8926 | 424 | -9.31 | <.0001 | 0.05 | -10.0626 | -6.5539 |
| All Other Races | 21 | 2 | -9.6889 | 1.7502 | 409 | -5.54 | <.0001 | 0.05 | -13.1294 | -6.2483 |
| White | 21 | 2 | -7.9419 | 0.9105 | 430 | -8.72 | <.0001 | 0.05 | -9.7315 | -6.1523 |
| All Other Races | 21 | 3 | -6.4777 | 2.0044 | 400 | -3.23 | 0.0013 | 0.05 | -10.4181 | -2.5374 |
| White | 21 | 3 | -6.5518 | 0.8889 | 429 | -7.37 | <.0001 | 0.05 | -8.2989 | -4.8047 |
| All Other Races | 28 | 1 | -11.3582 | 2.1608 | 444 | -5.26 | <.0001 | 0.05 | -15.6049 | -7.1116 |
| White | 28 | 1 | -9.2681 | 1.0250 | 433 | -9.04 | <.0001 | 0.05 | -11.2826 | -7.2535 |
| All Other Races | 28 | 2 | -12.7159 | 1.9930 | 408 | -6.38 | <.0001 | 0.05 | -16.6337 | -8.7982 |
| White | 28 | 2 | -8.7879 | 1.0386 | 442 | -8.46 | <.0001 | 0.05 | -10.8291 | -6.7467 |
| All Other Races | 28 | 3 | -5.5914 | 2.3069 | 414 | -2.42 | 0.0158 | 0.05 | -10.1261 | -1.0567 |
| White | 28 | 3 | -6.4036 | 1.0037 | 428 | -6.38 | <.0001 | 0.05 | -8.3764 | -4.4308 |
| All Other Races | 35 | 1 | -11.5318 | 2.2200 | 440 | -5.19 | <.0001 | 0.05 | -15.8948 | -7.1687 |
| White | 35 | 1 | -9.9860 | 1.0509 | 427 | -9.50 | <.0001 | 0.05 | -12.0515 | -7.9204 |
| All Other Races | 35 | 2 | -13.1394 | 2.0655 | 417 | -6.36 | <.0001 | 0.05 | -17.1995 | -9.0793 |
| White | 35 | 2 | -10.0665 | 1.0666 | 439 | -9.44 | <.0001 | 0.05 | -12.1627 | -7.9703 |
| All Other Races | 35 | 3 | -8.4240 | 2.3575 | 405 | -3.57 | 0.0004 | 0.05 | -13.0585 | -3.7896 |
| | All Other Races White | RACEGRP (N) All Other Races 14 White 14 All Other Races 21 White 21 All Other Races 21 White 21 All Other Races 21 White 21 All Other Races 21 White 21 All Other Races 28 White 28 All Other Races 28 White 28 All Other Races 28 White 28 All Other Races 28 White 28 All Other Races 35 White 35 All Other Races 35 White 35 White 35 White 35 | RACEGRP (N) (N) All Other Races 14 3 White 14 3 All Other Races 21 1 White 21 1 All Other Races 21 2 White 21 2 All Other Races 21 3 White 21 3 All Other Races 21 3 White 21 4 All Other Races 22 3 White 21 4 All Other Races 28 1 White 28 1 All Other Races 28 1 White 28 1 All Other Races 28 2 White 28 2 All Other Races 28 3 White 28 3 All Other Races 35 1 White 35 1 All Other Races 35 1 White 35 2 White 35 2 | RACEGRP (N) (N) Estimate All Other Races 14 3 -6.8926 White 14 3 -6.4045 All Other Races 21 1 -9.1324 White 21 1 -8.3083 All Other Races 21 2 -7.9419 White 21 2 -7.9419 All Other Races 21 3 -6.4777 White 21 3 -6.5518 All Other Races 28 1 -11.3582 White 28 1 -9.2681 All Other Races 28 2 -12.7159 White 28 2 -8.7879 All Other Races 28 3 -5.5914 White 28 3 -6.4036 All Other Races 35 1 -11.5318 White 35 1 -9.9860 All Other Races 35 1 -9.9860 All Other Races 35 2 -13.1394 White 35 2 -10.0665 | RACEGRP (N) Estimate Error All Other Races 14 3 -6.8926 1.8839 White 14 3 -6.4045 0.8426 All Other Races 21 1 -9.1324 1.8815 White 21 1 -8.3083 0.8926 All Other Races 21 2 -9.6889 1.7502 White 21 2 -7.9419 0.9105 All Other Races 21 3 -6.4777 2.0044 White 21 3 -6.5518 0.8889 All Other Races 28 1 -11.3582 2.1608 White 28 1 -9.2681 1.0250 All Other Races 28 2 -12.7159 1.9930 White 28 2 -8.7879 1.0386 All Other Races 28 3 -5.5914 2.3069 White 28 3 -6.4036 1.0037 All Other Races 35 1 -11.5318 2.2200 White 35 1 -9.9860 1.0509 All Other Races 35 1 -9.9860 1.0509 All Other Races 35 2 -13.1394 2.0665 White 35 2 -10.0665 1.0666 | RACEGRP (N) (N) Estimate Error DF All Other Races 14 3 -6.8926 1.8839 401 White 14 3 -6.4045 0.8426 433 All Other Races 21 1 -9.1324 1.8815 447 White 21 1 -8.3083 0.8926 424 All Other Races 21 2 -9.6889 1.7502 409 White 21 2 -7.9419 0.9105 430 All Other Races 21 3 -6.4777 2.0044 400 White 21 3 -6.5518 0.8889 429 All Other Races 28 1 -11.3582 2.1608 444 White 28 1 -9.2681 1.0250 433 All Other Races 28 2 -12.7159 1.9930 408 White 28 2 -8.7879 1.0386 442 All Other Races 28 3 -5.5914 2.3069 414 White 28 3 -6.4036 1.0037 428 All Other Races 35 1 -11.5318 2.2200 440 White 35 1 -9.9860 1.0509 427 All Other Races 35 2 -13.1394 2.0655 417 White 35 2 -13.1394 2.0655 417 White 35 2 -13.1394 2.0655 417 | RACEGRP (N) (N) Estimate Error DF t Value All Other Races 14 3 -6.8926 1.8839 401 -3.66 White 14 3 -6.4045 0.8426 433 -7.60 All Other Races 21 1 -9.1324 1.8815 447 -4.85 White 21 1 -8.3083 0.8926 424 -9.31 All Other Races 21 2 -9.6889 1.7502 409 -5.54 White 21 2 -7.9419 0.9105 430 -8.72 All Other Races 21 3 -6.4777 2.0044 400 -3.23 White 21 3 -6.5518 0.8889 429 -7.37 All Other Races 28 1 -11.3582 2.1608 444 -5.26 White 28 1 -9.2681 1.0250 433 -9.04 All Other Races 28 2 -12.7159 1.9930 408 -6.38 White 28 2 -8.7879 1.0386 442 -8.46 All Other Races 28 3 -5.5914 2.3069 414 -2.42 White 28 3 -6.4036 1.0037 428 -6.38 All Other Races 35 1 -11.5318 2.2200 440 -5.19 White 35 1 -9.9860 1.0509 427 -9.50 White 35 2 -13.1394 2.0655 417 -6.36 White 35 2 -13.1394 2.0655 417 -6.36 White 35 2 -13.1394 2.0655 417 -6.36 | RACEGRP (N) (N) Estimate Error DF t Value Pr > t All Other Races 14 3 -6.8926 1.8839 401 -3.66 0.0003 White 14 3 -6.4045 0.8426 433 -7.60 <.0001 All Other Races 21 1 -9.1324 1.8815 447 -4.85 <.0001 White 21 1 -8.3083 0.8926 424 -9.31 <.0001 All Other Races 21 2 -9.6889 1.7502 409 -5.54 <.0001 White 21 2 -7.9419 0.9105 430 -8.72 <.0001 White 21 3 -6.4777 2.0044 400 -3.23 0.0013 White 21 3 -6.5518 0.8889 429 -7.37 <.0001 All Other Races 28 1 -11.3582 2.1608 444 -5.26 <.0001 White 28 1 -9.2681 1.0250 433 -9.04 <.0001 White 28 1 -9.2681 1.0250 433 -9.04 <.0001 All Other Races 28 2 -12.7159 1.9930 408 -6.38 <.0001 White 28 2 -8.7879 1.0386 442 -8.46 <.0001 All Other Races 28 3 -5.5914 2.3069 414 -2.42 0.0158 White 28 3 -6.4036 1.0037 428 -6.38 <.0001 All Other Races 35 1 -11.5318 2.2200 440 -5.19 <.0001 All Other Races 35 1 -11.5318 2.2200 440 -5.19 <.0001 All Other Races 35 2 -13.1394 2.0655 417 -6.36 <.0001 White 35 2 -13.1394 2.0655 417 -6.36 <.0001 White 35 2 -10.0665 1.0666 439 -9.44 <.0001 | RACEGRP (N) (N) Estimate Error DF t Value Pr > t Alpha All Other Races 14 3 -6.8926 1.8839 401 -3.66 0.0003 0.05 White 14 3 -6.4045 0.8426 433 -7.60 <.0001 0.05 All Other Races 21 1 -9.1324 1.8815 447 -4.85 <.0001 0.05 White 21 1 -8.3083 0.8926 424 -9.31 <.0001 0.05 All Other Races 21 2 -9.6889 1.7502 409 -5.54 <.0001 0.05 White 21 2 -7.9419 0.9105 430 -8.72 <.0001 0.05 White 21 3 -6.4777 2.0044 400 -3.23 0.0013 0.05 White 21 3 -6.5518 0.8889 429 -7.37 <.0001 0.05 White 21 3 -6.5518 0.8889 429 -7.37 <.0001 0.05 White 21 3 -6.5518 0.8889 429 -7.37 <.0001 0.05 White 28 1 -9.2681 1.0250 433 -9.04 <.0001 0.05 White 28 1 -9.2681 1.0250 433 -9.04 <.0001 0.05 White 28 2 -8.7879 1.0386 442 -8.46 <.0001 0.05 White 28 2 -8.7879 1.0386 442 -8.46 <.0001 0.05 White 28 3 -6.4036 1.0037 428 -6.38 <.0001 0.05 White 28 3 -6.4036 1.0037 428 -6.38 <.0001 0.05 White 28 3 -6.4036 1.0037 428 -6.38 <.0001 0.05 White 28 3 -6.4036 1.0037 428 -6.38 <.0001 0.05 White 28 3 -6.4036 1.0037 428 -6.38 <.0001 0.05 White 35 1 -9.9860 1.0509 427 -9.50 <.0001 0.05 White 35 1 -9.9860 1.0509 427 -9.50 <.0001 0.05 White 35 2 -13.1394 2.0655 417 -6.36 <.0001 0.05 White 35 2 -13.1394 2.0655 417 -6.36 <.0001 0.05 White 35 2 -13.1394 2.0655 417 -6.36 <.0001 0.05 White 35 2 -13.1394 2.0655 417 -6.36 <.0001 0.05 | RACEGRP Visit (N) Estimate Error DF t Value Pr > t Alpha Lower All Other Races 14 3 -6.8926 1.8839 401 -3.66 0.0003 0.05 -10.5961 White 14 3 -6.4045 0.8426 433 -7.60 <.0001 0.05 -8.0607 All Other Races 21 1 -9.1324 1.8815 447 -4.85 <.0001 0.05 -12.8302 White 21 1 -8.3083 0.8926 424 -9.31 <.0001 0.05 -10.0626 All Other Races 21 2 -9.6889 1.7502 409 -5.54 <.0001 0.05 -13.1294 White 21 2 -9.6889 1.7502 409 -5.54 <.0001 0.05 -13.1294 White Races 21 2 -7.9419 0.9105 430 -8.72 <.0001 0.05 -9.7315 All Other Races 21 3 -6.4777 2.0044 400 -3.23 0.0013 0.05 -10.4181 White 21 3 -6.5518 0.8889 429 -7.37 <.0001 0.05 -8.2989 All Other Races 28 1 -11.3582 2.1608 444 -5.26 <.0001 0.05 -8.2989 White 28 1 -9.2681 1.0250 433 -9.04 <.0001 0.05 -15.6049 White Races 28 2 -12.7159 1.9930 408 -6.38 <.0001 0.05 -10.8266 All Other Races 28 3 -5.5914 2.3069 414 -2.42 0.0158 0.05 -10.8291 All Other Races 28 3 -5.5914 2.3069 414 -2.42 0.0158 0.05 -10.1261 White 28 3 -6.4036 1.0037 428 -6.38 <.0001 0.05 -15.8948 White 28 3 -6.4036 1.0037 428 -6.38 <.0001 0.05 -15.8948 White 35 1 -9.9860 1.0509 427 -9.50 <.0001 0.05 -15.8948 White 35 2 -13.1394 2.0655 417 -6.36 <.0001 0.05 -17.1995 White 35 2 -10.0665 1.0666 439 -9.44 <.0001 0.05 -17.1627 |

CENTANAFADINE 28 OF 28 PROTOCOL 405-201-00013

# $$\operatorname{STAT-3.2}$$ MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

#### The Mixed Procedure

# Least Squares Means

| Effect | RACEGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Ellecc | NACEGINI | (14) | (14) | E3 CIMACE | BITOI | DE | c varue | 11 > 0 | Aipha | HOWEL | opper |
| AVISIT*TRTPN*RACEGRP | White | 35 | 3 | -6.9780 | 1.0307 | 426 | -6.77 | <.0001 | 0.05 | -9.0039 | -4.9521 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 42 | 1 | -11.5976 | 2.2803 | 430 | -5.09 | < .0001 | 0.05 | -16.0795 | -7.1158 |
| AVISIT*TRTPN*RACEGRP | White | 42 | 1 | -9.8108 | 1.0918 | 431 | -8.99 | < .0001 | 0.05 | -11.9568 | -7.6648 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 42 | 2 | -11.4938 | 2.1175 | 406 | -5.43 | <.0001 | 0.05 | -15.6564 | -7.3313 |
| AVISIT*TRTPN*RACEGRP | White | 42 | 2 | -9.2764 | 1.0974 | 433 | -8.45 | <.0001 | 0.05 | -11.4333 | -7.1195 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 42 | 3 | -4.9221 | 2.4639 | 416 | -2.00 | 0.0464 | 0.05 | -9.7653 | -0.07897 |
| AVISIT*TRTPN*RACEGRP | White | 42 | 3 | -7.3460 | 1.0634 | 424 | -6.91 | < .0001 | 0.05 | -9.4363 | -5.2558 |

CENTANAFADINE 1 OF 18 PROTOCOL 405-201-00013

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure

Model Information

WORK.INDATA Data Set Dependent Variable CHG Covariance Structure Unstructured Subject Effect SUBJID Estimation Method REML Residual Variance Method None Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger

Class Level Information

Class Levels Values

AVISITN 6 7 14 21 28 35 42

TRTPN 3 1 2 3

POOLCNTR 38

CENTANAFADINE


STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure

Class Level Information

Class Levels Values

SUBJID 438



CENTANAFADINE


STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure




CENTANAFADINE 4 OF 18

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure



CENTANAFADINE 5 OF 18 PROTOCOL 405-201-00013

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure



CENTANAFADINE 6 OF 18

PROTOCOL 405-201-00013 STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

------

The Mixed Procedure



CENTANAFADINE 7 OF 18 PROTOCOL 405-201-00013

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

......

The Mixed Procedure



CENTANAFADINE


STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure

Dimensions

Covariance Parameters 21
Columns in X 72
Columns in Z 0
Subjects 438
Max Obs per Subject 6

Number of Observations

Number of Observations Read 2292
Number of Observations Used 2292
Number of Observations Not Used 0

Iteration History

 Iteration
 Evaluations
 -2 Res Log Like
 Criterion

 0
 1
 16529.25629156
 0.00013099

 1
 2
 14254.41720522
 0.00013099

 2
 1
 14253.71654441
 0.00000106

 3
 1
 14253.71110309
 0.00000000

CENTANAFADINE 9 OF 18

PROTOCOL 405-201-00013 STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

-----

The Mixed Procedure

Convergence criteria met.

#### Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | 52.4121 |
| UN(2,1) | SUBJID | 40.1625 |
| UN(2,2) | SUBJID | 72.3841 |
| UN(3,1) | SUBJID | 37.8797 |
| UN(3,2) | SUBJID | 62.0385 |
| UN(3,3) | SUBJID | 81.2283 |
| UN(4,1) | SUBJID | 37.2709 |
| UN(4,2) | SUBJID | 62.5977 |
| UN(4,3) | SUBJID | 77.1568 |
| UN (4,4) | SUBJID | 105.57 |
| UN(5,1) | SUBJID | 38.1278 |
| UN(5,2) | SUBJID | 63.2146 |
| UN(5,3) | SUBJID | 80.4768 |
| UN(5,4) | SUBJID | 95.8339 |
| UN(5,5) | SUBJID | 110.37 |
| UN(6,1) | SUBJID | 38.5259 |
| UN(6,2) | SUBJID | 64.2868 |
| UN(6,3) | SUBJID | 78.4374 |

CENTANAFADINE 10 OF 18


# STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

......

The Mixed Procedure

#### Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(6,4) | SUBJID | 96.1387 |
| UN(6,5) | SUBJID | 99.0726 |
| UN (6.6) | SUBJID | 117.05 |

# Fit Statistics

| -2 Res Log Likelihood | 14253.7 |
|--------------------------|---------|
| AIC (Smaller is Better) | 14295.7 |
| AICC (Smaller is Better) | 14296.1 |
| BIC (Smaller is Better) | 14381.4 |

# Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSo |
|----|------------|------------|
| 20 | 2275.55 | <.0001 |

CENTANAFADINE 11 OF 18

PROTOCOL 405-201-00013 STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure

Solution for Fixed Effects

| | Pooled | Analysis | Planned | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Center | Visit | Treatment | | Standard | | | |
| Effect | Number | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| Intercept | | | | 0.4831 | 4.8082 | 567 | 0.10 | 0.9200 |
| AVISITN | | 7 | | -0.7357 | 2.9385 | 398 | -0.25 | 0.8024 |
| AVISITN | | 14 | | -0.8075 | 2.4473 | 388 | -0.33 | 0.7416 |
| AVISITN | | 21 | | -2.8674 | 2.0446 | 361 | -1.40 | 0.1616 |
| AVISITN | | 28 | | 2.9224 | 1.7765 | 345 | 1.64 | 0.1009 |
| AVISITN | | 35 | | 0.5711 | 1.7576 | 352 | 0.32 | 0.7454 |
| AVISITN | | 42 | | 0 | | | | |
| TRTPN | | | 1 | -3.1497 | 1.3407 | 400 | -2.35 | 0.0193 |
| TRTPN | | | 2 | -2.7448 | 1.3267 | 392 | -2.07 | 0.0392 |
| TRTPN | | | 3 | 0 | | | | |
| AVISITN*TRTPN | | 7 | 1 | 1.8448 | 1.2086 | 398 | 1.53 | 0.1277 |
| AVISITN*TRTPN | | 7 | 2 | 2.8699 | 1.1928 | 393 | 2.41 | 0.0166 |
| AVISITN*TRTPN | | 7 | 3 | 0 | | | | |
| AVISITN*TRTPN | | 14 | 1 | 2.1849 | 1.0072 | 387 | 2.17 | 0.0307 |
| AVISITN*TRTPN | | 14 | 2 | 2.4905 | 0.9856 | 382 | 2.53 | 0.0119 |
| AVISITN*TRTPN | | 14 | 3 | 0 | | | | |
| AVISITN*TRTPN | | 21 | 1 | 1.2025 | 0.8417 | 362 | 1.43 | 0.1540 |
| AVISITN*TRTPN | | 21 | 2 | 0.9723 | 0.8240 | 360 | 1.18 | 0.2388 |
| AVISITN*TRTPN | | 21 | 3 | 0 | | | | |

SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 18JUN2020 10:00; ANALYSIS DATASET CREATED: 11JUN2020 07:28 PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC STAT/stat1.sas

OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-4.1.1 FINAL

CENTANAFADINE 12 OF 18 PROTOCOL 405-201-00013

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

# The Mixed Procedure

# Solution for Fixed Effects

| | Pooled<br>Center | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Number | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| AVISITN*TRTPN | | 28 | 1 | -0.2340 | 0.7283 | 342 | -0.32 | 0.7481 |
| AVISITN*TRTPN | | 28 | 2 | -0.6011 | 0.7150 | 343 | -0.84 | 0.4011 |
| AVISITN*TRTPN | | 28 | 3 | 0 | | | | |
| AVISITN*TRTPN | | 35 | 1 | 0.07206 | 0.7186 | 348 | 0.10 | 0.9202 |
| AVISITN*TRTPN | | 35 | 2 | -0.7607 | 0.7085 | 349 | -1.07 | 0.2837 |
| AVISITN*TRTPN | | 35 | 3 | 0 | | | | |
| AVISITN*TRTPN | | 42 | 1 | 0 | | | | |
| AVISITN*TRTPN | | 42 | 2 | 0 | | | | |
| AVISITN*TRTPN | | 42 | 3 | 0 | | | | |
| POOLCNTR | | | | -1.5781 | 3.9342 | 391 | -0.40 | 0.6885 |
| POOLCNTR | | | | -1.0310 | 3.8358 | 391 | -0.27 | 0.7882 |
| POOLCNTR | | | | -2.1594 | 3.9655 | 391 | -0.54 | 0.5864 |
| POOLCNTR | | | | -1.5289 | 3.7488 | 393 | -0.41 | 0.6836 |
| POOLCNTR | | | | -1.5067 | 3.8012 | 392 | -0.40 | 0.6920 |
| POOLCNTR | | | | -2.4888 | 4.2744 | 391 | -0.58 | 0.5607 |
| POOLCNTR | | | | -8.3662 | 4.3446 | 393 | -1.93 | 0.0549 |
| POOLCNTR | | | | -6.3243 | 5.3927 | 393 | -1.17 | 0.2416 |
| POOLCNTR | | | | -5.4404 | 3.9685 | 392 | -1.37 | 0.1712 |
| POOLCNTR | | | | -1.9497 | 4.7926 | 406 | -0.41 | 0.6844 |

CENTANAFADINE 13 OF 18 PROTOCOL 405-201-00013

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

#### The Mixed Procedure

# Solution for Fixed Effects

| | Pooled<br>Center | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Number | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| POOLCNTR | | | | -3.3328 | 3.7186 | 392 | -0.90 | 0.3707 |
| POOLCNTR | | | | -5.6893 | 4.1349 | 391 | -1.38 | 0.1696 |
| POOLCNTR | | | | 0.8859 | 4.2071 | 397 | 0.21 | 0.8333 |
| POOLCNTR | | | | -3.4584 | 4.1907 | 393 | -0.83 | 0.4097 |
| POOLCNTR | | | | -2.1719 | 4.2744 | 391 | -0.51 | 0.6117 |
| POOLCNTR | | | | -3.4300 | 4.7326 | 392 | -0.72 | 0.4690 |
| POOLCNTR | | | | -3.1079 | 3.9681 | 391 | -0.78 | 0.4340 |
| POOLCNTR | | | | -4.5105 | 4.3481 | 391 | -1.04 | 0.3002 |
| POOLCNTR | | | | -0.4554 | 5.3811 | 393 | -0.08 | 0.9326 |
| POOLCNTR | | | | -1.5914 | 4.4306 | 394 | -0.36 | 0.7197 |
| POOLCNTR | | | | -5.6339 | 5.0120 | 390 | -1.12 | 0.2617 |
| POOLCNTR | | | | 0.2294 | 4.7268 | 391 | 0.05 | 0.9613 |
| POOLCNTR | | | | -1.1086 | 4.7948 | 392 | -0.23 | 0.8173 |
| POOLCNTR | | | | -3.8392 | 4.5625 | 394 | -0.84 | 0.4006 |
| POOLCNTR | | | | -1.8688 | 3.8721 | 393 | -0.48 | 0.6296 |
| POOLCNTR | | | | -4.7987 | 4.2584 | 393 | -1.13 | 0.2605 |
| POOLCNTR | | | | -4.5967 | 4.1713 | 391 | -1.10 | 0.2712 |
| POOLCNTR | | | | -4.0969 | 4.7405 | 397 | -0.86 | 0.3880 |
| POOLCNTR | | | | -12.4605 | 3.8212 | 392 | -3.26 | 0.0012 |

CENTANAFADINE 14 OF 18 PROTOCOL 405-201-00013

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

\_\_\_\_\_

# The Mixed Procedure

# Solution for Fixed Effects

| | Pooled | Analysis | Planned | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Center | Visit | Treatment | | Standard | | | |
| Effect | Number | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| POOLCNTR | | | | 2.2378 | 5.3865 | 390 | 0.42 | 0.6780 |
| POOLCNTR | | | | 3.2557 | 4.5695 | 390 | 0.71 | 0.4766 |
| POOLCNTR | | | | -2.8411 | 4.9870 | 390 | -0.57 | 0.5692 |
| POOLCNTR | | | | -2.4274 | 5.0523 | 397 | -0.48 | 0.6312 |
| POOLCNTR | | | | -1.0008 | 3.9085 | 391 | -0.26 | 0.7980 |
| POOLCNTR | | | | -5.1075 | 3.8314 | 391 | -1.33 | 0.1833 |
| POOLCNTR | | | | -1.5870 | 4.9866 | 392 | -0.32 | 0.7505 |
| POOLCNTR | | | | -1.6255 | 4.9908 | 392 | -0.33 | 0.7448 |
| POOLCNTR | | | | 0 | | | | |
| BASE*AVISITN | | 7 | | -0.02833 | 0.06074 | 406 | -0.47 | 0.6411 |
| BASE*AVISITN | | 14 | | -0.08413 | 0.06890 | 455 | -1.22 | 0.2227 |
| BASE*AVISITN | | 21 | | -0.03354 | 0.07241 | 456 | -0.46 | 0.6434 |
| BASE*AVISITN | | 28 | | -0.1732 | 0.08145 | 469 | -2.13 | 0.0340 |
| BASE*AVISITN | | 35 | | -0.1373 | 0.08324 | 466 | -1.65 | 0.0998 |
| BASE*AVISITN | | 42 | | -0.1177 | 0.08570 | 465 | -1.37 | 0.1704 |

CENTANAFADINE 15 OF 18 PROTOCOL 405-201-00013

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

# The Mixed Procedure

# Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------------|-----------|-----------|---------|--------|
| AVISITN | 5 | 380 | 2.06 | 0.0694 |
| TRTPN | 2 | 400 | 3.05 | 0.0482 |
| AVISITN*TRTPN | 10 | 563 | 1.68 | 0.0815 |
| POOLCNTR | 37 | 396 | 2.25 | <.0001 |
| BASE*AVISITN | 6 | 405 | 2.18 | 0.0443 |

# Estimates

| | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| DAY7 1 vs 3 | -1.3049 | 0.8584 | 396 | -1.52 | 0.1292 | 0.05 | -2.9924 | 0.3826 |
| DAY7 2 vs 3 | 0.1251 | 0.8581 | 396 | 0.15 | 0.8841 | 0.05 | -1.5618 | 1.8121 |
| DAY14 1 vs 3 | -0.9648 | 1.0193 | 403 | -0.95 | 0.3444 | 0.05 | -2.9686 | 1.0390 |
| DAY14 2 vs 3 | -0.2542 | 1.0168 | 400 | -0.25 | 0.8027 | 0.05 | -2.2531 | 1.7446 |
| DAY21 1 vs 3 | -1.9472 | 1.0892 | 398 | -1.79 | 0.0746 | 0.05 | -4.0885 | 0.1941 |
| DAY21 2 vs 3 | -1.7725 | 1.0824 | 391 | -1.64 | 0.1023 | 0.05 | -3.9006 | 0.3556 |
| DAY28 1 vs 3 | -3.3837 | 1.2590 | 401 | -2.69 | 0.0075 | 0.05 | -5.8587 | -0.9087 |
| DAY28 2 vs 3 | -3.3458 | 1.2483 | 395 | -2.68 | 0.0077 | 0.05 | -5.8000 | -0.8917 |

CENTANAFADINE 16 OF 18 PROTOCOL 405-201-00013

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

......

#### The Mixed Procedure

#### Estimates

| Label | | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|
| DAY35 | 1 vs 3 | -3.0776 | 1.2921 | 398 | -2.38 | 0.0177 | 0.05 | -5.6178 | -0.5375 |
| DAY35 | 2 vs 3 | -3.5055 | 1.2838 | 394 | -2.73 | 0.0066 | 0.05 | -6.0294 | -0.9816 |
| DAY42 | 1 vs 3 | -3.1497 | 1.3407 | 400 | -2.35 | 0.0193 | 0.05 | -5.7855 | -0.5139 |
| DAY42 | 2 vs 3 | -2.7448 | 1.3267 | 392 | -2.07 | 0.0392 | 0.05 | -5.3532 | -0.1364 |

# Least Squares Means

| Effect | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN | 7 | 1 | -5.4832 | 0.6575 | 405 | -8.34 | <.0001 | 0.05 | -6.7757 | -4.1907 |
| AVISITN*TRTPN | 7 | 2 | -4.0531 | 0.6710 | 406 | -6.04 | <.0001 | 0.05 | -5.3721 | -2.7341 |
| AVISITN*TRTPN | 7 | 3 | -4.1783 | 0.6708 | 402 | -6.23 | <.0001 | 0.05 | -5.4970 | -2.8596 |
| AVISITN*TRTPN | 14 | 1 | -7.4261 | 0.7642 | 431 | -9.72 | <.0001 | 0.05 | -8.9281 | -5.9242 |
| AVISITN*TRTPN | 14 | 2 | -6.7156 | 0.7740 | 436 | -8.68 | <.0001 | 0.05 | -8.2368 | -5.1943 |
| AVISITN*TRTPN | 14 | 3 | -6.4613 | 0.7759 | 437 | -8.33 | <.0001 | 0.05 | -7.9862 | -4.9364 |
| AVISITN*TRTPN | 21 | 1 | -8.4638 | 0.8150 | 436 | -10.39 | <.0001 | 0.05 | -10.0655 | -6.8620 |
| AVISITN*TRTPN | 21 | 2 | -8.2891 | 0.8186 | 436 | -10.13 | <.0001 | 0.05 | -9.8980 | -6.6801 |

SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 18JUN2020 10:00; ANALYSIS DATASET CREATED: 11JUN2020 07:28 PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC STAT/statl.sas

OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-4.1.1 FINAL


CENTANAFADINE 17 OF 18

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure

Least Squares Means

| | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 21 | 3 | -6.5166 | 0.8184 | 435 | -7.96 | <.0001 | 0.05 | -8.1251 | -4.9080 |
| AVISITN*TRTPN | 28 | 1 | -9.6450 | 0.9350 | 444 | -10.32 | <.0001 | 0.05 | -11.4825 | -7.8075 |
| AVISITN*TRTPN | 28 | 2 | -9.6071 | 0.9317 | 446 | -10.31 | <.0001 | 0.05 | -11.4382 | -7.7761 |
| AVISITN*TRTPN | 28 | 3 | -6.2613 | 0.9266 | 437 | -6.76 | <.0001 | 0.05 | -8.0825 | -4.4401 |
| AVISITN*TRTPN | 35 | 1 | -10.2665 | 0.9572 | 438 | -10.73 | <.0001 | 0.05 | -12.1478 | -8.3852 |
| AVISITN*TRTPN | 35 | 2 | -10.6944 | 0.9567 | 446 | -11.18 | <.0001 | 0.05 | -12.5746 | -8.8143 |
| AVISITN*TRTPN | 35 | 3 | -7.1889 | 0.9493 | 434 | -7.57 | <.0001 | 0.05 | -9.0547 | -5.3231 |
| AVISITN*TRTPN | 42 | 1 | -10.1321 | 0.9918 | 440 | -10.22 | <.0001 | 0.05 | -12.0814 | -8.1829 |
| AVISITN*TRTPN | 42 | 2 | -9.7272 | 0.9830 | 439 | -9.89 | <.0001 | 0.05 | -11.6593 | -7.7951 |
| AVISITN*TRTPN | 42 | 3 | -6.9824 | 0.9807 | 436 | -7.12 | <.0001 | 0.05 | -8.9099 | -5.0549 |

CENTANAFADINE 18 OF 18


STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

......

The Mixed Procedure

Tests of Effect Slices

| | Analysis | | | | |
|---------------|----------|-----|-----|---------|--------|
| | Visit | Num | Den | | |
| Effect | (N) | DF | DF | F Value | Pr > F |
| | - | | 205 | | 0 1001 |
| AVISITN*TRTPN | 7 | 2 | 397 | 1.71 | 0.1821 |
| AVISITN*TRTPN | 14 | 2 | 402 | 0.48 | 0.6181 |
| AVISITN*TRTPN | 21 | 2 | 397 | 1.97 | 0.1409 |
| AVISITN*TRTPN | 28 | 2 | 400 | 4.82 | 0.0085 |
| AVISITN*TRTPN | 35 | 2 | 399 | 4.44 | 0.0124 |
| AVISITN*TRTPN | 42 | 2 | 398 | 3.30 | 0.0377 |

CENTANAFADINE 1 OF 14 PROTOCOL 405-201-00013

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

The Mixed Procedure

Model Information

WORK.INDATA Data Set Dependent Variable CHG Covariance Structure Unstructured Subject Effect SUBJID Estimation Method REML Residual Variance Method None Fixed Effects SE Method Model-Based Degrees of Freedom Method Satterthwaite

Class Level Information

Class Levels Values

AVISITN 6 7 14 21 28 35 42

TRTPN 3 1 2 3

POOLCNTR 38

CENTANAFADINE 2 OF 14 PROTOCOL 405-201-00013

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE

(Efficacy Sample)

The Mixed Procedure

Class Level Information

Values Class Levels

SUBJID 438



CENTANAFADINE

3 OF 14

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

......

The Mixed Procedure




CENTANAFADINE 4 OF 14

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

The Mixed Procedure



CENTANAFADINE 5 OF 14 PROTOCOL 405-201-00013

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

The Mixed Procedure




CENTANAFADINE 6 OF 14

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

The Mixed Procedure



CENTANAFADINE 7 OF 14 PROTOCOL 405-201-00013

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

The Mixed Procedure



| CENTANAFADINE | 8 OF 14 |
|------------------------|---------|

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE

(Efficacy Sample)

------

#### The Mixed Procedure

#### Dimensions

| Covariance | Parameters | 21 |
|------------|------------|-----|
| Columns in | X | 72 |
| Columns in | Z | 0 |
| Subjects | | 438 |
| Max Obs pe | r Subject | 6 |

# Number of Observations

| Number | of | Observations | Read | 2292 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 2292 |
| Number | of | Observations | Not Used | 0 |

# Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 16529.25629156 | |
| 1 | 2 | 14254.41720522 | 0.00013099 |
| 2 | 1 | 14253.71654441 | 0.00000106 |
| 3 | 1 | 14253.71110309 | 0.00000000 |

CENTANAFADINE 9 OF 14 PROTOCOL 405-201-00013

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

The Mixed Procedure

Convergence criteria met.

#### Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | 52.4121 |
| UN(2,1) | SUBJID | 40.1625 |
| UN(2,2) | SUBJID | 72.3841 |
| UN(3,1) | SUBJID | 37.8797 |
| UN(3,2) | SUBJID | 62.0385 |
| UN(3,3) | SUBJID | 81.2283 |
| UN(4,1) | SUBJID | 37.2709 |
| UN(4,2) | SUBJID | 62.5977 |
| UN(4,3) | SUBJID | 77.1568 |
| UN (4,4) | SUBJID | 105.57 |
| UN(5,1) | SUBJID | 38.1278 |
| UN(5,2) | SUBJID | 63.2146 |
| UN(5,3) | SUBJID | 80.4768 |
| UN(5,4) | SUBJID | 95.8339 |
| UN(5,5) | SUBJID | 110.37 |
| UN(6,1) | SUBJID | 38.5259 |
| UN(6,2) | SUBJID | 64.2868 |
| UN(6,3) | SUBJID | 78.4374 |

CENTANAFADINE 10 OF 14 PROTOCOL 405-201-00013

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

......

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|-----------|----------|----------|
| UN(6,4) | SUBJID | 96.1387 |
| UN(6,5) | SUBJID | 99.0726 |
| IIN (6 6) | SIIR.TTD | 117 05 |

# Fit Statistics

| -2 Res Log Likelihood | 14253.7 |
|--------------------------|---------|
| AIC (Smaller is Better) | 14295.7 |
| AICC (Smaller is Better) | 14296.1 |
| BIC (Smaller is Better) | 14381.4 |

# Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSc |
|----|------------|------------|
| 20 | 2275.55 | <.0001 |

CENTANAFADINE 11 OF 14 PROTOCOL 405-201-00013

# STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

# The Mixed Procedure

# Type 3 Tests of Fixed Effects

| | Num | Den | | |
|---------------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| AVISITN | 5 | 384 | 2.09 | 0.0662 |
| TRTPN | 2 | 400 | 3.06 | 0.0482 |
| AVISITN*TRTPN | 10 | 396 | 1.71 | 0.0774 |
| POOLCNTR | 37 | 396 | 2.31 | <.0001 |
| BASE*AVISITN | 6 | 404 | 2.21 | 0.0415 |

# Estimates

| | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| DAY7 1 vs 3 | -1.3049 | 0.8582 | 396 | -1.52 | 0.1291 | 0.05 | -2.9920 | 0.3822 |
| DAY7 2 vs 3 | 0.1251 | 0.8578 | 396 | 0.15 | 0.8841 | 0.05 | -1.5614 | 1.8116 |
| DAY14 1 vs 3 | -0.9648 | 1.0190 | 403 | -0.95 | 0.3443 | 0.05 | -2.9680 | 1.0384 |
| DAY14 2 vs 3 | -0.2542 | 1.0165 | 400 | -0.25 | 0.8026 | 0.05 | -2.2526 | 1.7442 |
| DAY21 1 vs 3 | -1.9472 | 1.0889 | 398 | -1.79 | 0.0745 | 0.05 | -4.0879 | 0.1935 |
| DAY21 2 vs 3 | -1.7725 | 1.0822 | 391 | -1.64 | 0.1022 | 0.05 | -3.9001 | 0.3551 |
| DAY28 1 vs 3 | -3.3837 | 1.2584 | 401 | -2.69 | 0.0075 | 0.05 | -5.8576 | -0.9098 |
| DAY28 2 vs 3 | -3.3458 | 1.2478 | 395 | -2.68 | 0.0076 | 0.05 | -5.7990 | -0.8927 |

CENTANAFADINE 12 OF 14 PROTOCOL 405-201-00013

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

......

#### The Mixed Procedure

# Estimates

| | | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Label | | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| DAY35 | 1 vs 3 | -3.0776 | 1.2914 | 398 | -2.38 | 0.0176 | 0.05 | -5.6164 | -0.5389 |
| DAY35 | 2 vs 3 | -3.5055 | 1.2831 | 394 | -2.73 | 0.0066 | 0.05 | -6.0281 | -0.9829 |
| DAY42 | 1 vs 3 | -3.1497 | 1.3398 | 400 | -2.35 | 0.0192 | 0.05 | -5.7836 | -0.5158 |
| DAY42 | 2 vs 3 | -2.7448 | 1.3259 | 392 | -2.07 | 0.0391 | 0.05 | -5.3516 | -0.1379 |

# Least Squares Means

| | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 7 | 1 | -5.4832 | 0.6561 | 405 | -8.36 | <.0001 | 0.05 | -6.7731 | -4.1934 |
| AVISITN*TRTPN | 7 | 2 | -4.0531 | 0.6693 | 406 | -6.06 | <.0001 | 0.05 | -5.3688 | -2.7374 |
| AVISITN*TRTPN | 7 | 3 | -4.1783 | 0.6693 | 402 | -6.24 | <.0001 | 0.05 | -5.4940 | -2.8626 |
| AVISITN*TRTPN | 14 | 1 | -7.4261 | 0.7629 | 431 | -9.73 | <.0001 | 0.05 | -8.9256 | -5.9266 |
| AVISITN*TRTPN | 14 | 2 | -6.7156 | 0.7725 | 436 | -8.69 | <.0001 | 0.05 | -8.2339 | -5.1972 |
| AVISITN*TRTPN | 14 | 3 | -6.4613 | 0.7745 | 437 | -8.34 | <.0001 | 0.05 | -7.9835 | -4.9392 |
| AVISITN*TRTPN | 21 | 1 | -8.4638 | 0.8137 | 436 | -10.40 | <.0001 | 0.05 | -10.0631 | -6.8645 |
| AVISITN*TRTPN | 21 | 2 | -8.2891 | 0.8172 | 436 | -10.14 | <.0001 | 0.05 | -9.8952 | -6.6829 |

SOURCE: MMRMOUT; TABLE: statlab.lis; RUN: 18JUN2020 10:00; ANALYSIS DATASET CREATED: 11JUN2020 07:28 PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC STAT/statl.sas

OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-4.1.2 FINAL

CENTANAFADINE 13 OF 14 PROTOCOL 405-201-00013

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

The Mixed Procedure

Least Squares Means

| | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 21 | 3 | -6.5166 | 0.8171 | 435 | -7.98 | <.0001 | 0.05 | -8.1225 | -4.9107 |
| AVISITN*TRTPN | 28 | 1 | -9.6450 | 0.9336 | 444 | -10.33 | <.0001 | 0.05 | -11.4799 | -7.8102 |
| AVISITN*TRTPN | 28 | 2 | -9.6071 | 0.9302 | 446 | -10.33 | <.0001 | 0.05 | -11.4353 | -7.7790 |
| AVISITN*TRTPN | 28 | 3 | -6.2613 | 0.9253 | 437 | -6.77 | <.0001 | 0.05 | -8.0799 | -4.4427 |
| AVISITN*TRTPN | 35 | 1 | -10.2665 | 0.9558 | 438 | -10.74 | <.0001 | 0.05 | -12.1451 | -8.3880 |
| AVISITN*TRTPN | 35 | 2 | -10.6944 | 0.9551 | 446 | -11.20 | <.0001 | 0.05 | -12.5714 | -8.8175 |
| AVISITN*TRTPN | 35 | 3 | -7.1889 | 0.9479 | 434 | -7.58 | <.0001 | 0.05 | -9.0520 | -5.3258 |
| AVISITN*TRTPN | 42 | 1 | -10.1321 | 0.9902 | 440 | -10.23 | <.0001 | 0.05 | -12.0783 | -8.1860 |
| AVISITN*TRTPN | 42 | 2 | -9.7272 | 0.9815 | 439 | -9.91 | <.0001 | 0.05 | -11.6561 | -7.7983 |
| AVISITN*TRTPN | 42 | 3 | -6.9824 | 0.9792 | 436 | -7.13 | <.0001 | 0.05 | -8.9069 | -5.0579 |

CENTANAFADINE 14 OF 14 PROTOCOL 405-201-00013

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

The Mixed Procedure

Tests of Effect Slices

| | Analysis | | | | |
|---------------|----------|-----|-----|---------|--------|
| | Visit | Num | Den | | |
| Effect | (N) | DF | DF | F Value | Pr > F |
| AVISITN*TRTPN | 7 | 2 | 397 | 1.71 | 0.1819 |
| AVISITN*TRTPN | 14 | 2 | 402 | 0.48 | 0.6179 |
| AVISITN*TRTPN | 21 | 2 | 397 | 1.97 | 0.1407 |
| AVISITN*TRTPN | 28 | 2 | 400 | 4.83 | 0.0085 |
| AVISITN*TRTPN | 35 | 2 | 399 | 4.44 | 0.0124 |
| AVISITN*TRTPN | 42 | 2 | 398 | 3.31 | 0.0376 |

CENTANAFADINE 1 OF 6 PROTOCOL 405-201-00013

STAT-4.2

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, LOCF (Efficacy Sample)

.....

The GLM Procedure

Class Level Information

Class Levels Values

TRTPN 3 1 2 3

POOLCNTR 38

Number of Observations Read 438 Number of Observations Used 438
CENTANAFADINE 2 OF 6 PROTOCOL 405-201-00013

STAT-4.2

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, LOCF (Efficacy Sample)

The GLM Procedure

Dependent Variable: CHG Change from Baseline

| Source | | DF | Sum<br>Squar | | Mean Sq | uare F | Value | Pr > F |
|---|---|---|---|---|---|---|---|---|
| Model | | 40 | 7613.605 | 24 | 190.3 | 4013 | 1.72 | 0.0053 |
| Error | | 397 | 43878.351 | .38 | 110.5 | 2481 | | |
| Corrected Total | | 437 | 51491.956 | 62 | | | | |
| | R-Square<br>0.147860 | | f Var | Root M: | | CHG Mean | | |
| Source | | DF | Type III | SS 1 | Mean Sq | uare F | Value | Pr > F |
| TRTPN<br>POOLCNTR<br>BASE | | 2<br>37<br>1 | 612.6426<br>5773.4495<br>231.3540 | 66 | 306.32<br>156.03<br>231.35 | 9177 | 2.77<br>1.41<br>2.09 | 0.0638<br>0.0603<br>0.1487 |

CENTANAFADINE 3 OF 6 PROTOCOL 405-201-00013

STAT-4.2 Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, LOCF (Efficacy Sample)

......

## The GLM Procedure

| Level of | | CHC | G | BA | SE |
|----------|-----|-------------|------------|------------|------------|
| TRTPN | N | Mean | Std Dev | Mean | Std Dev |
| 1 | 147 | -9.97278912 | 11.8933305 | 39.5986395 | 6.69354613 |
| 2 | 147 | -9.85714286 | 10.3632649 | 39.5646259 | 6.81664766 |
| 3 | 144 | -7.45833333 | 10.0959557 | 39.5347222 | 7.19840036 |

CENTANAFADINE 4 OF 6 PROTOCOL 405-201-00013

STAT-4.2

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, LOCF (Efficacy Sample)

The GLM Procedure Least Squares Means

| | | Standard | LSMEAN | |
|-------|-------------|-----------|---------|--------|
| TRTPN | CHG LSMEAN | Error | Pr > t | Number |
| 1 | -10.0466880 | 0.9524391 | <.0001 | 1 |
| 2 | -9.5942969 | 0.9741456 | <.0001 | 2 |
| 3 | -7.3212133 | 0.9759953 | <.0001 | 3 |

Least Squares Means for effect TRTPN Pr > |t| for H0: LSMean(i)=LSMean(j)

## Dependent Variable: CHG

| i/j | 1 | 2 | 3 |
|---|---|---|---|
| 1<br>2 | 0.7141 | 0.7141 | 0.0284<br>0.0674 |
| 3 | 0.0284 | 0.0674 | |
| TRTPN | CHG LSMEAN | 95% Confidence | ce Limits |
| 1<br>2 | -10.046688<br>-9.594297 | -11.919143<br>-11.509426 | -8.174233<br>-7.679168 |

CENTANAFADINE 5 OF 6 PROTOCOL 405-201-00013

STAT-4.2

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, LOCF (Efficacy Sample)

The GLM Procedure Least Squares Means

TRTPN CHG LSMEAN 95% Confidence Limits

3 -7.321213 -9.239979 -5.402448

Least Squares Means for Effect TRTPN

Difference 95% Confidence Limits for Between i LSMean(i)-LSMean(j) Means 2 -0.452391 -2.877963 1.973180 -2.725475 -5.161161 -0.289788 -2.273084 -4.709885 0.163718

NOTE: To ensure overall protection level, only probabilities associated with pre-planned comparisons should be used.

CENTANAFADINE 6 OF 6 PROTOCOL 405-201-00013

STAT-4.2

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, LOCF (Efficacy Sample)

The GLM Procedure

Dependent Variable: CHG Change from Baseline

| Parameter | Estimate | Standard<br>Error | t Value | Pr > t |
|-----------|-------------|-------------------|---------|---------|
| 1 vs 3 | -2.72547476 | 1.23893152 | -2.20 | 0.0284 |
| 2 vs 3 | -2.27308361 | 1.23949880 | -1.83 | 0.0674 |


STAT-4.3

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, OC (Efficacy Sample)

The GLM Procedure

Class Level Information

Class Levels Values
TRTPN 3 1 2 3

Number of Observations Read 438 Number of Observations Used 438


STAT-4.3

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, OC (Efficacy Sample)

The GLM Procedure

Dependent Variable: CHG Change from Baseline Sum of

| Source | | DF | Squar | res | Mean | Square | F Value | Pr > F |
|---|---|---|---|---|---|---|---|---|
| Model | | 3 | 1840.155 | 67 | 613 | 3.38522 | 5.36 | 0.0012 |
| Error | | 434 | 49651.800 | 95 | 114 | 1.40507 | | |
| Corrected Total | | 437 | 51491.956 | 62 | | | | |
| | R-Square<br>0.035737 | | f Var | Root N | | CHG Me | | |
| Source | | DF | Type III | SS | Mean | Square | F Value | Pr > F |
| TRTPN<br>BASE | | 2<br>1 | 578.7023<br>1255.8402 | | | 351182<br>840210 | 2.53<br>10.98 | 0.0809<br>0.0010 |


STAT-4.3

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, OC (Efficacy Sample)

## The GLM Procedure

| Level of | | CHC | G | BAS | SE |
|----------|-----|-------------|------------|------------|------------|
| TRTPN | N | Mean | Std Dev | Mean | Std Dev |
| 1 | 147 | -9.97278912 | 11.8933305 | 39.5986395 | 6.69354613 |
| 2 | 147 | -9.85714286 | 10.3632649 | 39.5646259 | 6.81664766 |
| 3 | 144 | -7.45833333 | 10.0959557 | 39.5347222 | 7.19840036 |


STAT-4.3

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, OC (Efficacy Sample)

\_\_\_\_\_

The GLM Procedure Least Squares Means

| | | Standard | | LSMEAN |
|-------|-------------|------------|---------|--------|
| TRTPN | CHG LSMEAN | Error | Pr > t | Number |
| 1 | -9.96480823 | 0.88219703 | <.0001 | 1 |
| 2 | -9.85753273 | 0.88219375 | <.0001 | 2 |
| 3 | -7.46608250 | 0.89133895 | <.0001 | 3 |

Least Squares Means for effect TRTPN Pr > |t| for H0: LSMean(i)=LSMean(j)

## Dependent Variable: CHG

| i/j | 1 | 2 | 3 |
|---|---|---|---|
| 1<br>2<br>3 | 0.9315<br>0.0469 | 0.9315<br>0.0572 | 0.0469<br>0.0572 |
| TRTPN | CHG LSMEAN | 95% Confidenc | ce Limits |
| 1<br>2 | -9.964808<br>-9.857533 | -11.698718<br>-11.591436 | -8.230898<br>-8.123629 |


STAT-4.3

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, OC (Efficacy Sample)

......

The GLM Procedure Least Squares Means

| TRTPN | CHG LSMEAN | 95% Confidence | ce Limits |
|-------|------------|----------------|-----------|
| 3 | -7.466082 | -9.217960 | -5.714205 |

Least Squares Means for Effect TRTPN

| | | DILIELEUCE | | |
|---|---|------------|----------------|------------|
| | | Between | 95% Confidence | Limits for |
| i | j | Means | LSMean(i)-L | SMean(j) |
| 1 | 2 | -0.107275 | -2.559390 | 2.344839 |
| 1 | 3 | -2.498726 | -4.963591 | -0.033860 |
| 2 | 3 | -2.391450 | -4.856302 | 0.073402 |

NOTE: To ensure overall protection level, only probabilities associated with pre-planned comparisons should be used.


STAT-4.3

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, OC (Efficacy Sample)

The GLM Procedure

Dependent Variable: CHG Change from Baseline

| Parameter | Estimate | Standard<br>Error | t Value | Pr > t |
|-----------|-------------|-------------------|---------|---------|
| 1 vs 3 | -2.49872573 | 1.25410047 | -1.99 | 0.0469 |
| 2 vs 3 | -2.39145023 | 1.25409345 | -1.91 | 0.0572 |

CENTANAFADINE 1 OF 2 PROTOCOL 405-201-00013

STAT-4.4

Proc GLM Output for Treatment by Center Interaction at Day 42 in AISRS Total Score, LOCF (Efficacy Sample)

(Efficacy Sample

------

The GLM Procedure

Class Level Information

Class Levels Values

TRTPN 3 1 2 3

POOLCNTR 38

Number of Observations Read 438 Number of Observations Used 438

CENTANAFADINE 2 OF 2


# STAT-4.4

Proc GLM Output for Treatment by Center Interaction at Day 42 in AISRS Total Score, LOCF (Efficacy Sample)

(Efficacy Sample

BASE

.------

The GLM Procedure

Dependent Variable: CHG Change from Baseline

| Source | | DF | Sum<br>Squar | | Mean : | Square | F | Value | Pr > F |
|---|---|---|---|---|---|---|---|---|---|
| Model | | 114 | 17280.040 | 47 | 151 | .57930 | | 1.43 | 0.0080 |
| Error | | 323 | 34211.916 | 15 | 105 | .91925 | | | |
| Corrected Total | | 437 | 51491.956 | 62 | | | | | |
| | R-Square | | f Var | Root M | | CHG Me | | | |
| | 0.335587 | -113 | .0050 | 10.291 | .71 | -9.1073 | 06 | | |
| Source | | DF | Type III | SS | Mean S | Square | F | Value | Pr > F |
| TRTPN POOLCNTR TRTPN*POOLCNTR | | 2<br>37<br>74 | 316.6105<br>5824.7243<br>9666.4352 | 54 | 157. | 305263<br>424983<br>627503 | | 1.49<br>1.49<br>1.23 | 0.2259<br>0.0390<br>0.1128 |
| TIVILIA LOODCIALIV | | / ユ | JUUU.4JJZ | JJ | ±00. | 021000 | | 1.20 | U. IIZO |

244.872536

244.872536 2.31 0.1294

CENTANAFADINE 1 OF 4 PROTOCOL 405-201-00013

STAT-4.5.1

Summary of Mean Change at Day 42 from Baseline in AISRS Total Score
By Center - LOCF (Efficacy Sample)

| | CTN SR 200MG | CTN SR 400MG | PLACEBO | TREATMENT | |
|---|---|---|---|---|---|
| CENTER | N LS MEAN (SE) | N LS MEAN (SE) | N LS MEAN (SE) | COMPARISON | LS MEAN DIFFERENCE <sup>1</sup> |
| OVERALL | 147 -10.0 (0.95) | 147 -9.59 (0.97) | 144 -7.32 (0.98) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -2.73 (-5.16, -0.29)<br>-2.27 (-4.71, 0.16) |
| | 5 -3.34 (4.60) | 6 -18.0 (4.20) | 6 -0.29 (4.20) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -3.04 (-15.3, 9.22)<br>-17.7 (-29.4, -6.05) |
| | 7 -7.96 (3.89) | 8 -1.67 (3.64) | 8 -5.76 (3.65) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -2.21 (-12.7, 8.30)<br>4.09 (-6.04, 14.22) |
| | 5 -12.9 (4.62) | 5 -12.1 (4.66) | 5 -11.3 (4.61) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -1.66 (-14.5, 11.15)<br>-0.78 (-13.6, 12.05) |
| | 11 -14.3 (3.10) | 11 -3.96 (3.10) | 10 -7.22 (3.31) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -7.07 (-16.0, 1.84)<br>3.26 (-5.68, 12.19) |
| | 9 -8.67 (3.44) | 8 -12.9 (3.65) | 8 -5.21 (3.65) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -3.46 (-13.3, 6.38)<br>-7.64 (-17.8, 2.48) |
| | 3 -11.5 (5.94) | 3 -16.1 (5.94) | 3 -11.3 (6.01) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -0.20 (-16.8, 16.40)<br>-4.82 (-21.4, 11.78) |
| | 3 -9.84 (5.95) | 2 -14.0 (7.28) | 3 -3.36 (5.95) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -6.47 (-23.0, 10.06)<br>-10.6 (-29.1, 7.84) |
| | 1 3.06 (10.3) | 1 -23.4 (10.3) | 1 -28.4 (10.3) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | 31.43 ( 2.79, 60.07)<br>5.01 (-23.7, 33.67) |
| | 5 -1.45 (4.61) | 5 -15.0 (4.62) | 6 -11.7 (4.20) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | 10.27 (-1.99, 22.54)<br>-3.24 (-15.5, 9.04) |
| | 2 -10.2 (7.29) | 1 -11.2 (10.3) | 2 -9.52 (7.31) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -0.64 (-20.9, 19.61)<br>-1.72 (-26.5, 23.08) |
| | 13 -6.23 (2.86) | 13 -11.4 (2.85) | 12 -2.49 (2.97) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -3.74 (-11.8, 4.37)<br>-8.92 (-17.0, -0.82) |

OVERALL TREATMENT DIFFERENCE IS DERIVED USING ANCOVA MODEL, WITH TREATMENT AND CENTER AS MAIN EFFECT AND BASELINE VALUE AS COVARIATE; BY CENTER DIFFERENCES ARE DERIVED USING ANCOVA MODEL, WITH TREATMENT AND CENTER AS MAIN EFFECT, TREATMENT BY CENTER INTERACTION, AND BASELINE VALUE AS COVARIATE.

NOTE: FOR ANALYSIS PURPOSE, SMALL CENTERS ARE POOLED TOGETHER.

CENTANAFADINE 2 OF 4

STAT-4.5.1

Summary of Mean Change at Day 42 from Baseline in AISRS Total Score
By Center - LOCF (Efficacy Sample)

AISRS TOTAL SCORE CTN SR 200MG \_\_\_ CTN SR 400MG \_\_\_ CENTER N LS MEAN (SE) N LS MEAN (SE) N LS MEAN (SE) COMPARISON LS MEAN DIFFERENCE<sup>1</sup> \_\_\_\_\_\_ 4 -9.58 (5.15) 4 -8.41 (5.15) 3 -11.5 (5.97) CTN SR 200MG VS. PLACEBO 1.87 (-13.6, 17.36) 3.05 (-12.5, 18.60) CTN SR 400MG VS. PLACEBO 4 -9.37 (5.15) 2 -8.00 (7.31) 4 -0.58 (5.15) CTN SR 200MG VS. PLACEBO -8.79 (-23.1, 5.54) CTN SR 400MG VS. PLACEBO -7.42 (-25.0, 10.15) 4 -11.1 (5.15) 3 -12.6 (5.95) 3 -0.13 (5.94) CTN SR 200MG VS. PLACEBO -11.0 (-26.4, 4.51) CTN SR 400MG VS. PLACEBO -12.5 (-29.1, 4.01) 3 0.78 (5.95) 3 -12.8 (5.99) 3 -2.84 (5.94) CTN SR 200MG VS. PLACEBO 3.62 (-12.9, 20.16) CTN SR 400MG VS. PLACEBO -9.99 (-26.6, 6.59) 2 -2.53 (7.40) -16.5 (-41.3, 8.32) 2 -16.7 (7.32) 1 -0.23 (10.3) CTN SR 200MG VS. PLACEBO CTN SR 400MG VS. PLACEBO -2.31 (-27.2, 22.60) 4 -9.65 (5.15) CTN SR 200MG VS. PLACEBO 5 -4.09 (4.61) 6 -14.0 (4.25) 5.57 (-8.02, 19.16) CTN SR 400MG VS. PLACEBO -4.37 (-17.5, 8.75) 3 -7.50 (5.97) 2 -8.00 (7.28) 3 -16.5 (5.94) CTN SR 200MG VS. PLACEBO 8.96 (-7.59, 25.51) CTN SR 400MG VS. PLACEBO 8.46 (-10.0, 26.94) 1 2.20 (10.3) 1 -21.1 (10.3) 1 -1.51 (10.3) CTN SR 200MG VS. PLACEBO 3.71 (-24.9, 32.35) CTN SR 400MG VS. PLACEBO -19.6 (-48.2, 9.07) 2 -7.22 (7.28) 2 -18.1 (7.29) 3 -17.8 (5.94) CTN SR 200MG VS. PLACEBO 10.62 (-7.87, 29.12) -0.24 (-18.7, 18.25) CTN SR 400MG VS. PLACEBO 2 -29.1 (7.30) 1 0.50 (10.3) 1 -3.51 (10.3) CTN SR 200MG VS. PLACEBO -25.6 (-50.5, -0.77) CTN SR 400MG VS. PLACEBO 4.01 (-24.7, 32.67) 2 -7.87 (7.28) 1 5.06 (10.3) 2 0.77 (7.28) CTN SR 200MG VS. PLACEBO -8.64 (-28.9, 11.60) 4.29 (-20.5, 29.09) CTN SR 400MG VS. PLACEBO 2 -0.78 (7.37) 2 -8.14 (7.33) 1 -1.66 (10.3) CTN SR 200MG VS. PLACEBO 0.88 (-24.1, 25.87) CTN SR 400MG VS. PLACEBO -6.48 (-31.4, 18.46)

NOTE: FOR ANALYSIS PURPOSE, SMALL CENTERS ARE POOLED TOGETHER.

OVERALL TREATMENT DIFFERENCE IS DERIVED USING ANCOVA MODEL, WITH TREATMENT AND CENTER AS MAIN EFFECT AND BASELINE VALUE AS COVARIATE; BY CENTER DIFFERENCES ARE DERIVED USING ANCOVA MODEL, WITH TREATMENT AND CENTER AS MAIN EFFECT, TREATMENT BY CENTER INTERACTION, AND BASELINE VALUE AS COVARIATE.

3 OF 4

CENTANAFADINE

STAT-4.5.1

Summary of Mean Change at Day 42 from Baseline in AISRS Total Score
By Center - LOCF (Efficacy Sample)

| | CTN SR 200MG | CTN SR 400MG | PLACEBO | TREATMENT | |
|---|---|---|---|---|---|
| CENTER | N LS MEAN (SE) | N LS MEAN (SE) | N LS MEAN (SE) | COMPARISON | LS MEAN DIFFERENCE¹ |
| | 2 -20.1 (7.29) | 2 -12.2 (7.28) | 2 1.85 (7.28) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -21.9 (-42.2, -1.68)<br>-14.0 (-34.2, 6.25) |
| | 7 -14.7 (3.91) | 8 -5.20 (3.65) | 7 -6.89 (3.90) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -7.81 (-18.6, 3.01)<br>1.69 (-8.79, 12.17) |
| | 3 -19.3 (5.96) | 4 -11.7 (5.15) | 2 -6.87 (7.28) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -12.4 (-31.0, 6.09)<br>-4.85 (-22.4, 12.69) |
| | 3 -11.0 (5.98) | 4 -7.26 (5.15) | 3 -15.9 (5.96) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | 4.95 (-11.6, 21.49)<br>8.69 (-6.80, 24.17) |
| | 1 -15.5 (10.3) | 2 -11.0 (7.34) | 2 -15.2 (7.32) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -0.28 (-25.1, 24.54)<br>4.28 (-16.0, 24.53) |
| | 9 -26.4 (3.52) | 13 -14.5 (2.95) | 12 -14.1 (3.10) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -12.3 (-21.2, -3.37)<br>-0.42 (-8.53, 7.69) |
| | 1 -5.95 (10.3) | 1 -2.53 (10.3) | 1 4.62 (10.3) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -10.6 (-39.2, 18.07)<br>-7.14 (-35.8, 21.49) |
| | 2 -1.93 (7.31) | 2 2.70 (7.30) | 2 -1.58 (7.28) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -0.35 (-20.6, 19.91)<br>4.27 (-16.0, 24.58) |
| | 1 -10.1 (10.3) | 2 -15.2 (7.28) | 1 -10.2 (10.3) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | 0.16 (-28.5, 28.83)<br>-4.99 (-29.8, 19.84) |
| | 2 -21.0 (7.28) | 1 -2.64 (10.3) | 1 -0.78 (10.3) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -20.2 (-45.0, 4.59)<br>-1.86 (-30.5, 26.78) |
| | 6 -4.42 (4.22) | 6 -3.87 (4.20) | 6 -8.94 (4.20) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | 4.52 (-7.22, 16.25)<br>5.07 (-6.62, 16.76) |
| | 7 -2.82 (3.89) | 7 -9.31 (3.92) | 8 -8.44 (3.66) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | 5.63 (-4.86, 16.11)<br>-0.87 (-11.4, 9.61) |

OVERALL TREATMENT DIFFERENCE IS DERIVED USING ANCOVA MODEL, WITH TREATMENT AND CENTER AS MAIN EFFECT AND BASELINE VALUE AS COVARIATE; BY CENTER DIFFERENCES ARE DERIVED USING ANCOVA MODEL, WITH TREATMENT AND CENTER AS MAIN EFFECT, TREATMENT BY CENTER INTERACTION, AND BASELINE VALUE AS COVARIATE.

NOTE: FOR ANALYSIS PURPOSE, SMALL CENTERS ARE POOLED TOGETHER.

CENTANAFADINE

4 OF 4

# STAT-4.5.1 Summary of Mean Change at Day 42 from Baseline in AISRS Total Score By Center - LOCF (Efficacy Sample)

------

| | | _AISRS TOTAL SCORE | | |
|---|---|---|---|---|
| | CTN SR 200MG | CTN SR 400MG | PLACEBO TREATMENT | |
| CENTER | N LS MEAN (SE) | N LS MEAN (SE) | N LS MEAN (SE) COMPARISON | LS MEAN DIFFERENCE¹ |
| | 2 1.21 (7.28) | 1 -14.2 (10.3) | 1 -12.9 (10.3) CTN SR 200MG VS. PLAC<br>CTN SR 400MG VS. PLAC | |
| | 2 -12.5 (7.29) | 1 -1.36 (10.3) | 1 -10.5 (10.3) CTN SR 200MG VS. PLACI<br>CTN SR 400MG VS. PLACI | |
| | 1 -23.9 (10.3) | 1 -1.23 (10.3) | 2 -6.52 (7.31) CTN SR 200MG VS. PLAC<br>CTN SR 400MG VS. PLAC | |

NOTE: FOR ANALYSIS PURPOSE, SMALL CENTERS ARE POOLED TOGETHER.

OVERALL TREATMENT DIFFERENCE IS DERIVED USING ANCOVA MODEL, WITH TREATMENT AND CENTER AS MAIN EFFECT AND BASELINE VALUE AS COVARIATE; BY CENTER DIFFERENCES ARE DERIVED USING ANCOVA MODEL, WITH TREATMENT AND CENTER AS MAIN EFFECT, TREATMENT BY CENTER INTERACTION, AND BASELINE VALUE AS COVARIATE.


 ${\tt STAT-4.5.2}$  Differences in Unadjusted Mean Changes of AISRS Total Score at Day 42 Among Treatment Groups By Center - LOCF (Efficacy Sample)

| | | _CTN | SR 200M | CTN | SR 400MG | PI | ACEBO | CTN SR 200MG VS.<br>PLACEBO | CTN SR 400MG VS.<br>PLACEBO |
|---|---|---|---|---|---|---|---|---|---|
| CENTER | COUNTRY | N | MEAN <sup>1</sup> | N | MEAN <sup>1</sup> | N | MEAN¹ | DIFF <sup>2</sup> | DIFF <sup>2</sup> |
| | USA | 1 | 3.00 | 1 | -21.00 | 1 | -1.00 | 4.00 | -20.00 |
| | USA | 5 | -3.40 | 6 | -18.00 | 6 | -0.50 | -2.90 | -17.50 |
| | USA | 2 | -19.50 | 2 | -12.00 | | 2.00 | -21.50 | -14.00 |
| | USA | 4 | -11.00 | 3 | -13.00 | 3 | -0.33 | -10.67 | |
| | USA | 3 | 0.33 | 3 | -14.00 | 3 | -3.00 | 3.33 | -11.00 |
| | USA | 3 | -10.33 | 2 | -14.00 | 3 | -3.67 | -6.67 | -10.33 |
| | USA | 13 | -6.08 | | -11.38 | 12 | -2.33 | -3.74 | -9.05 |
| | USA | 2 | -2.50 | 2 | -9.50 | 1 | -1.00 | -1.50 | -8.50 |
| | USA | 4 | -9.00 | 2 | -9.00 | 4 | -0.75 | -8.25 | -8.25 |
| | USA | 9 | -8.22 | 8 | | 8 | -4.75 | -3.47 | -7.63 |
| | USA | 1 | -5.00 | 1 | -1.00 | 1 | 6.00 | -11.00 | -7.00 |
| | USA | 1 | -10.00 | 2 | -15.00 | 1 | -9.00 | -1.00 | -6.00 |
| | USA | 3 | -20.00 | 4 | -11.75 | 2 | -6.50 | -13.50 | -5.25 |
| | USA | 5 | -1.80 | 5 | -15.60 | 6 | -11.83 | 10.03 | -3.77 |
| | USA | 3 | -11.67 | 3 | -16.33 | 3 | -12.67 | 1.00 | -3.67 |
| | USA | 5 | -3.60 | 6 | -13.00 | 4 | -9.50 | 5.90 | -3.50 |
| | USA | 2 | -21.50 | 1 | -4.00 | 1 | -2.00 | -19.50 | -2.00 |
| | USA | 2 | -9.50 | 1 | -10.00 | 2 | -8.50 | -1.00 | -1.50 |
| | USA | 2 | 1.00 | 1 | -13.00 | 1 | -12.00 | 13.00 | -1.00 |
| | USA | 7 | -2.57 | 7 | -8.57 | 8 | -7.88 | 5.30 | -0.70 |
| | USA | 2 | -15.50 | 2 | -0.50 | 1 | 0.00 | -15.50 | -0.50 |
| | USA | 5 | -12.40 | 5 | -11.00 | 5 | -10.80 | -1.60 | -0.20 |

 $<sup>^{\</sup>scriptscriptstyle 1}$  MEAN CHANGE FROM BASELINE AT DAY 42 (LOCF).

 $<sup>^{2}</sup>$  DIFFERENCE IN MEAN CHANGES AT DAY 42 BETWEEN TWO TREATMENT GROUPS. NOTE: FOR ANALYSIS PURPOSE, SMALL CENTERS ARE POOLED TOGETHER.

CENTANAFADINE 2 OF 2 PROTOCOL 405-201-00013

 ${\tt STAT-4.5.2}$  Differences in Unadjusted Mean Changes of AISRS Total Score at Day 42 Among Treatment Groups By Center - LOCF (Efficacy Sample)

| CTN SR 400MG VS.<br>PLACEBO | CTN SR 200MG VS.<br>PLACEBO | ACEBO | PL | SR 400MG | CTN | SR 200M | _CTN | | |
|---|---|---|---|---|---|---|---|---|---|
| DIFF <sup>2</sup> | DIFF <sup>2</sup> | MEAN 1 | N | MEAN <sup>1</sup> | N | MEAN 1 | N | COUNTRY | TER |
| -0.20 | -12.14 | -15.42 | 12 | -15.62 | 13 | -27.56 | 9 | USA | |
| 0.17 | 10.17 | -17.67 | 3 | -17.50 | 2 | -7.50 | 2 | USA | |
| 1.66 | -8.00 | -7.29 | 7 | -5.63 | 8 | -15.29 | 7 | USA | |
| 2.30 | -7.88 | -6.30 | 10 | -4.00 | 11 | -14.18 | 11 | USA | |
| 3.00 | -27.00 | -3.00 | 1 | 0.00 | 1 | -30.00 | 2 | USA | |
| 4.00 | 31.00 | -28.00 | 1 | -24.00 | 1 | 3.00 | 1 | USA | |
| 4.00 | -8.50 | 1.00 | 2 | 5.00 | 1 | -7.50 | 2 | USA | |
| 4.33 | 2.58 | -12.33 | 3 | -8.00 | 4 | -9.75 | 4 | USA | |
| 4.38 | -1.59 | -6.13 | 8 | -1.75 | 8 | -7.71 | 7 | USA | |
| 4.50 | -1.00 | -14.00 | 2 | -9.50 | 2 | -15.00 | 1 | USA | |
| 4.50 | -17.50 | -5.50 | 2 | -1.00 | 1 | -23.00 | 1 | USA | |
| 5.17 | 5.33 | -9.17 | 6 | -4.00 | 6 | -3.83 | 6 | USA | |
| 5.50 | -1.00 | -2.00 | 2 | 3.50 | 2 | -3.00 | 2 | USA | |
| 8.08 | 5.33 | -15.33 | 3 | -7.25 | 4 | -10.00 | 3 | USA | |
| 8.17 | 8.33 | -16.67 | 3 | -8.50 | 2 | -8.33 | 3 | USA | |
| 9.00 | -1.00 | -11.00 | 1 | -2.00 | 1 | -12.00 | 2 | USA | |

CEM CD 200MC T/C CEM CD 400MC T/C

<sup>&</sup>lt;sup>1</sup> MEAN CHANGE FROM BASELINE AT DAY 42 (LOCF).

 $<sup>^{2}</sup>$  DIFFERENCE IN MEAN CHANGES AT DAY 42 BETWEEN TWO TREATMENT GROUPS. NOTE: FOR ANALYSIS PURPOSE, SMALL CENTERS ARE POOLED TOGETHER.

CENTANAFADINE 1 OF 24 PROTOCOL 405-201-00013

STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

## The TTEST Procedure

| | Va | riable: CHG | (Change | from Baseline | e) | |
|---|---|---|---|---|---|---|
| TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 1 | 143 | -5.9580 | 8.6959 | 0.7272 | -40.0000 | 8.0000 |
| 3 | 142 | -4.8169 | 7.2284 | 0.6066 | -32.0000 | 7.0000 |
| Diff | (1-2) | -1.1411 | 7.9985 | 0.9476 | | |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 1 | | -5.9580 | -7.3955 | -4.5205 | 8.6959 | 7.7914 9.8398 |
| 3 | | -4.8169 | -6.0161 | -3.6177 | 7.2284 | 6.4742 8.1831 |
| Diff (1-2) | Pooled | -1.1411 | -3.0063 | 0.7241 | 7.9985 | 7.3903 8.7165 |
| Diff (1-2) | Satterthwaite | -1.1411 | -3.0054 | 0.7231 | | |
| | Method | Variances | DI | t Value | Pr > t | |
| | Pooled | Equal | 283 | 3 -1.20 | 0.2295 | |
| | Satterthwaite | Unequal | 274.5 | 1 -1.21 | 0.2292 | |

CENTANAFADINE 2 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF

(Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Num DF Den DF F Value Pr > FMethod Folded F 142 141 1.45 0.0287

CENTANAFADINE 3 OF 24


## STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=14 ------

## The TTEST Procedure

| | Va | riable: CHG | (Change | from Baseline | ∍) | |
|---|---|---|---|---|---|---|
| TRTPN | N N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 1 | 147 | -7.7823 | 9.5684 | 0.7892 | -41.0000 | 7.0000 |
| 3 | 144 | -6.9167 | 8.7909 | 0.7326 | -36.0000 | 8.0000 |
| Diff | (1-2) | -0.8656 | 9.1919 | 1.0777 | | |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 1 | | -7.7823 | -9.3420 | -6.2226 | 9.5684 | 8.5855 10.8076 |
| 3 | | -6.9167 | -8.3647 | -5.4686 | 8.7909 | 7.8794 9.9427 |
| Diff (1-2) | Pooled | -0.8656 | -2.9869 | 1.2556 | 9.1919 | 8.4998 10.0078 |
| Diff (1-2) | Satterthwaite | -0.8656 | -2.9850 | 1.2537 | | |
| | Method | Variances | DI | F t Value | Pr > t | |
| | Pooled | Equal | 289 | 9 -0.80 | 0.4225 | |
| | Satterthwaite | Unequal | 287 83 | 2 -0.80 | 0 4221 | |

CENTANAFADINE 4 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 146 143 1.18 0.3099

CENTANAFADINE 5 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=21 ------

The TTEST Procedure

| | Vai | riable: CHG | (Change | from Baselin | e) | |
|---|---|---|---|---|---|---|
| TRTPN | ı N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 1 | 147 | -8.5714 | 9.5530 | 0.7879 | -40.0000 | 7.0000 |
| 3 | 144 | -6.9792 | 8.8929 | 0.7411 | -39.0000 | 7.0000 |
| Diff | (1-2) | -1.5923 | 9.2323 | 1.0825 | | |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 1 | | -8.5714 | -10.1286 | -7.0142 | 9.5530 | 8.5717 10.7901 |
| 3 | | -6.9792 | -8.4440 | -5.5143 | 8.8929 | 7.9708 10.0581 |
| Diff (1-2) | Pooled | -1.5923 | -3.7228 | 0.5383 | 9.2323 | 8.5371 10.0517 |
| Diff (1-2) | Satterthwaite | -1.5923 | -3.7212 | 0.5367 | | |
| | Method | Variance | s D | F t Value | Pr > t | |
| | Pooled | Equal | 28 | 9 -1.47 | 0.1424 | |
| | Cattorthuaito | IInogual | 200 2 | 5 _1 /7 | 0 1/21 | |

CENTANAFADINE 6 OF 24 PROTOCOL 405-201-00013

STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=21 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > FFolded F 146 143 1.15 0.3909

CENTANAFADINE 7 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=28 ------

The TTEST Procedure

| | | | Variable: | CHG (Chang | e from Bas | eline) | | |
|---|---|---|---|---|---|---|---|---|
| | TRTPN | N | Mean | n Std Dev | Std E | rr Minimum | Maximum | |
| | 1<br>3<br>Diff | 147<br>144<br>(1-2) | -9.5578<br>-6.8613<br>-2.696 | 9.5972 | 0.79 | 98 -50.0000 | | |
| TRTPN | | Method | Mea | an 95% | CL Mean | Std Dev | 95% CL S | td Dev |
| 1<br>3<br>Diff (1-<br>Diff (1- | , | Pooled<br>Satterthwait | -9.557<br>-6.863<br>-2.696<br>e -2.696 | -8.442<br>-5.109 | 7 -7.7270<br>0 -5.2802<br>4 -0.2840<br>7 -0.2877 | 9.5972 | 8.6021 | 12.6863<br>10.8547<br>11.3829 |
| | | Method | Var | iances | DF t V | alue Pr > t | t | |
| | | Pooled<br>Satterthw | Equa<br>aite Uneo | | | 2.20 0.028<br>2.20 0.028 | | |

CENTANAFADINE 8 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 146 143 1.37 0.0599

CENTANAFADINE 9 OF 24


## STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

......

------ Analysis Visit (N)=35 ------

## The TTEST Procedure

| | | | Var | riable: CF | HG (Change | from Baseline | e) | |
|---|---|---|---|---|---|---|---|---|
| | TRTPN | | N | Mean | Std Dev | Std Err | Minimum | Maximum |
| | 1<br>3<br>Diff | | | -10.0816<br>-7.5694<br>-2.5122 | 11.1358<br>10.1545<br>10.6616 | 0.9185<br>0.8462<br>1.2501 | -46.0000<br>-41.0000 | 7.0000<br>11.0000 |
| TRTPN | | Method | | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 1<br>3<br>Diff (1-<br>Diff (1- | , | Pooled<br>Satterthw | aite | -10.0816<br>-7.5694<br>-2.5122<br>-2.5122 | -4.9725 | -5.8967<br>-0.0518 | 11.1358<br>10.1545<br>10.6616 | 9.9919 12.5779<br>9.1016 11.4850<br>9.8587 11.6079 |
| | | Method | | Variano | ces DI | f t Value | Pr > t | |
| | | Pooled<br>Satter | thwaite | Equal<br>Unequal | 289<br>L 287.53 | | | |

CENTANAFADINE 10 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=35 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 146 143 1.20 0.2691

CENTANAFADINE 11 OF 24


## STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

......

## The TTEST Procedure

| | Va | riable: CHG | (Change | from Baselin | e) | | |
|---|---|---|---|---|---|---|---|
| TRTI | PN N | Mean | Std Dev | Std Err | Minimum | Maximum | 1 |
| 1<br>3<br>Difi | 147<br>144<br>£ (1-2) | -7.4583 | 11.8933<br>10.0960<br>11.0406 | 0.9809<br>0.8413<br>1.2945 | -47.0000<br>-50.0000 | 7.0000<br>9.0000 | |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL S | Std Dev |
| 1<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -9.9728<br>-7.4583<br>-2.5145<br>-2.5145 | -11.9115<br>-9.1214<br>-5.0623<br>-5.0582 | -8.0341<br>-5.7953<br>0.0334<br>0.0293 | 11.8933<br>10.0960<br>11.0406 | | 13.4335<br>11.4188<br>12.0205 |
| | Method | Variances | DI | F t Value | Pr > t | | |
| | Pooled<br>Satterthwaite | Equal<br>Unequal | 289<br>283.29 | | | | |

CENTANAFADINE 12 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=42 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 146 143 1.39 0.0500

CENTANAFADINE 13 OF 24


## STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=7 ------

## The TTEST Procedure

| | | Variable: CH | G (Change f | rom Baseline | e) | |
|---|---|---|---|---|---|---|
| TRI | PN 1 | N Mean | Std Dev | Std Err | Minimum | Maximum |
| 2<br>3<br>Di f | 14<br>14:<br>Ef (1-2) | | 7.1088<br>7.2284<br>7.1684 | 0.5924<br>0.6066<br>0.8478 | -29.0000<br>-32.0000 | 11.0000<br>7.0000 |
| TRTPN | Method | Mean | 95% CL | | Std Dev | 95% CL Std Dev |
| 2<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwai | -4.7569<br>-4.8169<br>0.0600<br>te 0.0600 | -5.9279<br>-6.0161<br>-1.6088<br>-1.6090 | 1.7287 | 7.1088<br>7.2284<br>7.1684 | 6.3717 8.0402<br>6.4742 8.1831<br>6.6243 7.8108 |
| | Method | Varianc | es DF | t Value | Pr > t | |
| | Pooled | Equal | 284 | | 0.9437 | |

CENTANAFADINE 14 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Num DF Den DF F Value Pr > FMethod Folded F 141 143 1.03 0.8423

CENTANAFADINE 15 OF 24


## STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

......

## The TTEST Procedure

| | Vai | riable: CHG | (Change | from Baselin | e) | |
|---|---|---|---|---|---|---|
| TRTE | PN N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 2<br>3<br>Diff | 147<br>144<br>f (1-2) | -7.2245<br>-6.9167<br>-0.3078 | 8.6395<br>8.7909<br>8.7147 | 0.7126<br>0.7326<br>1.0218 | -42.0000<br>-36.0000 | 11.0000 |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -7.2245<br>-6.9167<br>-0.3078<br>-0.3078 | -8.6328<br>-8.3647<br>-2.3189<br>-2.3193 | | 8.6395<br>8.7909<br>8.7147 | 7.7520 9.7583<br>7.8794 9.9427<br>8.0585 9.4882 |
| | Method | Variances | D | F t Value | Pr > t | |
| | Pooled<br>Satterthwaite | Equal<br>Unequal | 28<br>288.5 | | | |

CENTANAFADINE 16 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Num DF Den DF F Value Pr > FMethod Folded F 143 146 1.04 0.8344

CENTANAFADINE 17 OF 24


## STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

......

## The TTEST Procedure

| | Va | riable: CHG | (Change | from Baseline | ∍) | |
|---|---|---|---|---|---|---|
| TRTPN | N N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 2 | 147 | -8.6871 | 9.4643 | 0.7806 | -41.0000 | 10.0000 |
| 3 | 144 | -6.9792 | 8.8929 | 0.7411 | -39.0000 | 7.0000 |
| Diff | (1-2) | -1.7079 | 9.1860 | 1.0770 | | |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2 | | -8.6871 | -10.2298 | -7.1443 | 9.4643 | 8.4920 10.6899 |
| 3 | | -6.9792 | -8.4440 | -5.5143 | 8.8929 | 7.9708 10.0581 |
| Diff (1-2) | Pooled | -1.7079 | -3.8277 | 0.4119 | 9.1860 | 8.4943 10.0013 |
| Diff (1-2) | Satterthwaite | -1.7079 | -3.8264 | 0.4106 | | |
| | Method | Variances | D. | F t Value | Pr > t | |
| | Pooled | Equal | 28 | 9 -1.59 | 0.1139 | |
| | Satterthwaite | Unequal | 288. | 5 -1.59 | 0.1137 | |
CENTANAFADINE 18 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=21 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 146 143 1.13 0.4555

CENTANAFADINE 19 OF 24


# STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

......

# The TTEST Procedure

| | Vai | riable: CHG | (Change | from Baselin | e) | |
|---|---|---|---|---|---|---|
| TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 2<br>3<br>Diff | 147<br>144<br>(1-2) | -9.7143<br>-6.8611<br>-2.8532 | 10.6179<br>9.5972<br>10.1257 | 0.8757<br>0.7998<br>1.1872 | -41.0000<br>-50.0000 | 10.0000 |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -9.7143<br>-6.8611<br>-2.8532<br>-2.8532 | -11.4451<br>-8.4420<br>-5.1899<br>-5.1875 | -5.2802<br>-0.5165 | 10.6179<br>9.5972<br>10.1257 | 9.5272 11.9929<br>8.6021 10.8547<br>9.3632 11.0244 |
| | Method | Variance: | s DI | f t Value | Pr > t | |
| | Pooled<br>Satterthwaite | Equal<br>Unequal | 289<br>287.1 | | | |

CENTANAFADINE 20 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

(HITTOGOY DAMPIC)

------ Analysis Visit (N)=28 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 146 143 1.22 0.2260

CENTANAFADINE 21 OF 24


# STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=35 -----

# The TTEST Procedure

| | Va | riable: CHG | (Change | from Baseline | e) | |
|---|---|---|---|---|---|---|
| TRTPN | N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 2<br>3<br>Diff | 147<br>144<br>(1-2) | -7.5694 | 11.0094<br>10.1545<br>10.5950 | 0.9080<br>0.8462<br>1.2422 | -43.0000<br>-41.0000 | 10.0000 |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -7.5694 | -12.4273<br>-9.2421<br>-5.5082<br>-5.5062 | -0.6182 | 11.0094<br>10.1545<br>10.5950 | 9.8784 12.4351<br>9.1016 11.4850<br>9.7972 11.5354 |
| | Method | Variances | DI | t Value | Pr > t | |
| | Pooled<br>Satterthwaite | Equal<br>Unequal | 289<br>287.96 | | 0.0142<br>0.0142 | |

CENTANAFADINE 22 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=35 -------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Num DF Den DF F Value Pr > FMethod Folded F 146 143 1.18 0.3328

CENTANAFADINE 23 OF 24


# STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

......

# The TTEST Procedure

| | Va | riable: CHG | (Change | from Baseline | ∌) | |
|---|---|---|---|---|---|---|
| TRTPN | N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 2 | 147 | -9.8571 | 10.3633 | 0.8547 | -38.0000 | 10.0000 |
| 2 | 144 | -7.4583 | 10.0960 | 0.8413 | -50.0000 | 9.0000 |
| Diff | (1-2) | -2.3988 | 10.2319 | 1.1997 | | |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2 | | -9.8571 | -11.5464 | -8.1679 | 10.3633 | 9.2987 11.7053 |
| 3 | | -7.4583 | -9.1214 | -5.7953 | 10.0960 | 9.0492 11.4188 |
| Diff (1-2) | Pooled | -2.3988 | -4.7600 | -0.0376 | 10.2319 | 9.4614 11.1400 |
| Diff (1-2) | Satterthwaite | -2.3988 | -4.7594 | -0.0383 | | |
| | Method | Variances | DI | F t Value | Pr > t | |
| | Pooled | Equal | 289 | 9 -2.00 | 0.0465 | |
| | Cattorthuaite | IInogual | 200 00 | -2 00 | 0 0464 | |

CENTANAFADINE 24 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Num DF Den DF F Value Pr > FMethod Folded F 146 143 1.05 0.7543


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

# The TTEST Procedure

| | Va | riable: CHG | (Change | from Baselin | e) | | |
|---|---|---|---|---|---|---|---|
| TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| 1 | 143 | -5.9580 | 8.6959 | 0.7272 | -40.0000 | 8.0000 | |
| 3 | 142 | -4.8169 | 7.2284 | 0.6066 | -32.0000 | 7.0000 | |
| Diff | (1-2) | -1.1411 | 7.9985 | 0.9476 | | | |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std | Dev |
| 1 | | -5.9580 | -7.3955 | -4.5205 | 8.6959 | 7.7914 9 | .8398 |
| 3 | | -4.8169 | -6.0161 | -3.6177 | 7.2284 | 6.4742 8 | .1831 |
| Diff (1-2) | Pooled | -1.1411 | -3.0063 | 0.7241 | 7.9985 | 7.3903 8 | .7165 |
| Diff (1-2) | Satterthwaite | -1.1411 | -3.0054 | 0.7231 | | | |
| | Method | Variances | D | F t Value | Pr > t | | |
| | Pooled<br>Satterthwaite | Equal<br>Unequal | 28:<br>274.5 | | | | |

CENTANAFADINE

STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC

(Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 142 141 1.45 0.0287

CENTANAFADINE 3 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

......

The TTEST Procedure

| | Va | riable: CHG | (Change | from Baselin | e) | |
|---|---|---|---|---|---|---|
| TRT | PN N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 1<br>3<br>Dif | 133<br>136<br>f (1-2) | -7.9699<br>-7.0588<br>-0.9111 | 9.5932<br>8.9648<br>9.2808 | 0.8318<br>0.7687<br>1.1318 | -41.0000<br>-36.0000 | 7.0000<br>8.0000 |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 1<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -7.9699<br>-7.0588<br>-0.9111<br>-0.9111 | -9.6154<br>-8.5791<br>-3.1395<br>-3.1412 | -6.3245<br>-5.5385<br>1.3173<br>1.3190 | 9.5932<br>8.9648<br>9.2808 | 8.5624 10.9084<br>8.0111 10.1782<br>8.5559 10.1408 |
| | Method | Variances | D | F t Value | Pr > t | |
| | Pooled<br>Satterthwaite | Equal | 26<br>264 8 | | 0.4215 | |

CENTANAFADINE 4 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 132 135 1.15 0.4343

CENTANAFADINE 5 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=21 ------

The TTEST Procedure

| | Va | riable: CHG | (Change | from Baseline | e) | |
|---|---|---|---|---|---|---|
| TRTPN | N N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 1<br>3<br>Diff | 124<br>134<br>(1-2) | -8.8871<br>-7.2910<br>-1.5961 | 9.8346<br>9.1255<br>9.4728 | 0.8832<br>0.7883<br>1.1804 | -40.0000<br>-39.0000 | 4.0000 |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 1<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -8.8871<br>-7.2910<br>-1.5961<br>-1.5961 | -10.6353<br>-8.8503<br>-3.9206<br>-3.9276 | -7.1389<br>-5.7318<br>0.7285<br>0.7355 | 9.8346<br>9.1255<br>9.4728 | 8.7442 11.2381<br>8.1483 10.3713<br>8.7186 10.3711 |
| | Method | Variances | DI | F t Value | Pr > t | |
| | Pooled<br>Satterthwaite | Equal<br>Unequal | 250.2 | | | |


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

(Efficacy Sample

\_\_\_\_\_\_

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 123 133 1.16 0.3970

CENTANAFADINE 7 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

......

The TTEST Procedure

| | Va | ariable: CHG | (Change | from Baseline | e) | | |
|---|---|---|---|---|---|---|---|
| TRTP | N N | Mean S | Std Dev | Std Err | Minimum | Maximum | |
| 1<br>3<br>Diff | 117<br>129<br>(1-2) | -7.2093 | 11.9391<br>10.0122<br>10.9706 | 1.1038<br>0.8815<br>1.4006 | -47.0000<br>-50.0000 | 8.0000<br>10.0000 | |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std | Dev |
| 1<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -10.4444<br>-7.2093<br>-3.2351<br>-3.2351 | -5.9939 | -8.2583<br>-5.4650<br>-0.4764<br>-0.4517 | 11.9391<br>10.0122<br>10.9706 | 8.9216 11 | .7010<br>.4091<br>.0386 |
| | Method | Variances | DI | F t Value | Pr > t | | |
| | Pooled<br>Satterthwaite | Equal<br>Unequal | 244<br>227.35 | | | | |

CENTANAFADINE

STAT-4.7 Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

\_\_\_\_\_\_

------ Analysis Visit (N)=28 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 116 128 1.42 0.0522

CENTANAFADINE 9 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=35 ------

The TTEST Procedure

| | | 7 | Variable: CHG | (Change | from Baseline | ∍) | | |
|---|---|---|---|---|---|---|---|---|
| TRT | PN | N | Mean | Std Dev | Std Err | Minimum | Maximu | m |
| 1<br>3<br>Dif | | 113<br>122 | -8.1721 | 11.7975<br>10.4405<br>11.1135 | 1.1098<br>0.9452<br>1.4510 | -46.0000<br>-41.0000 | 6.000<br>11.000 | |
| TRTPN | Method | | Mean | 95% CL | Mean | Std Dev | 95% CL | Std Dev |
| 1<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthw | aite | | -13.0751<br>-10.0435<br>-5.5627<br>-5.5767 | -8.6771<br>-6.3008<br>0.1548<br>0.1688 | 11.7975<br>10.4405<br>11.1135 | 10.4342<br>9.2744<br>10.1895 | 13.5739<br>11.9445<br>12.2231 |
| | Method | | Variances | D: | F t Value | Pr > t | | |
| | Pooled<br>Satter | | Equal<br>te Unequal | 23<br>224.2 | | 0.0636<br>0.0649 | | |

CENTANAFADINE 10 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

......

------ Analysis Visit (N)=35 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 112 121 1.28 0.1875

CENTANAFADINE 11 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=42 -----

The TTEST Procedure

| | Vā | ariable: CHG | (Change | from Baseline | e) | | |
|---|---|---|---|---|---|---|---|
| TRTPN | N N | Mean S | Std Dev | Std Err | Minimum | Maximum | |
| 1<br>3<br>Diff | 109<br>119<br>(1-2) | -7.7815 | 12.9332<br>10.5358<br>11.7427 | 1.2388<br>0.9658<br>1.5569 | -47.0000<br>-50.0000 | 7.0000<br>9.0000 | |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Sto | d Dev |
| 1<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -10.8349<br>-7.7815<br>-3.0533<br>-3.0533 | -13.2903<br>-9.6941<br>-6.1212<br>-6.1500 | -8.3794<br>-5.8689<br>0.0145<br>0.0433 | 12.9332<br>10.5358<br>11.7427 | 9.3460 12 | 1.9218<br>2.0755<br>2.9350 |
| | Method | Variances | DI | f t Value | Pr > t | | |
| | Pooled<br>Satterthwaite | Equal<br>Unequal | 228.64 | | 0.0511<br>0.0533 | | |

CENTANAFADINE 12 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

\_\_\_\_\_

------ Analysis Visit (N)=42 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 108 118 1.51 0.0297

CENTANAFADINE 13 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

......

------ Analysis Visit (N)=7 ------

The TTEST Procedure

| | | | Va | riable: CHG | (Change | from Baseline | ∋) | | |
|---|---|---|---|---|---|---|---|---|---|
| | TRTPN | 1 | N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 2 | | 144 | -4.7569 | 7.1088 | 0.5924 | -29.0000 | 11.0000 | |
| | 3 | | 142 | -4.8169 | 7.2284 | 0.6066 | -32.0000 | 7.0000 | |
| | Diff | (1-2) | | 0.0600 | 7.1684 | 0.8478 | | | |
| TRT | PN | Method | | Mean | 95% CL | Mean | Std Dev | 95% CL S | td Dev |
| 2 | | | | -4.7569 | -5.9279 | -3.5860 | 7.1088 | 6.3717 | 8.0402 |
| 3 | | | | -4.8169 | -6.0161 | -3.6177 | 7.2284 | 6.4742 | 8.1831 |
| Dif | f (1-2) | Pooled | | 0.0600 | -1.6088 | 1.7287 | 7.1684 | 6.6243 | 7.8108 |
| Dif | f (1-2) | Satterth | waite | 0.0600 | -1.6090 | 1.7289 | | | |
| | | Metho | d | Variances | D | F t Value | Pr > t | | |
| | | Poole | d | Equal | 28 | 4 0.07 | 0.9437 | | |
| | | Satto | rthwaita | Unogual | 293 7 | 3 0 07 | 0 9/37 | | |

CENTANAFADINE 14 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 141 143 1.03 0.8423

CENTANAFADINE 15 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

| | | Variable: CHG | (Change | from Baselin | e) | |
|---|---|---|---|---|---|---|
| TRT | PN N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 2<br>3<br>Dif | 137<br>136<br>f (1-2) | -7.5985<br>-7.0588<br>-0.5397 | 8.7737<br>8.9648<br>8.8694 | 0.7496<br>0.7687<br>1.0736 | -42.0000<br>-36.0000 | 11.0000 |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -7.5985<br>-7.0588<br>-0.5397<br>-0.5397 | -9.0809<br>-8.5791<br>-2.6534<br>-2.6536 | -6.1162<br>-5.5385<br>1.5740<br>1.5741 | 8.7737<br>8.9648<br>8.8694 | 7.8434 9.9563<br>8.0111 10.1782<br>8.1814 9.6847 |
| | Method | Variances | D | F t Value | Pr > t | |
| | Pooled<br>Satterthwai | Equal<br>te Unequal | 27<br>270.7 | | | |

CENTANAFADINE 16 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=14 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 135 136 1.04 0.8022

CENTANAFADINE 17 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=21 ------

The TTEST Procedure

| | Va | riable: CHG | (Change | from Baseline | e) | |
|---|---|---|---|---|---|---|
| TRTPN | N | Mean S | Std Dev | Std Err | Minimum | Maximum |
| 2 | 133 | -9.0902 | 9.5691 | 0.8297 | -41.0000 | 10.0000 |
| 3<br>Diff | 134 | -7.2910<br>-1.7992 | 9.1255<br>9.3491 | 0.7883<br>1.1443 | -39.0000 | 7.0000 |
| DIII | (1 2) | 1.7552 | J.J.J. | 1.1113 | | |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2 | | -9.0902 - | -10.7315 | -7.4489 | 9.5691 | 8.5409 10.8810 |
| 3 | | -7.2910 | -8.8503 | -5.7318 | 9.1255 | 8.1483 10.3713 |
| Diff (1-2) | Pooled | -1.7992 | -4.0523 | 0.4539 | 9.3491 | 8.6164 10.2191 |
| Diff (1-2) | Satterthwaite | -1.7992 | -4.0527 | 0.4544 | | |
| | Method | Variances | DI | F t Value | Pr > t | |
| | Pooled | Equal | 26 | 5 -1.57 | 0.1171 | |
| | Satterthwaite | Unequal | 264.2 | 2 -1.57 | 0.1171 | |

CENTANAFADINE 18 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=21 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > FFolded F 132 133 1.10 0.5855

CENTANAFADINE 19 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

| | Va | riable: CHG | (Change | from Baselin | e) | |
|---|---|---|---|---|---|---|
| TRTPN | N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 2<br>3<br>Diff | 129 | -7.2093 | 10.9092<br>10.0122<br>10.4614 | 0.9797<br>0.8815<br>1.3157 | -41.0000<br>-50.0000 | 10.0000 |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -10.6452<br>-7.2093<br>-3.4359<br>-3.4359 | | -5.4650<br>-0.8447 | 10.9092<br>10.0122<br>10.4614 | 9.6997 12.4662<br>8.9216 11.4091<br>9.6208 11.4642 |
| | Method | Variances | DI | F t Value | Pr > t | |
| | Pooled<br>Satterthwaite | Equal<br>Unequal | 253<br>247.13 | | | |

CENTANAFADINE 20 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

\_\_\_\_\_

------ Analysis Visit (N)=28 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 123 128 1.19 0.3369

CENTANAFADINE 21 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

......

The TTEST Procedure

| | | | Variable: CHG | (Change f | rom Baseline | ≘) | |
|---|---|---|---|---|---|---|---|
| | TRTPN | N | Mean | Std Dev | Std Err | Minimum | Maximum |
| | 2<br>3<br>Diff | 114<br>122<br>(1-2) | -8.1721 | 11.1993<br>10.4405<br>10.8136 | 1.0489<br>0.9452<br>1.4086 | -43.0000<br>-41.0000 | 10.0000<br>11.0000 |
| TRTPN | | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2<br>3<br>Diff (1-<br>Diff (1- | | Pooled<br>Satterthwaite | -8.1721<br>-3.8542 | | | 11.1993<br>10.4405<br>10.8136 | 9.9101 12.8770<br>9.2744 11.9445<br>9.9163 11.8907 |
| | | Method | Variances | DF | t Value | Pr > t | |
| | | Pooled<br>Satterthwa | Equal<br>ite Unequal | 234<br>229.63 | | 0.0067<br>0.0068 | |

CENTANAFADINE 22 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=35 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 113 121 1.15 0.4477

CENTANAFADINE 23 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

| | Vā | ariable: CHG | (Change | from Baseline | e) | |
|---|---|---|---|---|---|---|
| TRTPN | N N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 2<br>3<br>Diff | 119<br>119<br>(1-2) | -7.7815 | 10.6276<br>10.5358<br>10.5818 | 0.9742<br>0.9658<br>1.3718 | -38.0000<br>-50.0000 | 10.0000 9.0000 |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -10.8908<br>-7.7815<br>-3.1092<br>-3.1092 | | -5.8689<br>-0.4066 | 10.6276<br>10.5358<br>10.5818 | 9.4274 12.1807<br>9.3460 12.0755<br>9.7072 11.6310 |
| | Method | Variances | DI | F t Value | Pr > t | |
| | Pooled<br>Satterthwaite | Equal<br>Unequal | 236<br>235.98 | | 0.0243<br>0.0243 | |

CENTANAFADINE 24 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

\_\_\_\_\_\_

------ Analysis Visit (N)=42 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 118 118 1.02 0.9251


STAT-4.8

Non-Parametric Stratified by Center Analysis of Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=7 ------

The FREQ Procedure

Summary Statistics for TRTP by CHG Controlling for POOLCNTR

Cochran-Mantel-Haenszel Statistics (Based on Rank Scores)

| Statistic | Alternative Hypothesis | DF | Value | Prob |
|-----------|------------------------|----|--------|--------|
| 1 | Nonzero Correlation | 1 | 1.0718 | 0.3005 |
| 2 | Row Mean Scores Differ | 2 | 1.7562 | 0.4156 |

<sup>1</sup> WILCOXON TEST STRATIFIED BY (POOLED) CENTER.


STAT-4.8

Non-Parametric Stratified by Center Analysis of Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The FREQ Procedure

Summary Statistics for TRTP by CHG Controlling for POOLCNTR

Cochran-Mantel-Haenszel Statistics (Based on Rank Scores)

| Statistic | Alternative Hypothesis | DF | Value | Prob |
|-----------|------------------------|----|--------|--------|
| 1 | Nonzero Correlation | 1 | 0.7626 | 0.3825 |
| 2 | Row Mean Scores Differ | 2 | 1.6961 | 0.4283 |

<sup>1</sup> WILCOXON TEST STRATIFIED BY (POOLED) CENTER.


STAT-4.8

Non-Parametric Stratified by Center Analysis of Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=21 ------

The FREQ Procedure

Summary Statistics for TRTP by CHG
Controlling for POOLCNTR

Cochran-Mantel-Haenszel Statistics (Based on Rank Scores)

| Statistic | Alternative Hypothesis | DF | Value | Prob |
|-----------|------------------------|----|--------|--------|
| 1 | Nonzero Correlation | 1 | 1.0930 | 0.2958 |
| 2 | Row Mean Scores Differ | 2 | 1 6783 | 0 4321 |

<sup>1</sup> WILCOXON TEST STRATIFIED BY (POOLED) CENTER.


STAT-4.8

Non-Parametric Stratified by Center Analysis of Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=28 ------

The FREQ Procedure

Summary Statistics for TRTP by CHG Controlling for POOLCNTR

Cochran-Mantel-Haenszel Statistics (Based on Rank Scores)

| Statistic | Alternative Hypothesis | DF | Value | Prob |
|-----------|------------------------|----|--------|--------|
| 1 | Nonzero Correlation | 1 | 3.4385 | 0.0637 |
| 2 | Row Mean Scores Differ | 2 | 5.1565 | 0.0759 |

<sup>1</sup> WILCOXON TEST STRATIFIED BY (POOLED) CENTER.


STAT-4.8

Non-Parametric Stratified by Center Analysis of Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=35 ------

The FREQ Procedure

Summary Statistics for TRTP by CHG Controlling for POOLCNTR

Cochran-Mantel-Haenszel Statistics (Based on Rank Scores)

| Statistic | Alternative Hypothesis | DF | Value | Prob |
|-----------|------------------------|----|--------|--------|
| 1 | Nonzero Correlation | 1 | 3.8708 | 0.0491 |
| 2 | Row Mean Scores Differ | 2 | 6 2158 | 0 0447 |

<sup>1</sup> WILCOXON TEST STRATIFIED BY (POOLED) CENTER.

STAT-4.8

Non-Parametric Stratified by Center Analysis of Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=42 ------

The FREQ Procedure

Summary Statistics for TRTP by CHG Controlling for POOLCNTR

Cochran-Mantel-Haenszel Statistics (Based on Rank Scores)

| Statistic | Alternative Hypothesis | DF | Value | Prob |
|-----------|------------------------|----|--------|--------|
| 1 | Nonzero Correlation | 1 | 3.0224 | 0.0821 |
| 2 | Row Mean Scores Differ | 2 | 3 9747 | 0 1371 |

\_\_\_\_\_\_

<sup>1</sup> WILCOXON TEST STRATIFIED BY (POOLED) CENTER.

CENTANAFADINE 1 OF 9 PROTOCOL 405-201-00013

STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure
Variable: RESID (Residual)
AVISITN = 42
AVISIT = DAY 42

#### Moments

| N | 347 | Sum Weights | 347 |
|-----------------|------------|------------------|------------|
| Mean | -0.3635827 | Sum Observations | -126.16319 |
| Std Deviation | 10.8189753 | Variance | 117.050226 |
| Skewness | -0.8029258 | Kurtosis | 0.15184193 |
| Uncorrected SS | 40545.2491 | Corrected SS | 40499.3783 |
| Coeff Variation | -2975.6575 | Std Error Mean | 0.58079302 |

# Basic Statistical Measures

| Location | Variabilitv |
|----------|-------------|

| Mean | -0.36358 | Std Deviation | 10.81898 |
|--------|----------|---------------------|-----------|
| Median | 1.86002 | Variance | 117.05023 |
| Mode | 0.60473 | Range | 53.83629 |
| | | Interguartile Range | 14.88131 |

Note: The mode displayed is the smallest of 4 modes with a count of 2.

CENTANAFADINE 2 OF 9


STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure
Variable: RESID (Residual)
 AVISITN = 42
 AVISIT = DAY 42

Tests for Location: Mu0=0

| Test | -Statistic- | p Value |
|---|---|---|
| Student's t<br>Sign<br>Signed Rank | t -0.62601<br>M 28.5<br>S 1596 | Pr > t 0.5317<br>Pr >= M 0.0026<br>Pr >= S 0.3942 |
| orgined hallh | 5 1330 | 11 /- 0 0.3342 |

Quantiles (Definition 5)

| Level | Quantile |
|------------|-----------|
| 100% Max | 19.94892 |
| 99% | 17.59826 |
| 95% | 13.42180 |
| 90% | 11.14587 |
| 75% Q3 | 7.91676 |
| 50% Median | 1.86002 |
| 25% O1 | -6.96455 |
| 10% | -15.95262 |
| 5% | -21.57855 |
| 1% | -31.78702 |
| 0% Min | -33.88736 |

CENTANAFADINE 3 OF 9 PROTOCOL 405-201-00013

STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure
Variable: RESID (Residual)

AVISITN = 42

AVISIT = DAY 42

# Extreme Observations

| | Lowe | st | High | est | | | |
|---|---|---|---|---|---|---|---|
| | Value | Obs | Value | Obs | | | |
| | -33.8874 | 1677 | 16.6970 | 714 | | | |
| | -33.3787 | 1554 | 17.5983 | 1295 | | | |
| | -33.1571 | 411 | 18.8332 | 2204 | | | |
| | -31.7870 | 1798 | 19.4803 | 2243 | | | |
| | -28.1267 | 1406 | 19.9489 | 1355 | | | |
| Histogram | # | Boxplot | | | Normal Probabi | lity Plot | |
| 17.5+**** | 9 | Ī | | 17.5+ | | _ | ++++ ***** |
| ********** | 45 | | | 1 | | *** | ***** |
| .********* | 76 | ++ | | 1 | | ***** | |
| .******** | 72 | ** | | 1 | **** | *+ | |
| .********** | 46 | + | | 1 | ****++ | | |
| -7.5+********* | 30 | ++ | | -7.5+ | ***+ | | |
| .******* | 29 | | | 1 | +*** | | |
| .****** | 18 | | | 1 | +++*** | | |
| ***** | 12 | | | - | +++*** | | |
| .*** | 6 | | | +++ | *** | | |
| -32.5+** | 4 | 0 | | -32.5+*** | | | |
| +++++++ | | | | + | ++ | ++ | ++ |
| * may represent up to 2 counts | | | | | -2 -1 0 | +1 | +2 |

CENTANAFADINE 4 OF 9


STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

AVISITN = 42 AVISIT = DAY 42

# Moments

| N | 347 | Sum Weights | 347 |
|-----------------|------------|------------------|------------|
| Mean | -0.0353861 | Sum Observations | -12.278976 |
| Std Deviation | 1.02339086 | Variance | 1.04732886 |
| Skewness | -0.8014075 | Kurtosis | 0.14366209 |
| Uncorrected SS | 362.810289 | Corrected SS | 362.375784 |
| Coeff Variation | -2892.0705 | Std Error Mean | 0.0549385 |

# Basic Statistical Measures

# Location Variability

| Mean | -0.03539 | Std Deviation | 1.02339 |
|--------|----------|---------------------|---------|
| Median | 0.17390 | Variance | 1.04733 |
| Mode | 0.05664 | Range | 5.12952 |
| | | Interquartile Range | 1.41016 |

Note: The mode displayed is the smallest of 4 modes with a count of 2.

CENTANAFADINE 5 OF 9


STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

AVISITN = 42 AVISIT = DAY 42

Tests for Location: Mu0=0

| Test | -St | atistic- | p Valı | ıe |
|-------------|-----|----------|----------|--------|
| Student's t | t | -0.6441 | Pr > t | 0.5199 |
| Sign | M | 28.5 | Pr >= M | 0.0026 |
| Signed Rank | S | 1567 | Pr >= S | 0.4028 |

Quantiles (Definition 5)

| Level | Quantile |
|---------------|-----------|
| 100% Max | 1.902521 |
| 99% | 1.671961 |
| 95% | 1.269575 |
| 90%<br>75% Q3 | 1.049981 |
| 50% Median | 0.173896 |
| 25% Q1 | -0.660998 |
| 10% | -1.496158 |
| 5% | -2.066916 |
| 1% | -2.976287 |
| 0% Min | -3.227003 |

CENTANAFADINE 6 OF 9


STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure
Variable: STUDENTRESID (Studentized Residual)
AVISITN = 42
AVISIT = DAY 42

# Extreme Observations

| Lowes | st | Highest | |
|----------------------|--------------|--------------------|--------------|
| Value | Obs | Value | Obs |
| -3.22700<br>-3.14078 | 1677<br>1554 | 1.65677<br>1.67196 | 1295<br>714 |
| -3.10521<br>-2.97629 | 411<br>1798 | 1.76566<br>1.82508 | 2204<br>2243 |
| -2 70089 | 1406 | 1 90252 | 1355 |

CENTANAFADINE 7 OF 9 PROTOCOL 405-201-00013

STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

| | | The UNIVARIATE Pro | cedure | |
|---|---|---|---|---|
| | Variable: | STUDENTRESID (Stude | entized Residual) | |
| | | AVISITN = 42 | | |
| | | AVISIT = DAY 4 | 2 | |
| Leaf | # | Boxplot | | Normal Probability Plot |
| 30 | 2 | Ī | 1.9+ | ++ * |
| 677 | 3 | 1 | 1 | ++ *** |
| 5711 | 4 | 1 | 1 | + ** |
| 16777700777 | 11 | 1 | 1 | ++ *** |
| 00011123555667711666789 | 23 | 1 | 1 | +**** |
| 000012566777889000112344555555666778 | 36 | 1 | 1 | **** |
| 00011222333445566778899112222355556788 | 38 | ++ | 1 | **** |
| 111122344588889111466899 | 24 | 1 1 | I | ***++ |
| 0134556677888999044555666788888 | 31 | 1 1 | 1 | ***++ |
| 111223345666677900122445556779 | 30 | ** | 1 | ***++ |
| 9753329887665443322 | 19 | + | 1 | **++ |
| 977654111998877631 | 18 | I I | 1 | **++ |
| 99855427665543000 | 17 | I I | 1 | **+ |
| 88652998765321 | 14 | ++ | -0.7+ | *** |
| 86541766431 | 11 | 1 | 1 | ** |
| 8755332865333 | 13 | 1 | 1 | +** |
| 76407765541 | 11 | 1 | 1 | +*** |
| 3007666310 | 10 | 1 | 1 | ++** |
| 985100642 | 9 | 1 | 1 | ++** |
| 977 | 3 | 1 | + | + ** |
| 4418720 | 7 | 1 | ++ | *** |
| 7865 | 4 | 1 | ++ * | * |
| 105 | 3 | į | ++ ** | |
| 03 | 2 | ĺ | ** | |
| 8 | 1 | 0 | * | |
| 41 | 2 | 0 | * * | |
| | Leaf 30 677 5711 16777700777 00011123555667711666789 000012566777889000112344555555666778 00011222333445566778899112222355556788 11122344588889111466899 0134556677888999044555666788888 111223345666677900122445556779 9753329887665443322 977654111998877631 99855427665543000 88652998765321 86541766431 8755332865333 76407765541 3007666310 985100642 977 4418720 7865 105 03 8 41 | Leaf # 30 | Variable: STUDENTRESID (Stude AVISITN = 42 AVISITN = 42 AVISITN = 42 AVISITN = 42 AVISITN = 42 AVISIT = DAY 4 Leaf | Leaf |

| The UNIVARIATE Procedure | |
|---|---|
| Variable: STUDENTRESID (Studentized Residual) AVISITN = 42 AVISIT = DAY 42 | |
| -32 3 1 0 -3.3+*++ | + |

CENTANAFADINE 9 OF 9

STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)





CENTANAFADINE 1 OF 26 PROTOCOL 405-201-00013

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

# The Mixed Procedure

#### Model Information

Data Set WORK.INDATA
Dependent Variable CHG
Covariance Structure Unstructured
Subject Effect SUBJID
Group Effect TRTFN
Estimation Method REML
Residual Variance Method None
Fixed Effects SE Method Kenward-Roger

Fixed Effects SE Method Kenward-Roger
Degrees of Freedom Method Kenward-Roger

# Class Level Information

| Class | Levels | Values |
|------------------------------|--------------|---------------------------|
| AVISITN<br>TRTPN<br>POOLCNTR | 6<br>3<br>38 | 7 14 21 28 35 42<br>1 2 3 |

CENTANAFADINE 2 OF 26 PROTOCOL 405-201-00013

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

The Mixed Procedure

Class Level Information

Class Levels Values
SUBJID 438

CENTANAFADINE 3 OF 26 PROTOCOL 405-201-00013

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure



CENTANAFADINE 4 OF 26 PROTOCOL 405-201-00013

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

The Mixed Procedure



CENTANAFADINE 5 OF 26 PROTOCOL 405-201-00013

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

The Mixed Procedure



CENTANAFADINE 6 OF 26 PROTOCOL 405-201-00013

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

......

The Mixed Procedure



CENTANAFADINE 7 OF 26 PROTOCOL 405-201-00013

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

#### The Mixed Procedure



#### Dimensions

| Covariance | Parameters | 63 |
|------------|------------|-----|
| Columns in | X | 72 |
| Columns in | Z | 0 |
| Subjects | | 438 |
| Max Obs pe | r Subiect | 6 |

#### Number of Observations

| Number | of | Observations | Read | 2292 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 2292 |
| Number | of | Observations | Not Used | 0 |

CENTANAFADINE


8 OF 26

# STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

#### The Mixed Procedure

#### Iteration History

| Iterati | on 1 | Evaluations | -2 Res Log Like | Criterion |
|---------|------|-------------|-----------------|------------|
| | 0 | 1 | 16529.25629156 | |
| | 1 | 2 | 14188.42661779 | 0.00057908 |
| | 2 | 1 | 14185.23002848 | 0.00001628 |
| | 3 | 1 | 14185.14601175 | 0.00000002 |
| | 4 | 1 | 14185.14589278 | 0.00000000 |

Convergence criteria met.

| | | Estimated 1 | R Matrix for | SUBJID | | |
|-----|---------|-------------|--------------|---------|---------|---------|
| Row | Col1 | Co12 | Col3 | Col4 | Co15 | Col6 |
| 1 | 46.0381 | 41.1715 | 36.7487 | 32.9053 | 36.5459 | 38.5770 |
| 2 | 41.1715 | 72.3189 | 63.2366 | 57.9165 | 61.0600 | 61.5916 |
| 3 | 36.7487 | 63.2366 | 85.0775 | 79.2283 | 82.7270 | 77.0389 |
| 4 | 32.9053 | 57.9165 | 79.2283 | 109.98 | 96.5075 | 92.0782 |
| 5 | 36.5459 | 61.0600 | 82.7270 | 96.5075 | 108.06 | 90.3451 |
| 6 | 38.5770 | 61.5916 | 77.0389 | 92.0782 | 90.3451 | 107.13 |

CENTANAFADINE 9 OF 26 PROTOCOL 405-201-00013

STAT-4.10
Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups
(Efficacy Sample)

#### The Mixed Procedure

| | | The | e Mixed Proce | edure | | |
|---|---|---|---|---|---|---|
| | Estima | ated R Corre | lation Matrix | for SUBJID | | |
| Row | Col1 | Col2 | Col3 | Col4 | Col5 | Col6 |
| 1 | 1.0000 | 0.7135 | 0.5872 | 0.4624 | 0.5182 | 0.5493 |
| 2 | 0.7135 | 1.0000 | 0.8062 | 0.6494 | 0.6907 | 0.6997 |
| 3 | 0.5872 | 0.8062 | 1.0000 | 0.8191 | 0.8628 | 0.8069 |
| 4 | 0.4624 | 0.6494 | 0.8191 | 1.0000 | 0.8853 | 0.8483 |
| 5 | 0.5182 | 0.6907 | 0.8628 | 0.8853 | 1.0000 | 0.8397 |
| 6 | 0.5493 | 0.6997 | 0.8069 | 0.8483 | 0.8397 | 1.0000 |
| | | Estimated R | Matrix for S | SUBJID | | |
| Row | Col1 | Col2 | Col3 | Col4 | Col5 | Col6 |
| 1 | 65.6662 | 44.0115 | 46.3127 | 47.7634 | 47.6829 | 43.0330 |
| 2 | 44.0115 | 78.8090 | 65.0532 | 70.3450 | 71.8874 | 74.0759 |
| 3 | 46.3127 | 65.0532 | 84.1997 | 82.8999 | 84.5571 | 87.9428 |
| 4 | 47.7634 | 70.3450 | 82.8999 | 117.91 | 107.76 | 115.71 |
| 5 | 47.6829 | 71.8874 | 84.5571 | 107.76 | 118.69 | 119.10 |
| 6 | 43.0330 | 74.0759 | 87.9428 | 115.71 | 119.10 | 146.06 |

CENTANAFADINE 10 OF 26 PROTOCOL 405-201-00013

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

#### The Mixed Procedure

| | | Estimated F | Matrix for | SUBJID | | |
|-----|---------|-------------|------------|---------|---------|---------|
| Row | Col1 | Col2 | Col3 | Col4 | Col5 | Col6 |
| 1 | 46.3693 | 34.8314 | 31.0449 | 30.9025 | 30.4290 | 32.7595 |
| 2 | 34.8314 | 65.0980 | 57.0928 | 58.3247 | 56.0968 | 55.8943 |
| 3 | 31.0449 | 57.0928 | 73.8230 | 68.5633 | 73.5792 | 69.9148 |
| 4 | 30.9025 | 58.3247 | 68.5633 | 88.3257 | 83.0181 | 81.2208 |
| 5 | 30.4290 | 56.0968 | 73.5792 | 83.0181 | 104.07 | 88.0138 |
| 6 | 32.7595 | 55.8943 | 69.9148 | 81.2208 | 88.0138 | 99.0964 |

#### Covariance Parameter Estimates

| Cov Parm | Subject | Group | Estimate |
|----------|---------|---------|----------|
| UN(1,1) | SUBJID | TRTPN 1 | 65.6662 |
| UN(2,1) | SUBJID | TRTPN 1 | 44.0115 |
| UN(2,2) | SUBJID | TRTPN 1 | 78.8090 |
| UN(3,1) | SUBJID | TRTPN 1 | 46.3127 |
| UN(3,2) | SUBJID | TRTPN 1 | 65.0532 |
| UN(3,3) | SUBJID | TRTPN 1 | 84.1997 |
| UN(4,1) | SUBJID | TRTPN 1 | 47.7634 |
| UN(4,2) | SUBJID | TRTPN 1 | 70.3450 |
| UN(4,3) | SUBJID | TRTPN 1 | 82.8999 |
| UN (4,4) | SUBJID | TRTPN 1 | 117.91 |
| UN(5,1) | SUBJID | TRTPN 1 | 47.6829 |
| UN(5,2) | SUBJID | TRTPN 1 | 71.8874 |

CENTANAFADINE 11 OF 26 PROTOCOL 405-201-00013

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm | Subject | Group | Estimate |
|----------|---------|---------|----------|
| UN(5,3) | SUBJID | TRTPN 1 | 84.5571 |
| UN(5,4) | SUBJID | TRTPN 1 | 107.76 |
| UN(5,5) | SUBJID | TRTPN 1 | 118.69 |
| UN(6,1) | SUBJID | TRTPN 1 | 43.0330 |
| UN(6,2) | SUBJID | TRTPN 1 | 74.0759 |
| UN(6,3) | SUBJID | TRTPN 1 | 87.9428 |
| UN(6,4) | SUBJID | TRTPN 1 | 115.71 |
| UN(6,5) | SUBJID | TRTPN 1 | 119.10 |
| UN(6,6) | SUBJID | TRTPN 1 | 146.06 |
| UN(1,1) | SUBJID | TRTPN 2 | 46.0381 |
| UN(2,1) | SUBJID | TRTPN 2 | 41.1715 |
| UN(2,2) | SUBJID | TRTPN 2 | 72.3189 |
| UN(3,1) | SUBJID | TRTPN 2 | 36.7487 |
| UN(3,2) | SUBJID | TRTPN 2 | 63.2366 |
| UN(3,3) | SUBJID | TRTPN 2 | 85.0775 |
| UN(4,1) | SUBJID | TRTPN 2 | 32.9053 |
| UN(4,2) | SUBJID | TRTPN 2 | 57.9165 |
| UN(4,3) | SUBJID | TRTPN 2 | 79.2283 |
| UN (4,4) | SUBJID | TRTPN 2 | 109.98 |
| UN(5,1) | SUBJID | TRTPN 2 | 36.5459 |
| UN(5,2) | SUBJID | TRTPN 2 | 61.0600 |
| UN(5,3) | SUBJID | TRTPN 2 | 82.7270 |
| UN (5,4) | SUBJID | TRTPN 2 | 96.5075 |
| UN(5,5) | SUBJID | TRTPN 2 | 108.06 |

CENTANAFADINE 12 OF 26 PROTOCOL 405-201-00013

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm | Subject | Group | Estimate |
|----------|---------|---------|----------|
| UN(6,1) | SUBJID | TRTPN 2 | 38.5770 |
| UN(6,2) | SUBJID | TRTPN 2 | 61.5916 |
| UN(6,3) | SUBJID | TRTPN 2 | 77.0389 |
| UN(6,4) | SUBJID | TRTPN 2 | 92.0782 |
| UN(6,5) | SUBJID | TRTPN 2 | 90.3451 |
| UN(6,6) | SUBJID | TRTPN 2 | 107.13 |
| UN(1,1) | SUBJID | TRTPN 3 | 46.3693 |
| UN(2,1) | SUBJID | TRTPN 3 | 34.8314 |
| UN(2,2) | SUBJID | TRTPN 3 | 65.0980 |
| UN(3,1) | SUBJID | TRTPN 3 | 31.0449 |
| UN(3,2) | SUBJID | TRTPN 3 | 57.0928 |
| UN(3,3) | SUBJID | TRTPN 3 | 73.8230 |
| UN(4,1) | SUBJID | TRTPN 3 | 30.9025 |
| UN(4,2) | SUBJID | TRTPN 3 | 58.3247 |
| UN(4,3) | SUBJID | TRTPN 3 | 68.5633 |
| UN (4,4) | SUBJID | TRTPN 3 | 88.3257 |
| UN(5,1) | SUBJID | TRTPN 3 | 30.4290 |
| UN(5,2) | SUBJID | TRTPN 3 | 56.0968 |
| UN(5,3) | SUBJID | TRTPN 3 | 73.5792 |
| UN (5,4) | SUBJID | TRTPN 3 | 83.0181 |
| UN(5,5) | SUBJID | TRTPN 3 | 104.07 |
| UN(6,1) | SUBJID | TRTPN 3 | 32.7595 |
| UN(6,2) | SUBJID | TRTPN 3 | 55.8943 |
| UN(6,3) | SUBJID | TRTPN 3 | 69.9148 |

CENTANAFADINE 13 OF 26 PROTOCOL 405-201-00013

# STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

......

The Mixed Procedure

#### Covariance Parameter Estimates

| Cov Parm | Subject | Group | Estimate |
|----------|---------|---------|----------|
| UN(6,4) | SUBJID | TRTPN 3 | 81.2208 |
| UN(6,5) | SUBJID | TRTPN 3 | 88.0138 |
| UN(6,6) | SUBJID | TRTPN 3 | 99.0964 |

# Fit Statistics

| -2 Res Log Likelihood | 14185.1 |
|--------------------------|---------|
| AIC (Smaller is Better) | 14311.1 |
| AICC (Smaller is Better) | 14314.9 |
| BIC (Smaller is Better) | 14568.3 |

# Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 62 | 2344.11 | < .0001 |

CENTANAFADINE 14 OF 26


# STAT-4.10 Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

\_\_\_\_\_

# The Mixed Procedure

# Solution for Fixed Effects

| <b>7</b> 66 | Pooled<br>Center | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Number | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| Intercept | | | | 0.4124 | 4.8142 | 479 | 0.09 | 0.9318 |
| AVISITN | | 7 | | -0.8831 | 2.8978 | 372 | -0.30 | 0.7607 |
| AVISITN | | 14 | | -0.7454 | 2.4446 | 354 | -0.30 | 0.7606 |
| AVISITN | | 21 | | -2.9398 | 2.0177 | 326 | -1.46 | 0.1461 |
| AVISITN | | 28 | | 2.5080 | 1.7494 | 323 | 1.43 | 0.1526 |
| AVISITN | | 35 | | 0.3320 | 1.7659 | 337 | 0.19 | 0.8510 |
| AVISITN | | 42 | | 0 | | | | |
| TRTPN | | | 1 | -3.0330 | 1.3769 | 249 | -2.20 | 0.0285 |
| TRTPN | | | 2 | -2.7565 | 1.2456 | 260 | -2.21 | 0.0278 |
| TRTPN | | | 3 | 0 | | | | |
| AVISITN*TRTPN | | 7 | 1 | 1.7304 | 1.2761 | 241 | 1.36 | 0.1764 |
| AVISITN*TRTPN | | 7 | 2 | 2.8863 | 1.0986 | 274 | 2.63 | 0.0091 |
| AVISITN*TRTPN | | 7 | 3 | 0 | | | | |
| AVISITN*TRTPN | | 14 | 1 | 2.0397 | 1.0425 | 235 | 1.96 | 0.0516 |
| AVISITN*TRTPN | | 14 | 2 | 2.4871 | 0.9315 | 261 | 2.67 | 0.0081 |
| AVISITN*TRTPN | | 14 | 3 | 0 | | | | |
| AVISITN*TRTPN | | 21 | 1 | 1.0810 | 0.8683 | 218 | 1.24 | 0.2145 |
| AVISITN*TRTPN | | 21 | 2 | 0.9914 | 0.7662 | 241 | 1.29 | 0.1969 |
| AVISITN*TRTPN | | 21 | 3 | 0 | | | | |
| AVISITN*TRTPN | | 28 | 1 | -0.3136 | 0.7115 | 221 | -0.44 | 0.6598 |
| AVISITN*TRTPN | | 28 | 2 | -0.5811 | 0.6981 | 233 | -0.83 | 0.4061 |
| AVISITN*TRTPN | | 28 | 3 | 0 | | | | |

CENTANAFADINE 15 OF 26 PROTOCOL 405-201-00013

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ ({\tt Efficacy\ Sample})$ 

\_\_\_\_\_

#### The Mixed Procedure

# Solution for Fixed Effects

| Effect | Pooled<br>Center<br>Number | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | 35 | 1 | -0.02212 | 0.6892 | 228 | -0.03 | 0.9744 |
| AVISITN*TRTPN | | 35 | 2 | -0.7416 | 0.7276 | 234 | -1.02 | 0.3091 |
| AVISITN*TRTPN | | 35 | 3 | 0 | | | | |
| AVISITN*TRTPN | | 42 | 1 | 0 | | | | |
| AVISITN*TRTPN | | 42 | 2 | 0 | | | | |
| AVISITN*TRTPN | | 42 | 3 | 0 | | | | |
| POOLCNTR | | | | -1.3093 | 3.9540 | 335 | -0.33 | 0.7408 |
| POOLCNTR | | | | -0.7279 | 3.8546 | 333 | -0.19 | 0.8503 |
| POOLCNTR | | | | -1.6459 | 3.9898 | 337 | -0.41 | 0.6802 |
| POOLCNTR | | | | -1.6408 | 3.7641 | 330 | -0.44 | 0.6632 |
| POOLCNTR | | | | -1.6465 | 3.8229 | 333 | -0.43 | 0.6670 |
| POOLCNTR | | | | -2.4145 | 4.3086 | 350 | -0.56 | 0.5756 |
| POOLCNTR | | | | -6.6124 | 4.3891 | 343 | -1.51 | 0.1328 |
| POOLCNTR | | | | -7.0649 | 5.4521 | 366 | -1.30 | 0.1959 |
| POOLCNTR | | | | -5.7267 | 3.9888 | 333 | -1.44 | 0.1520 |
| POOLCNTR | | | | -2.2694 | 4.8320 | 342 | -0.47 | 0.6389 |
| POOLCNTR | | | | -3.1596 | 3.7355 | 330 | -0.85 | 0.3983 |
| POOLCNTR | | | | -6.0142 | 4.1721 | 353 | -1.44 | 0.1503 |
| POOLCNTR | | | | 0.8807 | 4.2539 | 340 | 0.21 | 0.8361 |
| POOLCNTR | | | | -3.8300 | 4.2304 | 355 | -0.91 | 0.3659 |
| POOLCNTR | | | | -2.5117 | 4.3115 | 345 | -0.58 | 0.5606 |
| POOLCNTR | | | | -2.7422 | 4.8000 | 380 | -0.57 | 0.5681 |

CENTANAFADINE 16 OF 26 PROTOCOL 405-201-00013

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ ({\tt Efficacy\ Sample})$ 

\_\_\_\_\_

Parameter Code=AISRSTOT ------

# The Mixed Procedure

# Solution for Fixed Effects

| | Pooled | Analysis | Planned | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Center | Visit | Treatment | | Standard | | | |
| Effect | Number | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| POOLCNTR | | | | -2.6550 | 3.9942 | 344 | -0.66 | 0.5067 |
| POOLCNTR | | | | -5.0193 | 4.3859 | 342 | -1.14 | 0.2533 |
| POOLCNTR | | | | 0.07424 | 5.4356 | 368 | 0.01 | 0.9891 |
| POOLCNTR | | | | -2.1018 | 4.4549 | 338 | -0.47 | 0.6374 |
| POOLCNTR | | | | -4.1304 | 5.1284 | 376 | -0.81 | 0.4211 |
| POOLCNTR | | | | 0.3290 | 4.7835 | 343 | 0.07 | 0.9452 |
| POOLCNTR | | | | -1.2695 | 4.8590 | 375 | -0.26 | 0.7940 |
| POOLCNTR | | | | -3.0686 | 4.5967 | 355 | -0.67 | 0.5048 |
| POOLCNTR | | | | -2.1150 | 3.8922 | 338 | -0.54 | 0.5872 |
| POOLCNTR | | | | -4.1346 | 4.2846 | 359 | -0.96 | 0.3352 |
| POOLCNTR | | | | -4.7395 | 4.1998 | 347 | -1.13 | 0.2599 |
| POOLCNTR | | | | -4.0008 | 4.7432 | 345 | -0.84 | 0.3995 |
| POOLCNTR | | | | -11.9023 | 3.8364 | 333 | -3.10 | 0.0021 |
| POOLCNTR | | | | 2.1419 | 5.4591 | 363 | 0.39 | 0.6950 |
| POOLCNTR | | | | 3.1038 | 4.6133 | 353 | 0.67 | 0.5015 |
| POOLCNTR | | | | -2.8280 | 5.0206 | 357 | -0.56 | 0.5736 |
| POOLCNTR | | | | -2.0196 | 5.1661 | 388 | -0.39 | 0.6961 |
| POOLCNTR | | | | -1.0234 | 3.9312 | 338 | -0.26 | 0.7948 |
| POOLCNTR | | | | -5.1194 | 3.8469 | 331 | -1.33 | 0.1842 |
| POOLCNTR | | | | -1.7274 | 5.0914 | 377 | -0.34 | 0.7346 |
| POOLCNTR | | | | -1.2967 | 5.0881 | 378 | -0.25 | 0.7990 |
| POOLCNTR | | | | 0 | | | | |

CENTANAFADINE 17 OF 26 PROTOCOL 405-201-00013

# STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

Parameter Code=AISRSTOT ------

#### The Mixed Procedure

# Solution for Fixed Effects

| | Pooled<br>Center | Analysis<br>Visit | Treatment | | Standard | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Number | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| BASE*AVISITN | | 7 | | -0.02539 | 0.06167 | 394 | -0.41 | 0.6808 |
| BASE*AVISITN | | 14 | | -0.08601 | 0.07029 | 442 | -1.22 | 0.2217 |
| BASE*AVISITN | | 21 | | -0.03257 | 0.07393 | 445 | -0.44 | 0.6597 |
| BASE*AVISITN | | 28 | | -0.1639 | 0.08209 | 447 | -2.00 | 0.0465 |
| BASE*AVISITN | | 35 | | -0.1325 | 0.08419 | 458 | -1.57 | 0.1163 |
| BASE*AVISITN | | 42 | | -0.1191 | 0.08648 | 447 | -1.38 | 0.1690 |

# Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------------|-----------|-----------|---------|--------|
| AVISITN | 5 | 369 | 1.80 | 0.1124 |
| TRTPN | 2 | 259 | 3.15 | 0.0444 |
| AVISITN*TRTPN | 10 | 316 | 1.70 | 0.0795 |
| POOLCNTR | 37 | 387 | 2.00 | 0.0007 |
| BASE*AVISITN | 6 | 392 | 1.99 | 0.0662 |

CENTANAFADINE 18 OF 26 PROTOCOL 405-201-00013

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ ({\tt Efficacy\ Sample})$ 

\_\_\_\_\_

# The Mixed Procedure

# Least Squares Means

| Effect | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN | 7 | 1 | -5.4621 | 0.7260 | 152 | -7.52 | <.0001 | 0.05 | -6.8964 | -4.0278 |
| AVISITN*TRTPN | 7 | 2 | -4.0298 | 0.6402 | 174 | -6.29 | <.0001 | 0.05 | -5.2934 | -2.7661 |
| AVISITN*TRTPN | 7 | 3 | -4.1595 | 0.6417 | 166 | -6.48 | <.0001 | 0.05 | -5.4263 | -2.8926 |
| AVISITN*TRTPN | 14 | 1 | -7.4177 | 0.7968 | 154 | -9.31 | <.0001 | 0.05 | -8.9917 | -5.8437 |
| AVISITN*TRTPN | 14 | 2 | -6.6938 | 0.7750 | 166 | -8.64 | <.0001 | 0.05 | -8.2239 | -5.1637 |
| AVISITN*TRTPN | 14 | 3 | -6.4243 | 0.7445 | 165 | -8.63 | <.0001 | 0.05 | -7.8943 | -4.9544 |
| AVISITN*TRTPN | 21 | 1 | -8.4528 | 0.8292 | 144 | -10.19 | <.0001 | 0.05 | -10.0918 | -6.8137 |
| AVISITN*TRTPN | 21 | 2 | -8.2660 | 0.8380 | 158 | -9.86 | <.0001 | 0.05 | -9.9212 | -6.6108 |
| AVISITN*TRTPN | 21 | 3 | -6.5008 | 0.7887 | 165 | -8.24 | <.0001 | 0.05 | -8.0580 | -4.9436 |
| AVISITN*TRTPN | 28 | 1 | -9.6039 | 0.9837 | 145 | -9.76 | <.0001 | 0.05 | -11.5482 | -7.6596 |
| AVISITN*TRTPN | 28 | 2 | -9.5949 | 0.9555 | 153 | -10.04 | <.0001 | 0.05 | -11.4827 | -7.7071 |
| AVISITN*TRTPN | 28 | 3 | -6.2572 | 0.8577 | 160 | -7.30 | <.0001 | 0.05 | -7.9511 | -4.5634 |
| AVISITN*TRTPN | 35 | 1 | -10.2433 | 0.9879 | 145 | -10.37 | <.0001 | 0.05 | -12.1959 | -8.2908 |
| AVISITN*TRTPN | 35 | 2 | -10.6864 | 0.9502 | 152 | -11.25 | <.0001 | 0.05 | -12.5638 | -8.8090 |
| AVISITN*TRTPN | 35 | 3 | -7.1882 | 0.9300 | 159 | -7.73 | <.0001 | 0.05 | -9.0250 | -5.3515 |
| AVISITN*TRTPN | 42 | 1 | -10.0246 | 1.1034 | 141 | -9.09 | <.0001 | 0.05 | -12.2058 | -7.8433 |
| AVISITN*TRTPN | 42 | 2 | -9.7481 | 0.9464 | 155 | -10.30 | <.0001 | 0.05 | -11.6176 | -7.8787 |
| AVISITN*TRTPN | 42 | 3 | -6.9916 | 0.9122 | 159 | -7.66 | <.0001 | 0.05 | -8.7932 | -5.1899 |

CENTANAFADINE 19 OF 26


# STAT-4.10 Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

\_\_\_\_\_\_

------ Parameter Code=AISRSTOT ------

#### The Mixed Procedure

# Differences of Least Squares Means

| | Analysis | Planned | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | Treatment | Visit | Treatment | | Standard | | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 7 | 1 | 7 | 2 | -1.4324 | 0.8834 | 249 | -1.62 | 0.1062 | 0.05 | -3.1723 | 0.3075 |
| AVISITN*TRTPN | 7 | 1 | 7 | 3 | -1.3027 | 0.8872 | 253 | -1.47 | 0.1433 | 0.05 | -3.0499 | 0.4446 |
| AVISITN*TRTPN | 7 | 1 | 14 | 1 | 1.9555 | 0.6484 | 129 | 3.02 | 0.0031 | 0.05 | 0.6726 | 3.2385 |
| AVISITN*TRTPN | 7 | 1 | 14 | 2 | 1.2316 | 0.9852 | 263 | 1.25 | 0.2124 | 0.05 | -0.7083 | 3.1716 |
| AVISITN*TRTPN | 7 | 1 | 14 | 3 | 0.9622 | 0.9628 | 263 | 1.00 | 0.3186 | 0.05 | -0.9337 | 2.8580 |
| AVISITN*TRTPN | 7 | 1 | 21 | 1 | 2.9906 | 0.6630 | 136 | 4.51 | <.0001 | 0.05 | 1.6796 | 4.3017 |
| AVISITN*TRTPN | 7 | 1 | 21 | 2 | 2.8038 | 1.0353 | 258 | 2.71 | 0.0072 | 0.05 | 0.7650 | 4.8426 |
| AVISITN*TRTPN | 7 | 1 | 21 | 3 | 1.0387 | 0.9969 | 266 | 1.04 | 0.2984 | 0.05 | -0.9242 | 3.0015 |
| AVISITN*TRTPN | 7 | 1 | 28 | 1 | 4.1417 | 0.8366 | 125 | 4.95 | <.0001 | 0.05 | 2.4860 | 5.7975 |
| AVISITN*TRTPN | 7 | 1 | 28 | 2 | 4.1328 | 1.1322 | 242 | 3.65 | 0.0003 | 0.05 | 1.9026 | 6.3630 |
| AVISITN*TRTPN | 7 | 1 | 28 | 3 | 0.7951 | 1.0524 | 262 | 0.76 | 0.4506 | 0.05 | -1.2771 | 2.8673 |
| AVISITN*TRTPN | 7 | 1 | 35 | 1 | 4.7812 | 0.8422 | 126 | 5.68 | <.0001 | 0.05 | 3.1144 | 6.4480 |
| AVISITN*TRTPN | 7 | 1 | 35 | 2 | 5.2243 | 1.1280 | 240 | 4.63 | <.0001 | 0.05 | 3.0022 | 7.4463 |
| AVISITN*TRTPN | 7 | 1 | 35 | 3 | 1.7261 | 1.1120 | 255 | 1.55 | 0.1219 | 0.05 | -0.4638 | 3.9160 |
| AVISITN*TRTPN | 7 | 1 | 42 | 1 | 4.5625 | 1.0080 | 124 | 4.53 | <.0001 | 0.05 | 2.5674 | 6.5575 |
| AVISITN*TRTPN | 7 | 1 | 42 | 2 | 4.2860 | 1.1248 | 243 | 3.81 | 0.0002 | 0.05 | 2.0703 | 6.5017 |
| AVISITN*TRTPN | 7 | 1 | 42 | 3 | 1.5294 | 1.0974 | 255 | 1.39 | 0.1646 | 0.05 | -0.6317 | 3.6905 |
| AVISITN*TRTPN | 7 | 2 | 7 | 3 | 0.1297 | 0.8064 | 260 | 0.16 | 0.8723 | 0.05 | -1.4582 | 1.7177 |
| AVISITN*TRTPN | 7 | 2 | 14 | 1 | 3.3879 | 0.9433 | 247 | 3.59 | 0.0004 | 0.05 | 1.5300 | 5.2459 |
| AVISITN*TRTPN | 7 | 2 | 14 | 2 | 2.6640 | 0.5142 | 139 | 5.18 | <.0001 | 0.05 | 1.6473 | 3.6807 |
| AVISITN*TRTPN | 7 | 2 | 14 | 3 | 2.3946 | 0.8886 | 255 | 2.69 | 0.0075 | 0.05 | 0.6447 | 4.1445 |
| AVISITN*TRTPN | 7 | 2 | 21 | 1 | 4.4230 | 0.9707 | 233 | 4.56 | <.0001 | 0.05 | 2.5105 | 6.3355 |

CENTANAFADINE 20 OF 26 PROTOCOL 405-201-00013

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ ({\tt Efficacy\ Sample})$ 

------

#### The Mixed Procedure

# Differences of Least Squares Means

| | Analysis | Planned | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | Treatment | Visit | Treatment | | Standard | | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 7 | 2 | 21 | 2 | 4.2362 | 0.6527 | 138 | 6.49 | <.0001 | 0.05 | 2.9457 | 5.5267 |
| AVISITN*TRTPN | 7 | 2 | 21 | 3 | 2.4711 | 0.9253 | 248 | 2.67 | 0.0081 | 0.05 | 0.6486 | 4.2936 |
| AVISITN*TRTPN | 7 | 2 | 28 | 1 | 5.5741 | 1.1055 | 214 | 5.04 | <.0001 | 0.05 | 3.3950 | 7.7532 |
| AVISITN*TRTPN | 7 | 2 | 28 | 2 | 5.5651 | 0.8296 | 133 | 6.71 | <.0001 | 0.05 | 3.9243 | 7.2060 |
| AVISITN*TRTPN | 7 | 2 | 28 | 3 | 2.2275 | 0.9848 | 232 | 2.26 | 0.0246 | 0.05 | 0.2872 | 4.1678 |
| AVISITN*TRTPN | 7 | 2 | 35 | 1 | 6.2136 | 1.1092 | 214 | 5.60 | <.0001 | 0.05 | 4.0273 | 8.3998 |
| AVISITN*TRTPN | 7 | 2 | 35 | 2 | 6.6566 | 0.7932 | 130 | 8.39 | <.0001 | 0.05 | 5.0873 | 8.2260 |
| AVISITN*TRTPN | 7 | 2 | 35 | 3 | 3.1585 | 1.0483 | 227 | 3.01 | 0.0029 | 0.05 | 1.0928 | 5.2241 |
| AVISITN*TRTPN | 7 | 2 | 42 | 1 | 5.9948 | 1.2133 | 198 | 4.94 | <.0001 | 0.05 | 3.6023 | 8.3874 |
| AVISITN*TRTPN | 7 | 2 | 42 | 2 | 5.7184 | 0.7711 | 134 | 7.42 | <.0001 | 0.05 | 4.1932 | 7.2435 |
| AVISITN*TRTPN | 7 | 2 | 42 | 3 | 2.9618 | 1.0328 | 226 | 2.87 | 0.0045 | 0.05 | 0.9267 | 4.9970 |
| AVISITN*TRTPN | 7 | 3 | 14 | 1 | 3.2582 | 0.9468 | 250 | 3.44 | 0.0007 | 0.05 | 1.3935 | 5.1229 |
| AVISITN*TRTPN | 7 | 3 | 14 | 2 | 2.5343 | 0.9168 | 245 | 2.76 | 0.0061 | 0.05 | 0.7286 | 4.3400 |
| AVISITN*TRTPN | 7 | 3 | 14 | 3 | 2.2649 | 0.5534 | 139 | 4.09 | <.0001 | 0.05 | 1.1708 | 3.3589 |
| AVISITN*TRTPN | 7 | 3 | 21 | 1 | 4.2933 | 0.9741 | 231 | 4.41 | <.0001 | 0.05 | 2.3741 | 6.2125 |
| AVISITN*TRTPN | 7 | 3 | 21 | 2 | 4.1065 | 0.9705 | 231 | 4.23 | <.0001 | 0.05 | 2.1944 | 6.0186 |
| AVISITN*TRTPN | 7 | 3 | 21 | 3 | 2.3413 | 0.6524 | 140 | 3.59 | 0.0005 | 0.05 | 1.0515 | 3.6311 |
| AVISITN*TRTPN | 7 | 3 | 28 | 1 | 5.4444 | 1.1085 | 215 | 4.91 | <.0001 | 0.05 | 3.2595 | 7.6293 |
| AVISITN*TRTPN | 7 | 3 | 28 | 2 | 5.4354 | 1.0732 | 214 | 5.06 | <.0001 | 0.05 | 3.3200 | 7.5508 |
| AVISITN*TRTPN | 7 | 3 | 28 | 3 | 2.0978 | 0.7357 | 142 | 2.85 | 0.0050 | 0.05 | 0.6435 | 3.5521 |
| AVISITN*TRTPN | 7 | 3 | 35 | 1 | 6.0839 | 1.1121 | 215 | 5.47 | <.0001 | 0.05 | 3.8918 | 8.2760 |
| AVISITN*TRTPN | 7 | 3 | 35 | 2 | 6.5269 | 1.0688 | 214 | 6.11 | <.0001 | 0.05 | 4.4202 | 8.6336 |

CENTANAFADINE 21 OF 26 PROTOCOL 405-201-00013

# STAT-4.10 Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

------

#### The Mixed Procedure

# Differences of Least Squares Means

| | Analysis | Planned | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | Treatment | Visit | Treatment | | Standard | | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 7 | 3 | 35 | 3 | 3.0287 | 0.8227 | 140 | 3.68 | 0.0003 | 0.05 | 1.4022 | 4.6552 |
| AVISITN*TRTPN | 7 | 3 | 42 | 1 | 5.8651 | 1.2160 | 198 | 4.82 | <.0001 | 0.05 | 3.4673 | 8.2630 |
| AVISITN*TRTPN | 7 | 3 | 42 | 2 | 5.5886 | 1.0654 | 221 | 5.25 | <.0001 | 0.05 | 3.4889 | 7.6884 |
| AVISITN*TRTPN | 7 | 3 | 42 | 3 | 2.8321 | 0.7825 | 140 | 3.62 | 0.0004 | 0.05 | 1.2850 | 4.3792 |
| AVISITN*TRTPN | 14 | 1 | 14 | 2 | -0.7239 | 1.0393 | 273 | -0.70 | 0.4867 | 0.05 | -2.7701 | 1.3222 |
| AVISITN*TRTPN | 14 | 1 | 14 | 3 | -0.9933 | 1.0181 | 261 | -0.98 | 0.3301 | 0.05 | -2.9980 | 1.0113 |
| AVISITN*TRTPN | 14 | 1 | 21 | 1 | 1.0351 | 0.5228 | 121 | 1.98 | 0.0500 | 0.05 | 0.000165 | 2.0701 |
| AVISITN*TRTPN | 14 | 1 | 21 | 2 | 0.8483 | 1.0869 | 271 | 0.78 | 0.4358 | 0.05 | -1.2916 | 2.9882 |
| AVISITN*TRTPN | 14 | 1 | 21 | 3 | -0.9169 | 1.0504 | 265 | -0.87 | 0.3835 | 0.05 | -2.9850 | 1.1513 |
| AVISITN*TRTPN | 14 | 1 | 28 | 1 | 2.1862 | 0.6913 | 123 | 3.16 | 0.0020 | 0.05 | 0.8179 | 3.5545 |
| AVISITN*TRTPN | 14 | 1 | 28 | 2 | 2.1772 | 1.1796 | 259 | 1.85 | 0.0661 | 0.05 | -0.1455 | 4.5000 |
| AVISITN*TRTPN | 14 | 1 | 28 | 3 | -1.1604 | 1.1031 | 267 | -1.05 | 0.2938 | 0.05 | -3.3324 | 1.0115 |
| AVISITN*TRTPN | 14 | 1 | 35 | 1 | 2.8257 | 0.6812 | 124 | 4.15 | <.0001 | 0.05 | 1.4775 | 4.1738 |
| AVISITN*TRTPN | 14 | 1 | 35 | 2 | 3.2687 | 1.1755 | 256 | 2.78 | 0.0058 | 0.05 | 0.9538 | 5.5837 |
| AVISITN*TRTPN | 14 | 1 | 35 | 3 | -0.2295 | 1.1602 | 265 | -0.20 | 0.8434 | 0.05 | -2.5137 | 2.0548 |
| AVISITN*TRTPN | 14 | 1 | 42 | 1 | 2.6069 | 0.8200 | 121 | 3.18 | 0.0019 | 0.05 | 0.9836 | 4.2302 |
| AVISITN*TRTPN | 14 | 1 | 42 | 2 | 2.3305 | 1.1725 | 260 | 1.99 | 0.0479 | 0.05 | 0.02168 | 4.6392 |
| AVISITN*TRTPN | 14 | 1 | 42 | 3 | -0.4261 | 1.1462 | 266 | -0.37 | 0.7104 | 0.05 | -2.6828 | 1.8306 |
| AVISITN*TRTPN | 14 | 2 | 14 | 3 | -0.2694 | 0.9898 | 261 | -0.27 | 0.7857 | 0.05 | -2.2183 | 1.6795 |
| AVISITN*TRTPN | 14 | 2 | 21 | 1 | 1.7590 | 1.0642 | 265 | 1.65 | 0.0995 | 0.05 | -0.3364 | 3.8545 |
| AVISITN*TRTPN | 14 | 2 | 21 | 2 | 1.5722 | 0.4849 | 133 | 3.24 | 0.0015 | 0.05 | 0.6131 | 2.5313 |
| AVISITN*TRTPN | 14 | 2 | 21 | 3 | -0.1929 | 1.0229 | 262 | -0.19 | 0.8505 | 0.05 | -2.2071 | 1.8212 |

CENTANAFADINE 22 OF 26 PROTOCOL 405-201-00013

# ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ ({\tt Efficacy\ Sample})$

------

Parameter Code=AISRSTOT ------

#### The Mixed Procedure

# Differences of Least Squares Means

| | Analysis | Planned | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | Treatment | Visit | Treatment | | Standard | | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 14 | 2 | 28 | 1 | 2.9101 | 1.1885 | 251 | 2.45 | 0.0150 | 0.05 | 0.5695 | 5.2508 |
| AVISITN*TRTPN | 14 | 2 | 28 | 2 | 2.9011 | 0.7202 | 131 | 4.03 | <.0001 | 0.05 | 1.4764 | 4.3259 |
| AVISITN*TRTPN | 14 | 2 | 28 | 3 | -0.4365 | 1.0770 | 256 | -0.41 | 0.6856 | 0.05 | -2.5574 | 1.6844 |
| AVISITN*TRTPN | 14 | 2 | 35 | 1 | 3.5496 | 1.1919 | 249 | 2.98 | 0.0032 | 0.05 | 1.2022 | 5.8970 |
| AVISITN*TRTPN | 14 | 2 | 35 | 2 | 3.9926 | 0.6830 | 132 | 5.85 | <.0001 | 0.05 | 2.6415 | 5.3438 |
| AVISITN*TRTPN | 14 | 2 | 35 | 3 | 0.4945 | 1.1353 | 251 | 0.44 | 0.6636 | 0.05 | -1.7415 | 2.7304 |
| AVISITN*TRTPN | 14 | 2 | 42 | 1 | 3.3308 | 1.2893 | 232 | 2.58 | 0.0104 | 0.05 | 0.7906 | 5.8711 |
| AVISITN*TRTPN | 14 | 2 | 42 | 2 | 3.0544 | 0.6732 | 131 | 4.54 | <.0001 | 0.05 | 1.7227 | 4.3861 |
| AVISITN*TRTPN | 14 | 2 | 42 | 3 | 0.2978 | 1.1211 | 251 | 0.27 | 0.7907 | 0.05 | -1.9101 | 2.5057 |
| AVISITN*TRTPN | 14 | 3 | 21 | 1 | 2.0285 | 1.0435 | 246 | 1.94 | 0.0530 | 0.05 | -0.02684 | 4.0838 |
| AVISITN*TRTPN | 14 | 3 | 21 | 2 | 1.8416 | 1.0397 | 252 | 1.77 | 0.0777 | 0.05 | -0.2060 | 3.8892 |
| AVISITN*TRTPN | 14 | 3 | 21 | 3 | 0.07648 | 0.4315 | 135 | 0.18 | 0.8596 | 0.05 | -0.7769 | 0.9299 |
| AVISITN*TRTPN | 14 | 3 | 28 | 1 | 3.1795 | 1.1699 | 236 | 2.72 | 0.0071 | 0.05 | 0.8747 | 5.4844 |
| AVISITN*TRTPN | 14 | 3 | 28 | 2 | 3.1706 | 1.1362 | 239 | 2.79 | 0.0057 | 0.05 | 0.9323 | 5.4088 |
| AVISITN*TRTPN | 14 | 3 | 28 | 3 | -0.1671 | 0.5311 | 135 | -0.31 | 0.7536 | 0.05 | -1.2175 | 0.8833 |
| AVISITN*TRTPN | 14 | 3 | 35 | 1 | 3.8190 | 1.1734 | 236 | 3.25 | 0.0013 | 0.05 | 1.5074 | 6.1306 |
| AVISITN*TRTPN | 14 | 3 | 35 | 2 | 4.2621 | 1.1320 | 238 | 3.76 | 0.0002 | 0.05 | 2.0320 | 6.4921 |
| AVISITN*TRTPN | 14 | 3 | 35 | 3 | 0.7639 | 0.6655 | 135 | 1.15 | 0.2530 | 0.05 | -0.5522 | 2.0799 |
| AVISITN*TRTPN | 14 | 3 | 42 | 1 | 3.6003 | 1.2722 | 219 | 2.83 | 0.0051 | 0.05 | 1.0929 | 6.1076 |
| AVISITN*TRTPN | 14 | 3 | 42 | 2 | 3.3238 | 1.1289 | 246 | 2.94 | 0.0035 | 0.05 | 1.1003 | 5.5473 |
| AVISITN*TRTPN | 14 | 3 | 42 | 3 | 0.5672 | 0.6438 | 130 | 0.88 | 0.3799 | 0.05 | -0.7064 | 1.8409 |
| AVISITN*TRTPN | 21 | 1 | 21 | 2 | -0.1868 | 1.1108 | 266 | -0.17 | 0.8666 | 0.05 | -2.3740 | 2.0003 |

CENTANAFADINE 23 OF 26 PROTOCOL 405-201-00013

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ ({\tt Efficacy\ Sample})$ 

------

# The Mixed Procedure

# Differences of Least Squares Means

| | Analysis | Planned | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | Treatment | Visit | Treatment | | Standard | | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 21 | 1 | 21 | 3 | -1.9520 | 1.0750 | 255 | -1.82 | 0.0706 | 0.05 | -4.0690 | 0.1651 |
| AVISITN*TRTPN | 21 | 1 | 28 | 1 | 1.1511 | 0.5594 | 117 | 2.06 | 0.0418 | 0.05 | 0.04332 | 2.2589 |
| AVISITN*TRTPN | 21 | 1 | 28 | 2 | 1.1421 | 1.2016 | 261 | 0.95 | 0.3427 | 0.05 | -1.2240 | 3.5082 |
| AVISITN*TRTPN | 21 | 1 | 28 | 3 | -2.1955 | 1.1266 | 259 | -1.95 | 0.0524 | 0.05 | -4.4141 | 0.02302 |
| AVISITN*TRTPN | 21 | 1 | 35 | 1 | 1.7906 | 0.5443 | 116 | 3.29 | 0.0013 | 0.05 | 0.7125 | 2.8687 |
| AVISITN*TRTPN | 21 | 1 | 35 | 2 | 2.2336 | 1.1977 | 257 | 1.86 | 0.0633 | 0.05 | -0.1249 | 4.5921 |
| AVISITN*TRTPN | 21 | 1 | 35 | 3 | -1.2646 | 1.1825 | 260 | -1.07 | 0.2859 | 0.05 | -3.5931 | 1.0640 |
| AVISITN*TRTPN | 21 | 1 | 42 | 1 | 1.5718 | 0.6948 | 117 | 2.26 | 0.0255 | 0.05 | 0.1959 | 2.9478 |
| AVISITN*TRTPN | 21 | 1 | 42 | 2 | 1.2953 | 1.1947 | 261 | 1.08 | 0.2792 | 0.05 | -1.0571 | 3.6478 |
| AVISITN*TRTPN | 21 | 1 | 42 | 3 | -1.4612 | 1.1688 | 259 | -1.25 | 0.2124 | 0.05 | -3.7628 | 0.8404 |
| AVISITN*TRTPN | 21 | 2 | 21 | 3 | -1.7652 | 1.0712 | 256 | -1.65 | 0.1006 | 0.05 | -3.8748 | 0.3444 |
| AVISITN*TRTPN | 21 | 2 | 28 | 1 | 1.3379 | 1.2304 | 259 | 1.09 | 0.2779 | 0.05 | -1.0849 | 3.7607 |
| AVISITN*TRTPN | 21 | 2 | 28 | 2 | 1.3289 | 0.5423 | 125 | 2.45 | 0.0156 | 0.05 | 0.2557 | 2.4021 |
| AVISITN*TRTPN | 21 | 2 | 28 | 3 | -2.0087 | 1.1231 | 257 | -1.79 | 0.0749 | 0.05 | -4.2203 | 0.2029 |
| AVISITN*TRTPN | 21 | 2 | 35 | 1 | 1.9774 | 1.2336 | 257 | 1.60 | 0.1102 | 0.05 | -0.4519 | 4.4067 |
| AVISITN*TRTPN | 21 | 2 | 35 | 2 | 2.4204 | 0.4860 | 122 | 4.98 | <.0001 | 0.05 | 1.4583 | 3.3826 |
| AVISITN*TRTPN | 21 | 2 | 35 | 3 | -1.0778 | 1.1791 | 254 | -0.91 | 0.3616 | 0.05 | -3.3998 | 1.2443 |
| AVISITN*TRTPN | 21 | 2 | 42 | 1 | 1.7586 | 1.3280 | 243 | 1.32 | 0.1867 | 0.05 | -0.8572 | 4.3745 |
| AVISITN*TRTPN | 21 | 2 | 42 | 2 | 1.4822 | 0.5617 | 123 | 2.64 | 0.0094 | 0.05 | 0.3702 | 2.5941 |
| AVISITN*TRTPN | 21 | 2 | 42 | 3 | -1.2744 | 1.1654 | 254 | -1.09 | 0.2752 | 0.05 | -3.5694 | 1.0206 |
| AVISITN*TRTPN | 21 | 3 | 28 | 1 | 3.1031 | 1.1982 | 247 | 2.59 | 0.0102 | 0.05 | 0.7431 | 5.4630 |
| AVISITN*TRTPN | 21 | 3 | 28 | 2 | 3.0941 | 1.1652 | 246 | 2.66 | 0.0084 | 0.05 | 0.7991 | 5.3891 |

CENTANAFADINE 24 OF 26 PROTOCOL 405-201-00013

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ ({\tt Efficacy\ Sample})$ 

------

# The Mixed Procedure

# Differences of Least Squares Means

| | Analysis | Planned | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | Treatment | Visit | Treatment | | Standard | | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 21 | 3 | 28 | 3 | -0.2436 | 0.4409 | 129 | -0.55 | 0.5816 | 0.05 | -1.1158 | 0.6287 |
| AVISITN*TRTPN | 21 | 3 | 35 | 1 | 3.7425 | 1.2015 | 247 | 3.11 | 0.0021 | 0.05 | 1.3760 | 6.1091 |
| AVISITN*TRTPN | 21 | 3 | 35 | 2 | 4.1856 | 1.1611 | 246 | 3.60 | 0.0004 | 0.05 | 1.8987 | 6.4725 |
| AVISITN*TRTPN | 21 | 3 | 35 | 3 | 0.6874 | 0.4989 | 125 | 1.38 | 0.1707 | 0.05 | -0.2999 | 1.6747 |
| AVISITN*TRTPN | 21 | 3 | 42 | 1 | 3.5238 | 1.2982 | 229 | 2.71 | 0.0071 | 0.05 | 0.9658 | 6.0817 |
| AVISITN*TRTPN | 21 | 3 | 42 | 2 | 3.2473 | 1.1580 | 252 | 2.80 | 0.0054 | 0.05 | 0.9667 | 5.5279 |
| AVISITN*TRTPN | 21 | 3 | 42 | 3 | 0.4908 | 0.5209 | 118 | 0.94 | 0.3481 | 0.05 | -0.5408 | 1.5223 |
| AVISITN*TRTPN | 28 | 1 | 28 | 2 | -0.00898 | 1.3130 | 269 | -0.01 | 0.9945 | 0.05 | -2.5940 | 2.5760 |
| AVISITN*TRTPN | 28 | 1 | 28 | 3 | -3.3466 | 1.2447 | 256 | -2.69 | 0.0076 | 0.05 | -5.7977 | -0.8955 |
| AVISITN*TRTPN | 28 | 1 | 35 | 1 | 0.6395 | 0.4336 | 113 | 1.47 | 0.1430 | 0.05 | -0.2195 | 1.4985 |
| AVISITN*TRTPN | 28 | 1 | 35 | 2 | 1.0825 | 1.3093 | 266 | 0.83 | 0.4091 | 0.05 | -1.4955 | 3.6605 |
| AVISITN*TRTPN | 28 | 1 | 35 | 3 | -2.4157 | 1.2955 | 265 | -1.86 | 0.0633 | 0.05 | -4.9664 | 0.1351 |
| AVISITN*TRTPN | 28 | 1 | 42 | 1 | 0.4207 | 0.5447 | 112 | 0.77 | 0.4416 | 0.05 | -0.6586 | 1.5001 |
| AVISITN*TRTPN | 28 | 1 | 42 | 2 | 0.1442 | 1.3066 | 267 | 0.11 | 0.9122 | 0.05 | -2.4283 | 2.7168 |
| AVISITN*TRTPN | 28 | 1 | 42 | 3 | -2.6123 | 1.2830 | 261 | -2.04 | 0.0427 | 0.05 | -5.1386 | -0.08601 |
| AVISITN*TRTPN | 28 | 2 | 28 | 3 | -3.3376 | 1.2130 | 252 | -2.75 | 0.0064 | 0.05 | -5.7265 | -0.9488 |
| AVISITN*TRTPN | 28 | 2 | 35 | 1 | 0.6485 | 1.3160 | 268 | 0.49 | 0.6226 | 0.05 | -1.9426 | 3.2395 |
| AVISITN*TRTPN | 28 | 2 | 35 | 2 | 1.0915 | 0.4672 | 117 | 2.34 | 0.0212 | 0.05 | 0.1662 | 2.0168 |
| AVISITN*TRTPN | 28 | 2 | 35 | 3 | -2.4067 | 1.2650 | 256 | -1.90 | 0.0582 | 0.05 | -4.8978 | 0.08446 |
| AVISITN*TRTPN | 28 | 2 | 42 | 1 | 0.4297 | 1.4049 | 260 | 0.31 | 0.7600 | 0.05 | -2.3367 | 3.1961 |
| AVISITN*TRTPN | 28 | 2 | 42 | 2 | 0.1532 | 0.5269 | 120 | 0.29 | 0.7717 | 0.05 | -0.8901 | 1.1966 |
| AVISITN*TRTPN | 28 | 2 | 42 | 3 | -2.6033 | 1.2522 | 255 | -2.08 | 0.0386 | 0.05 | -5.0693 | -0.1373 |

CENTANAFADINE 25 OF 26 PROTOCOL 405-201-00013

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ ({\tt Efficacy\ Sample})$ 

\_\_\_\_\_\_

#### The Mixed Procedure

# Differences of Least Squares Means

| | Analysis | Planned | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | Treatment | Visit | Treatment | | Standard | | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 28 | 3 | 35 | 1 | 3.9861 | 1.2479 | 256 | 3.19 | 0.0016 | 0.05 | 1.5286 | 6.4436 |
| AVISITN*TRTPN | 28 | 3 | 35 | 2 | 4.4291 | 1.2091 | 256 | 3.66 | 0.0003 | 0.05 | 2.0482 | 6.8101 |
| AVISITN*TRTPN | 28 | 3 | 35 | 3 | 0.9310 | 0.4637 | 127 | 2.01 | 0.0468 | 0.05 | 0.01342 | 1.8485 |
| AVISITN*TRTPN | 28 | 3 | 42 | 1 | 3.7673 | 1.3413 | 241 | 2.81 | 0.0054 | 0.05 | 1.1252 | 6.4095 |
| AVISITN*TRTPN | 28 | 3 | 42 | 2 | 3.4909 | 1.2061 | 259 | 2.89 | 0.0041 | 0.05 | 1.1159 | 5.8659 |
| AVISITN*TRTPN | 28 | 3 | 42 | 3 | 0.7343 | 0.4577 | 117 | 1.60 | 0.1113 | 0.05 | -0.1721 | 1.6408 |
| AVISITN*TRTPN | 35 | 1 | 35 | 2 | 0.4430 | 1.3124 | 264 | 0.34 | 0.7359 | 0.05 | -2.1410 | 3.0271 |
| AVISITN*TRTPN | 35 | 1 | 35 | 3 | -3.0551 | 1.2986 | 265 | -2.35 | 0.0194 | 0.05 | -5.6120 | -0.4983 |
| AVISITN*TRTPN | 35 | 1 | 42 | 1 | -0.2188 | 0.4942 | 109 | -0.44 | 0.6589 | 0.05 | -1.1982 | 0.7607 |
| AVISITN*TRTPN | 35 | 1 | 42 | 2 | -0.4952 | 1.3097 | 266 | -0.38 | 0.7056 | 0.05 | -3.0739 | 2.0834 |
| AVISITN*TRTPN | 35 | 1 | 42 | 3 | -3.2518 | 1.2861 | 261 | -2.53 | 0.0121 | 0.05 | -5.7843 | -0.7193 |
| AVISITN*TRTPN | 35 | 2 | 35 | 3 | -3.4982 | 1.2613 | 258 | -2.77 | 0.0059 | 0.05 | -5.9819 | -1.0145 |
| AVISITN*TRTPN | 35 | 2 | 42 | 1 | -0.6618 | 1.4015 | 256 | -0.47 | 0.6372 | 0.05 | -3.4217 | 2.0981 |
| AVISITN*TRTPN | 35 | 2 | 42 | 2 | -0.9383 | 0.5462 | 119 | -1.72 | 0.0884 | 0.05 | -2.0198 | 0.1432 |
| AVISITN*TRTPN | 35 | 2 | 42 | 3 | -3.6948 | 1.2485 | 258 | -2.96 | 0.0034 | 0.05 | -6.1533 | -1.2363 |
| AVISITN*TRTPN | 35 | 3 | 42 | 1 | 2.8364 | 1.3886 | 253 | 2.04 | 0.0421 | 0.05 | 0.1018 | 5.5710 |
| AVISITN*TRTPN | 35 | 3 | 42 | 2 | 2.5599 | 1.2584 | 261 | 2.03 | 0.0429 | 0.05 | 0.08197 | 5.0379 |
| AVISITN*TRTPN | 35 | 3 | 42 | 3 | -0.1966 | 0.4806 | 120 | -0.41 | 0.6832 | 0.05 | -1.1482 | 0.7549 |
| AVISITN*TRTPN | 42 | 1 | 42 | 2 | -0.2765 | 1.3989 | 258 | -0.20 | 0.8435 | 0.05 | -3.0313 | 2.4783 |
| AVISITN*TRTPN | 42 | 1 | 42 | 3 | -3.0330 | 1.3769 | 249 | -2.20 | 0.0285 | 0.05 | -5.7448 | -0.3212 |
| AVISITN*TRTPN | 42 | 2 | 42 | 3 | -2.7565 | 1.2456 | 260 | -2.21 | 0.0278 | 0.05 | -5.2094 | -0.3037 |

CENTANAFADINE 26 OF 26 PROTOCOL 405-201-00013

# STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

The Mixed Procedure

Tests of Effect Slices

| | Analysis | | | | |
|---------------|----------|-----|-----|---------|--------|
| | Visit | Num | Den | | |
| Effect | (N) | DF | DF | F Value | Pr > F |
| AVISITN*TRTPN | 7 | 2 | 257 | 1.52 | 0.2216 |
| AVISITN*TRTPN | 14 | 2 | 265 | 0.50 | 0.6098 |
| AVISITN*TRTPN | 21 | 2 | 259 | 2.06 | 0.1301 |
| AVISITN*TRTPN | 28 | 2 | 261 | 5.16 | 0.0063 |
| AVISITN*TRTPN | 35 | 2 | 262 | 4.53 | 0.0117 |
| AVISITN*TRTPN | 42 | 2 | 260 | 3.39 | 0.0352 |

STAT-5.1

Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN) (Efficacy Sample)

\_\_\_\_\_

------ Parameter Code=CGI0201 ------

The Mixed Procedure

Model Information

Data Set WORK.INDATA
Dependent Variable CHG
Covariance Structure Unstructured
Subject Effect SUBJID
Estimation Method REML
Residual Variance Method None

Fixed Effects SE Method Kenward-Roger
Degrees of Freedom Method Kenward-Roger

Class Level Information

Class Levels Values

AVISITN 6 7 14 21 28 35 42

TRTPN 3 1 2 3

POOLCNTR 38


Levels

STAT-5.1 Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN) (Efficacy Sample)

The Mixed Procedure

Class Level Information Values

SUBJID 437

SOURCE: MMRMOUT; TABLE: stat1cgisa.lis; RUN: 18JUN2020 10:00; ANALYSIS DATASET CREATED: 11JUN2020 07:28 PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-5.1 FINAL

Class

CENTANAFADINE

3 OF 14

STAT-5.1
Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN)
(Efficacy Sample)

......

The Mixed Procedure



CENTANAFADINE 4 OF 14 PROTOCOL 405-201-00013

STAT-5.1
Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN)
(Efficacy Sample)

The Mixed Procedure




STAT-5.1
Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN)
(Efficacy Sample)

The Mixed Procedure



CENTANAFADINE 6 OF 14 PROTOCOL 405-201-00013

STAT-5.1
Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN)
(Efficacy Sample)

......

The Mixed Procedure




STAT-5.1
Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN)
(Efficacy Sample)

......

The Mixed Procedure



CENTANAFADINE


8 OF 14

STAT-5.1

Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN) (Efficacy Sample)

------ Parameter Code=CGI0201 ------

### The Mixed Procedure

### Dimensions

| Covariance | Parameters | 21 |
|------------|------------|-----|
| Columns in | X | 72 |
| Columns in | Z | 0 |
| Subjects | | 437 |
| Max Obs pe | r Subject | 6 |

### Number of Observations

| Number | of | Observations | Read | 2288 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 2288 |
| Number | of | Observations | Not Used | 0 |

### Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 5394.49812760 | |
| 1 | 2 | 3445.02451748 | 0.00188171 |
| 2 | 1 | 3444.38818261 | 0.00001015 |
| 3 | 1 | 3444.38487436 | 0.00000000 |


STAT-5.1

Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN) (Efficacy Sample)

The Mixed Procedure

Convergence criteria met.

### Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | |
| UN(2,1) | SUBJID | 0.2034 |
| UN(2,2) | SUBJID | 0.4814 |
| UN(3,1) | SUBJID | 0.1871 |
| UN(3,2) | SUBJID | 0.4119 |
| UN(3,3) | SUBJID | 0.6159 |
| UN(4,1) | SUBJID | 0.1907 |
| UN(4,2) | SUBJID | 0.3954 |
| UN(4,3) | SUBJID | 0.5303 |
| UN (4,4) | SUBJID | 0.6979 |
| UN(5,1) | SUBJID | 0.1737 |
| UN(5,2) | SUBJID | 0.4163 |
| UN(5,3) | SUBJID | 0.5399 |
| UN (5,4) | SUBJID | 0.5865 |
| UN(5,5) | SUBJID | 0.7044 |
| UN(6,1) | SUBJID | 0.2284 |
| UN(6,2) | SUBJID | 0.4456 |
| UN(6,3) | SUBJID | 0.5853 |

| CENTANAFADINE | 10 OF 14 |
|------------------------|----------|

STAT-5.

Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN) (Efficacy Sample)

......

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(6,4) | SUBJID | 0.6539 |
| UN(6,5) | SUBJID | 0.6649 |
| UN(6,6) | SUBJID | 0.8820 |

### Fit Statistics

| -2 Res Log Likelihood | 3444.4 |
|--------------------------|--------|
| AIC (Smaller is Better) | 3486.4 |
| AICC (Smaller is Better) | 3486.8 |
| BIC (Smaller is Better) | 3572.1 |

### Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|-----|------------|------------|
| 2.0 | 1050 11 | < 0001 |


# STAT-5.1 Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN) (Efficacy Sample)

------ Parameter Code=CGI0201 ------

The Mixed Procedure

### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------------|-----------|-----------|---------|--------|
| AVISITN | 5 | 380 | 2.29 | 0.0451 |
| TRTPN | 2 | 400 | 2.66 | 0.0431 |
| AVISITN*TRTPN | 10 | 562 | 1.94 | 0.0710 |
| | 37 | 395 | 1.94 | |
| POOLCNTR | | | | 0.0694 |
| BASE*AVISITN | 6 | 423 | 4.40 | 0.0003 |

### Estimates

| | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| DAY7 1 vs 3 | -0.07467 | 0.06756 | 397 | -1.11 | 0.2697 | 0.05 | -0.2075 | 0.05815 |
| DAY7 2 vs 3 | -0.01014 | 0.06743 | 397 | -0.15 | 0.8805 | 0.05 | -0.1427 | 0.1224 |
| DAY14 1 vs 3 | -0.04254 | 0.08369 | 401 | -0.51 | 0.6115 | 0.05 | -0.2071 | 0.1220 |
| DAY14 2 vs 3 | -0.04226 | 0.08328 | 398 | -0.51 | 0.6121 | 0.05 | -0.2060 | 0.1215 |
| DAY21 1 vs 3 | -0.1321 | 0.09557 | 392 | -1.38 | 0.1678 | 0.05 | -0.3200 | 0.05583 |
| DAY21 2 vs 3 | -0.1574 | 0.09468 | 385 | -1.66 | 0.0971 | 0.05 | -0.3436 | 0.02870 |
| DAY28 1 vs 3 | -0.1752 | 0.1030 | 403 | -1.70 | 0.0898 | 0.05 | -0.3778 | 0.02735 |
| DAY28 2 vs 3 | -0.2175 | 0.1019 | 396 | -2.13 | 0.0334 | 0.05 | -0.4178 | -0.01719 |

CENTANAFADINE 12 OF 14


# STAT-5.1 Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN) (Efficacy Sample)

.------

------Parameter Code=CGI0201 ------

### The Mixed Procedure

### Estimates

| | | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Label | | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| DAY35 | 1 vs 3 | -0.1864 | 0.1039 | 401 | -1.79 | 0.0736 | 0.05 | -0.3907 | 0.01789 |
| DAY35 | 2 vs 3 | -0.3316 | 0.1032 | 398 | -3.21 | 0.0014 | 0.05 | -0.5345 | -0.1288 |
| DAY42 | 1 vs 3 | -0.2664 | 0.1169 | 407 | -2.28 | 0.0232 | 0.05 | -0.4963 | -0.03659 |
| DAY42 | 2 vs 3 | -0.2789 | 0.1155 | 399 | -2.42 | 0.0162 | 0.05 | -0.5059 | -0.05194 |

### Least Squares Means

| 766 | Analysis<br>Visit | Planned<br>Treatment | <b>7</b> .1.1 | Standard | 25 | | 5. 2. 11.1 | 22.2 | • | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 7 | 1 | -0.3156 | 0.05150 | 409 | -6.13 | <.0001 | 0.05 | -0.4169 | -0.2144 |
| AVISITN*TRTPN | 7 | 2 | -0.2511 | 0.05228 | 413 | -4.80 | <.0001 | 0.05 | -0.3539 | -0.1483 |
| AVISITN*TRTPN | 7 | 3 | -0.2410 | 0.05226 | 411 | -4.61 | <.0001 | 0.05 | -0.3437 | -0.1383 |
| AVISITN*TRTPN | 14 | 1 | -0.4574 | 0.06241 | 434 | -7.33 | <.0001 | 0.05 | -0.5801 | -0.3348 |
| AVISITN*TRTPN | 14 | 2 | -0.4571 | 0.06273 | 440 | -7.29 | <.0001 | 0.05 | -0.5804 | -0.3339 |
| AVISITN*TRTPN | 14 | 3 | -0.4149 | 0.06281 | 439 | -6.61 | <.0001 | 0.05 | -0.5383 | -0.2914 |
| AVISITN*TRTPN | 21 | 1 | -0.5918 | 0.07085 | 432 | -8.35 | <.0001 | 0.05 | -0.7311 | -0.4526 |
| AVISITN*TRTPN | 21 | 2 | -0.6172 | 0.07042 | 432 | -8.76 | <.0001 | 0.05 | -0.7556 | -0.4788 |


# STAT-5.1 Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN) (Efficacy Sample)

------ Parameter Code=CGI0201 ------

The Mixed Procedure

Least Squares Means

| | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 21 | 3 | -0.4598 | 0.07038 | 430 | -6.53 | <.0001 | 0.05 | -0.5981 | -0.3214 |
| AVISITN*TRTPN | 28 | 1 | -0.6662 | 0.07633 | 445 | -8.73 | <.0001 | 0.05 | -0.8162 | -0.5162 |
| AVISITN*TRTPN | 28 | 2 | -0.7085 | 0.07549 | 445 | -9.38 | <.0001 | 0.05 | -0.8569 | -0.5601 |
| AVISITN*TRTPN | 28 | 3 | -0.4910 | 0.07503 | 437 | -6.54 | <.0001 | 0.05 | -0.6385 | -0.3435 |
| AVISITN*TRTPN | 35 | 1 | -0.6877 | 0.07674 | 439 | -8.96 | <.0001 | 0.05 | -0.8385 | -0.5369 |
| AVISITN*TRTPN | 35 | 2 | -0.8330 | 0.07652 | 449 | -10.89 | <.0001 | 0.05 | -0.9833 | -0.6826 |
| AVISITN*TRTPN | 35 | 3 | -0.5013 | 0.07580 | 435 | -6.61 | <.0001 | 0.05 | -0.6503 | -0.3523 |
| AVISITN*TRTPN | 42 | 1 | -0.7818 | 0.08592 | 443 | -9.10 | <.0001 | 0.05 | -0.9507 | -0.6130 |
| AVISITN*TRTPN | 42 | 2 | -0.7943 | 0.08453 | 440 | -9.40 | <.0001 | 0.05 | -0.9605 | -0.6282 |
| AVISITN*TRTPN | 42 | 3 | -0.5154 | 0.08437 | 438 | -6.11 | <.0001 | 0.05 | -0.6812 | -0.3496 |


CENTANAFADINE 14 OF 14

STAT-5.1

Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN) (Efficacy Sample)

The Mixed Procedure

Tests of Effect Slices

| | Analysis | | | | |
|---------------|----------|-----|-----|---------|--------|
| | Visit | Num | Den | | |
| Effect | (N) | DF | DF | F Value | Pr > F |
| AVISITN*TRTPN | 7 | 2 | 397 | 0.72 | 0.4872 |
| AVISITN*TRTPN | 14 | 2 | 400 | 0.17 | 0.8421 |
| AVISITN*TRTPN | 21 | 2 | 390 | 1.59 | 0.2056 |
| AVISITN*TRTPN | 28 | 2 | 402 | 2.56 | 0.0788 |
| AVISITN*TRTPN | 35 | 2 | 402 | 5.19 | 0.0059 |
| AVISITN*TRTPN | 42 | 2 | 405 | 3.70 | 0.0257 |


STAT-5.2

Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, LOCF (Efficacy Sample)

\_\_\_\_\_

The GLM Procedure

Class Level Information

Class Levels Values
TRTPN 3 1 2 3

POOLCNTR 38

Number of Observations Read 437 Number of Observations Used 437

CENTANAFADINE 2 OF 6

PROTOCOL 405-201-00013 STAT-5.2

Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, LOCF (Efficacy Sample)

......

The GLM Procedure

Dependent Variable: CHG Change from Baseline

| Source | | DF | Sum o<br>Square | | Square | F Value | Pr > F |
|---|---|---|---|---|---|---|---|
| Model | | 40 | 46.660795 | 2 1.1 | 1665199 | 1.38 | 0.0659 |
| Error | | 396 | 333.888403 | 9 0.8 | 3431525 | | |
| Corrected Total | | 436 | 380.549199 | 1 | | | |
| | R-Square | Coef | f Var | Root MSE | CHG M | ean | |
| | 0.122614 | -136 | .9515 | 0.918233 | -0.670 | 481 | |
| Source | | DF | Type III S | S Mean | Square | F Value | Pr > F |
| TRTPN<br>POOLCNTR<br>BASE | | 2<br>37<br>1 | 4.3720202<br>31.8559979<br>9.9661752 | 3 0.86 | 3601011<br>5097292<br>5617520 | 2.59<br>1.02<br>11.82 | 0.0761<br>0.4390<br>0.0006 |


 $$\tt STAT-5.2$$  Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, LOCF (Efficacy Sample)

### The GLM Procedure

| Level of | | CHC | 3 | BAS | SE |
|----------|-----|-------------|------------|------------|------------|
| TRTPN | N | Mean | Std Dev | Mean | Std Dev |
| 1 | 146 | -0.71917808 | 1.02212187 | 4.47945205 | 0.60136830 |
| 2 | 147 | -0.76190476 | 0.94603233 | 4.53061224 | 0.60029813 |
| 3 | 144 | -0.52777778 | 0.81028739 | 4.51388889 | 0.55452507 |


 $$\tt STAT-5.2$$  Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, LOCF (Efficacy Sample)

The GLM Procedure Least Squares Means

| TRTPN | CHG LSMEAN | Standard<br>Error | Pr > t | Number |
|-------|-------------|-------------------|---------|--------|
| 1 | -0.71916295 | 0.08370474 | <.0001 | 1 |
| 2 | -0.72793134 | 0.08502853 | <.0001 | 2 |
| 3 | -0.50965777 | 0.08513983 | <.0001 | 3 |

Least Squares Means for effect TRTPN
Pr > |t| for H0: LSMean(i)=LSMean(j)

### Dependent Variable: CHG

| i/j | 1 | 2 | 3 |
|---|---|---|---|
| 1<br>2<br>3 | 0.9353<br>0.0543 | 0.9353 0.054<br>0.044 | |
| TRTPN | CHG LSMEAN | 95% Confidence Limit | s |
| 1<br>2 | -0.719163<br>-0.727931 | -0.883724 -0.554<br>-0.895095 -0.560 | |


STAT-5.2

Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, LOCF (Efficacy Sample)

The GLM Procedure Least Squares Means

TRTPN CHG LSMEAN 95% Confidence Limits

3 -0.509658 -0.677040 -0.342275

Least Squares Means for Effect TRTPN

Difference
Between 95% Confidence Limits for
i j Means LSMean(i)-LSMean(j)

1 2 0.008768 -0.203504 0.221040
1 3 -0.209505 -0.422864 0.003854
2 3 -0.218274 -0.431132 -0.005415

NOTE: To ensure overall protection level, only probabilities associated with pre-planned comparisons should be used.


STAT-5.2

Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, LOCF (Efficacy Sample)

The GLM Procedure

Dependent Variable: CHG Change from Baseline

| Parameter | Estimate | Standard<br>Error | t Value | Pr > t |
|-----------|-------------|-------------------|---------|---------|
| 1 vs 3 | -0.20950519 | 0.10852592 | -1.93 | 0.0543 |
| 2 vs 3 | -0.21827357 | 0.10827131 | -2.02 | 0.0445 |


STAT-5.3

Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, OC (Efficacy Sample)

\_\_\_\_\_

The GLM Procedure

Class Level Information

Class Levels Values
TRTPN 3 1 2 3

Number of Observations Read 437 Number of Observations Used 437


> STAT-5.3 Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, OC (Efficacy Sample)

The GLM Procedure

Dependent Variable: CHG Change from Baseline

| Source | | DF | Sum (<br>Square | | Mean S | Square | F Value | Pr > F |
|---|---|---|---|---|---|---|---|---|
| Model | | 3 | 14.80479 | 73 | 4.93 | 349324 | 5.84 | 0.0006 |
| Error | | 433 | 365.74440 | 18 | 0.84 | 146753 | | |
| Corrected Total | | 436 | 380.54919 | 91 | | | | |
| | R-Square<br>0.038904 | | f Var<br>.0751 | Root M:<br>0.9190 | | CHG Mea | | |
| Source | | DF | Type III : | SS 1 | Mean 9 | Square | F Value | Pr > F |
| TRTPN<br>BASE | | 2 1 | 4.531629-<br>10.297455 | 49 | 2.265 | 581475<br>745513 | 2.68<br>12.19 | 0.0695 |

SOURCE: GLMOUT; TABLE: stat1cgisc.lis; RUN: 18JUN2020 10:00; ANALYSIS DATASET CREATED: 11JUN2020 07:28 PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-5.3 FINAL


STAT-5.3 Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, OC (Efficacy Sample)

### The GLM Procedure

| Level of | | СНО | ; | BAS | E |
|----------|-----|-------------|------------|------------|------------|
| TRTPN | N | Mean | Std Dev | Mean | Std Dev |
| 1 | 146 | -0.71917808 | 1.02212187 | 4.47945205 | 0.60136830 |
| 2 | 147 | -0.76190476 | 0.94603233 | 4.53061224 | 0.60029813 |
| 3 | 144 | -0.52777778 | 0.81028739 | 4.51388889 | 0.55452507 |


## STAT-5.3

Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, OC (Efficacy Sample)

\_\_\_\_\_

### The GLM Procedure Least Squares Means

| | | Standard | | LSMEAN |
|-------|-------------|------------|---------|--------|
| TRTPN | CHG LSMEAN | Error | Pr > t | Number |
| 1 | -0.72668484 | 0.07609251 | <.0001 | 1 |
| 2 | -0.75596312 | 0.07582207 | <.0001 | 2 |
| 3 | -0.52623218 | 0.07658979 | <.0001 | 3 |

Least Squares Means for effect TRTPN Pr > |t| for H0: LSMean(i)=LSMean(j)

### Dependent Variable: CHG

| i/j | 1 | 2 | 3 |
|---|---|---|---|
| 1<br>2<br>3 | 0.7854<br>0.0641 | 0.7854 | 0.0641<br>0.0336 |
| TRTPN | CHG LSMEAN | 95% Confidence | ce Limits |
| 1<br>2 | -0.726685<br>-0.755963 | -0.876241<br>-0.904988 | -0.577128<br>-0.606938 |


STAT-5.3

Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, OC (Efficacy Sample)

The GLM Procedure Least Squares Means

TRTPN CHG LSMEAN 95% Confidence Limits

3 -0.526232 -0.676766 -0.375698

Least Squares Means for Effect TRTPN

Difference
Between 95% Confidence Limits for
i j Means LSMean(i)-LSMean(j)

1 2 0.029278 -0.181918 0.240475
1 3 -0.200453 -0.412667 0.011762
2 3 -0.229731 -0.441540 -0.017922

NOTE: To ensure overall protection level, only probabilities associated with pre-planned comparisons should be used.

CENTANAFADINE 6 OF 6


STAT-5.3

Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, OC (Efficacy Sample)

The GLM Procedure

Dependent Variable: CHG Change from Baseline

| Parameter | Estimate | Standard<br>Error | t Value | Pr > t |
|-----------|-------------|-------------------|---------|---------|
| 1 vs 3 | -0.20045266 | 0.10797208 | -1.86 | 0.0641 |
| 2 vs 3 | -0.22973094 | 0.10776584 | -2.13 | 0.0336 |

CENTANAFADINE 1 OF 1 PROTOCOL 405-201-00013

STAT-6.1.1
Shapiro-Wilk Test for Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_\_

| | | | | GOODNESS OF FIT | |
|---|---|---|---|---|---|
| | | TEST | GOODNESS OF FIT | TEST | |
| PROTOCOL | Day | VARIABLE | TEST | STATISTICS | Pvalue |
| 40520100013 | DAY 7 | RESID | Shapiro-Wilk | 0.9505 | <0.0001 |
| | | STUDENTRESID | Shapiro-Wilk | 0.9512 | <0.0001 |
| | DAY 14 | RESID | Shapiro-Wilk | 0.9461 | <0.0001 |
| | | STUDENTRESID | Shapiro-Wilk | 0.9474 | <0.0001 |
| | DAY 21 | RESID | Shapiro-Wilk | 0.9557 | <0.0001 |
| | | STUDENTRESID | Shapiro-Wilk | 0.9575 | <0.0001 |
| | DAY 28 | RESID | Shapiro-Wilk | 0.9600 | <0.0001 |
| | | STUDENTRESID | Shapiro-Wilk | 0.9604 | <0.0001 |
| | DAY 35 | RESID | Shapiro-Wilk | 0.9643 | <0.0001 |
| | | STUDENTRESID | Shapiro-Wilk | 0.9645 | <0.0001 |
| | DAY 42 | RESID | Shapiro-Wilk | 0.9468 | <0.0001 |
| | | STUDENTRESID | Shapiro-Wilk | 0.9468 | <0.0001 |

.\_\_\_\_\_

FILE: normality ba.lis, RUN: 18JUN2020 10:00

PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC\_STAT/normality\_b.sas
OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-6.1.1 FINAL

CENTANAFADINE 1 OF 48 PROTOCOL 405-201-00013

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

The UNIVARIATE Procedure Variable: RESID (Residual)

#### Moments

| N | 429 | Sum Weights | 429 |
|-----------------|------------|------------------|------------|
| Mean | -0.0358232 | Sum Observations | -15.368154 |
| Std Deviation | 6.92317198 | Variance | 47.9303103 |
| Skewness | -0.8989502 | Kurtosis | 1.59121128 |
| Uncorrected SS | 20514.7234 | Corrected SS | 20514.1728 |
| Coeff Variation | -19325.943 | Std Error Mean | 0.33425389 |

### Basic Statistical Measures

Location Variability

| Mean | -0.03582 | Std Deviation | 6.92317 |
|--------|----------|---------------------|----------|
| Median | 1.02764 | Variance | 47.93031 |
| Mode | -5.95541 | Range | 44.54954 |
| | | Interguartile Range | 7.44768 |

Note: The mode displayed is the smallest of 2 modes with a count of 2.

-----

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-6.1.2 FINAL

| CENTANAFADINE | 2 OF 48 |
|---------------|---------|


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

Tests for Location: Mu0=0

| Test | -S | tatistic- | p Valı | ue |
|-------------|----|-----------|----------|--------|
| Student's t | t | -0.10717 | Pr > t | 0.9147 |
| Sign | M | 30.5 | Pr >= M | 0.0037 |
| Signed Rank | S | 4507.5 | Pr >= S | 0.0794 |

### Tests for Normality

| Test | Sta | tistic | p Va | lue |
|--------------------|------|----------|-----------|---------|
| Shapiro-Wilk | W | 0.950477 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.096707 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 1.114552 | Pr > W-Sq | <0.0050 |
| Anderson-Darling | A-Sq | 6.25502 | Pr > A-Sq | <0.0050 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-6.1.2 FINAL

| CENTANAFADINE | 3 OF 48 |
|------------------------|---------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

Quantiles (Definition 5)

| Level | Quantile |
|------------|-----------|
| 100% Max | 18.12976 |
| 99% | 14.28640 |
| 95% | 9.63500 |
| 90% | 7.03550 |
| 75% Q3 | 4.19872 |
| 50% Median | 1.02764 |
| 25% Q1 | -3.24896 |
| 10% | -9.50864 |
| 5% | -13.14533 |
| 1% | -22.53575 |
| 0% Min | -26.41979 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-6.1.2 FINA

CENTANAFADINE

4 OF 48

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

(ZZZZGG) Cumpz

------ Analysis Visit (N)=7 ------

The UNIVARIATE Procedure
Variable: RESID (Residual)

Extreme Observations

| | Lowest | | | | Highest |
|----------|--------------|-----|---------|--------------|---------|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -26.4198 | 40520100013- | 31 | 14.2864 | 40520100013- | 253 |
| -25.0595 | 40520100013- | 241 | 14.5137 | 40520100013- | 127 |
| -24.7070 | 40520100013- | 345 | 15.9196 | 40520100013- | 344 |
| -23.8012 | 40520100013- | 126 | 17.4347 | 40520100013- | 336 |
| -22.5358 | 40520100013- | 215 | 18.1298 | 40520100013- | 348 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-6.1.2 FINAL

CENTANAFADINE 5 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Moments

 N
 429
 Sum Weights
 429

 Mean
 -0.0055696
 Sum Observations
 -2.3893447

 Std Deviation
 0.99907873
 Variance
 0.99815832

 Skewness
 -0.8889627
 Kurtosis
 1.51349761

 Uncorrected SS
 427.225068
 Corrected SS
 427.21176

 Coeff Variation
 -17938.172
 Std Error Mean
 0.04823598

Basic Statistical Measures

Location Variability

 Mean
 -0.00557
 Std Deviation
 0.99908

 Median
 0.14511
 Variance
 0.99816

 Mode
 -0.84411
 Range
 6.28819

 Interquartile Range
 1.08259

Note: The mode displayed is the smallest of 2 modes with a count of 2.

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-6.1.2 FINAL

| CENTANAFADINE | 6 OF 48 |
|------------------------|---------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: STUDENTRESID (Studentized Residual)

Tests for Location: Mu0=0

Test -Statistic- ----p Value-----Student's t t -0.11547 Pr > |t| 0.9081 Sign M 30.5 Pr >= |M| 0.0037 Signed Rank S 4427.5 Pr >= |S| 0.0849

Tests for Normality

| Test | Sta | tistic | p Val | ue |
|--------------------|------|----------|-----------|---------|
| Shapiro-Wilk | W | 0.951168 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.096496 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 1.109796 | Pr > W-Sq | <0.0050 |
| Anderson-Darling | A-Sq | 6.205792 | Pr > A-Sq | <0.0050 |

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC STAT/normality.sas OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-6.1.2

| CENTANAFADINE 7 OF 48 |
|------------------------|
| CENTANAFADINE // OF 40 |


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

### The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Quantiles (Definition 5)

| Level | Quantile |
|---|---|
| 100% Max<br>99%<br>95%<br>90%<br>75% Q3<br>50% Median<br>25% Q1 | 2.547354<br>2.106636<br>1.406654<br>1.041059<br>0.623263<br>0.145113<br>-0.459331 |
| 10% | -1.394934<br>-1 925385 |
| ~ | |
| 5%<br>1% | -1.925385<br>-3.293143 |
| 0% Min | -3.740832 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-6.1.2 FIN

CENTANAFADINE 8 OF 48 PROTOCOL 405-201-00013

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------

The UNIVARIATE Procedure
Variable: STUDENTRESID (Studentized Residual)

Extreme Observations

| Lowest | | | | Highest | |
|----------|--------------|-----|---------|--------------|-----|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -3.74083 | 40520100013- | 31 | 2.10664 | 40520100013- | 253 |
| -3.59734 | 40520100013- | 241 | 2.14602 | 40520100013- | 127 |
| -3.51327 | 40520100013- | 126 | 2.23609 | 40520100013- | 344 |
| -3.47412 | 40520100013- | 345 | 2.45134 | 40520100013- | 336 |
| -3.29314 | 40520100013- | 215 | 2.54735 | 40520100013- | 348 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-6.1.2 FINAL

CENTANAFADINE 9 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

The UNIVARIATE Procedure Variable: RESID (Residual)

### Moments

| N | 406 | Sum Weights | 406 |
|-----------------|------------|------------------|------------|
| Mean | -0.0512213 | Sum Observations | -20.795843 |
| Std Deviation | 8.29126377 | Variance | 68.745055 |
| Skewness | -0.918599 | Kurtosis | 0.87158088 |
| Uncorrected SS | 27842.8125 | Corrected SS | 27841.7473 |
| Coeff Variation | -16187.144 | Std Error Mean | 0.41148851 |

### Basic Statistical Measures

Location Variability

| Mean | -0.05122 | Std Deviation | 8.29126 |
|--------|----------|---------------------|----------|
| Median | 1.44518 | Variance | 68.74505 |
| Mode | -4.28518 | Range | 45.92221 |
| | | Interquartile Range | 10 09103 |

Note: The mode displayed is the smallest of 4 modes with a count of 2.

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-6.1.2 FINAL
| 0 OF 48 |
|---------|
|---------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------ Analysis Visit (N)=14 ------

The UNIVARIATE Procedure Variable: RESID (Residual)

Tests for Location: Mu0=0

| Test | -Statistic- | p Value |
|-------------|-------------|------------------|
| Student's t | t -0.12448 | Pr > t 0.9010 |
| Sign | M 33 | Pr >= M 0.0012 |
| Signed Rank | S 4233.5 | Pr >= S 0.0735 |

#### Tests for Normality

| Test | Sta | tistic | p V | alue |
|--------------------|------|----------|----------|-----------|
| Shapiro-Wilk | W | 0.946146 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.091654 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 1.123579 | Pr > W-S | q <0.0050 |
| Anderson-Darling | A-Sq | 6.515695 | Pr > A-S | q <0.0050 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| CENTANAFADINE | 11 OF 48 |
|---------------|----------|
|---------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

.------

The UNIVARIATE Procedure Variable: RESID (Residual)

Quantiles (Definition 5)

| Level | Quantile |
|-----------------|----------------------|
| 100% Max<br>99% | 18.12438<br>15.31626 |
| 95% | 10.82306 |
| 90% | 8.96116 |
| 75% Q3 | 5.77732 |
| 50% Median | 1.44518 |
| 25% Q1 | -4.31372 |
| 10% | -11.65152 |
| 5% | -16.87371 |
| 1% | -25.37928 |
| 0% Min | -27.79784 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 12 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------

The UNIVARIATE Procedure Variable: RESID (Residual)

Extreme Observations

Highogt

| Lowest | | | | Hignest | |
|----------|--------------|-----|---------|--------------|-----|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -27.7978 | 40520100013- | 729 | 15.3163 | 40520100013- | 630 |
| -26.3480 | 40520100013- | 701 | 15.4412 | 40520100013- | 549 |
| -26.1345 | 40520100013- | 586 | 15.9561 | 40520100013- | 747 |
| -25.7353 | 40520100013- | 459 | 17.3297 | 40520100013- | 748 |
| -25.3793 | 40520100013- | 664 | 18.1244 | 40520100013- | 746 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 13 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Moments

| N | 406 | Sum Weights | 406 |
|-----------------|------------|------------------|------------|
| Mean | -0.0056236 | Sum Observations | -2.283187 |
| Std Deviation | 1.0070444 | Variance | 1.01413842 |
| Skewness | -0.9021239 | Kurtosis | 0.83485956 |
| Uncorrected SS | 410.738899 | Corrected SS | 410.726059 |
| Coeff Variation | -17907.426 | Std Error Mean | 0.04997877 |

Basic Statistical Measures

Location Variability

| Mean | -0.00562 | Std Deviation | 1.00704 |
|--------|----------|---------------------|---------|
| Median | 0.17363 | Variance | 1.01414 |
| Mode | -0.51324 | Range | 5.55938 |
| | | Interquartile Range | 1 22582 |

Note: The mode displayed is the smallest of 4 modes with a count of 2.

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| OF | 4 | 8 | |
|----|----|------|-------|
| | OF | OF 4 | OF 48 |

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Tests for Location: Mu0=0

| Test | -S | tatistic- | p Valı | ue |
|-------------|----|-----------|----------|--------|
| Student's t | t | -0.11252 | Pr > t | 0.9105 |
| Sign | M | 33 | Pr >= M | 0.0012 |
| Signed Rank | S | 4183.5 | Pr >= S | 0.0770 |

#### Tests for Normality

| Test | Sta | tistic | p Va | lue |
|--------------------|------|----------|-----------|---------|
| Shapiro-Wilk | W | 0.947415 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.091557 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 1.124298 | Pr > W-Sq | <0.0050 |
| Anderson-Darling | A-Sq | 6.464081 | Pr > A-Sq | <0.0050 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_

## The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Quantiles (Definition 5)

| Level | Quantile |
|---------------|------------------------|
| 100% Max | 2.162711 |
| 99% | 1.902737 |
| 95% | 1.310225 |
| 90%<br>75% Q3 | 1.083757 |
| 50% Median | 0.173632 |
| 25% Q1 | -0.519422 |
| 10% | -1.416902<br>-2.033019 |
| 1% | -3.115779 |
| 0% Min | -3.396667 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 16 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------

------ Analysis Visit (N)=14 ------

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Extreme Observations

| Howest | | | | nighesc | | |
|----------|--------------|----|---------|-----------------|---|-----|
| Value | USUBJID | Ob | s Val | ue USUBJID | | Obs |
| -3.39667 | 40520100013- | 72 | 9 1.902 | 74 40520100013- | - | 747 |
| -3.16989 | 40520100013- | 70 | 1 1.905 | 42 40520100013- | - | 549 |
| -3.12956 | 40520100013- | 66 | 4 2.011 | 27 40520100013- | - | 554 |
| -3.11745 | 40520100013- | 54 | 7 2.066 | 17 40520100013- | - | 748 |
| -3.11578 | 40520100013- | 58 | 6 2.162 | 71 40520100013- | - | 746 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 17 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

The UNIVARIATE Procedure Variable: RESID (Residual)

#### Moments

| N | 391 | Sum Weights | 391 |
|-----------------|------------|------------------|------------|
| Mean | -0.1603789 | Sum Observations | -62.708169 |
| Std Deviation | 8.75757561 | Variance | 76.6951306 |
| Skewness | -0.7967468 | Kurtosis | 0.37509191 |
| Uncorrected SS | 29921.158 | Corrected SS | 29911.101 |
| Coeff Variation | -5460.5518 | Std Error Mean | 0.44288964 |

## Basic Statistical Measures

# Location Variability

| Mean | -0.16038 | Std Deviation | 8.75758 |
|--------|----------|---------------------|----------|
| Median | 1.40218 | Variance | 76.69513 |
| Mode | -4.23564 | Range | 49.66442 |
| | | Interquartile Range | 11.21801 |

Note: The mode displayed is the smallest of 3 modes with a count of 2.

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| .8 OF 48 |
|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_

------ Analysis Visit (N)=21 ------

The UNIVARIATE Procedure Variable: RESID (Residual)

Tests for Location: Mu0=0

| Test | -St | atistic- | p Va | lue |
|-------------|-----|----------|----------|--------|
| Student's t | t | -0.36212 | Pr > t | 0.7175 |
| Sign | M | 24.5 | Pr >= M | 0.0151 |
| Signed Rank | S | 2593 | Pr >= S | 0.2467 |

#### Tests for Normality

| Test | Sta | tistic | p Val | ue |
|--------------------|------|----------|-----------|---------|
| Shapiro-Wilk | W | 0.95566 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.082594 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.827025 | Pr > W-Sq | <0.0050 |
| Anderson-Darling | A-Sq | 5.002996 | Pr > A-Sq | <0.0050 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| CENTANAFADINE | 19 OF 48 |
|------------------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

Quantiles (Definition 5)

| Level | Quantile |
|------------|-----------|
| 100% Max | 17.73069 |
| 99% | 14.32811 |
| 95% | 11.25169 |
| 90% | 9.52209 |
| 75% O3 | 6.20743 |
| 50% Median | 1.40218 |
| 25% Q1 | -5.01058 |
| 10% | -12.76245 |
| 5% | -17.32377 |
| 1% | -23.46337 |
| 0% Min | -31.93373 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 20 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------

------ Analysis Visit (N)=21 ------

The UNIVARIATE Procedure
Variable: RESID (Residual)

Extreme Observations

| Howest | | | 1111 | 911000 | |
|----------|-------------|------|---------|--------------|------|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -31.9337 | 40520100013 | 988 | 14.1209 | 40520100013- | 1020 |
| -30.9690 | 40520100013 | 1101 | 14.3281 | 40520100013- | 1146 |
| -24.7107 | 40520100013 | 1129 | 14.3988 | 40520100013- | 1192 |
| -23.4634 | 40520100013 | 865 | 15.9977 | 40520100013- | 958 |
| -22.6585 | 40520100013 | 952 | 17.7307 | 40520100013- | 955 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 21 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Moments

| N | 391 | Sum Weights | 391 |
|-----------------|------------|------------------|------------|
| Mean | -0.0173302 | Sum Observations | -6.7761143 |
| Std Deviation | 1.0026023 | Variance | 1.00521137 |
| Skewness | -0.7767798 | Kurtosis | 0.33565986 |
| Uncorrected SS | 392.149864 | Corrected SS | 392.032433 |
| Coeff Variation | -5785.2846 | Std Error Mean | 0.05070378 |

Basic Statistical Measures

Location Variability

| Mean | -0.01733 | Std Deviation | 1.00260 |
|--------|----------|---------------------|---------|
| Median | 0.15766 | Variance | 1.00521 |
| Mode | -0.47523 | Range | 5.64738 |
| | | Interquartile Range | 1.29404 |

Note: The mode displayed is the smallest of 3 modes with a count of 2.

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

------ Analysis Visit (N)=21 ------

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Tests for Location: Mu0=0

| Test | -Sta | tistic- | p Valu | le |
|-------------|------|----------|----------|--------|
| Student's t | t - | -0.34179 | Pr > t | 0.7327 |
| Sign | M | 24.5 | Pr >= M | 0.0151 |
| Signed Rank | S | 2567 | Pr >= S | 0.2515 |

#### Tests for Normality

| Test | Sta | tistic | p Va | lue |
|--------------------|------|----------|-----------|---------|
| Shapiro-Wilk | W | 0.957454 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.082316 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.809936 | Pr > W-Sq | <0.0050 |
| Anderson-Darling | A-Sq | 4.874627 | Pr > A-Sq | (0.0050 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| OF 48 |
|-------|
|-------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Quantiles (Definition 5)

| Level | Quantile |
|---|---|
| 100% Max<br>99%<br>95%<br>90%<br>75% Q3<br>50% Median<br>25% Q1 | 2.056753<br>1.617161<br>1.320311<br>1.079049<br>0.709824<br>0.157662<br>-0.584218<br>-1.446331 |
| 5% | -2.015562 |
| 1% | -2.649605 |
| 0% Min | -3.590625 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 24 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------

The UNIVARIATE Procedure
Variable: STUDENTRESID (Studentized Residual)

Extreme Observations

| Lowest | | | Highest | | |
|----------|--------------|------|---------|--------------|------|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -3.59062 | 40520100013- | 988 | 1.61159 | 40520100013- | 1146 |
| -3.51155 | 40520100013- | 1101 | 1.61716 | 40520100013- | 1020 |
| -2.83912 | 40520100013- | 1129 | 1.63078 | 40520100013- | 1192 |
| -2.64961 | 40520100013- | 865 | 1.99613 | 40520100013- | 958 |
| -2.63088 | 40520100013- | 952 | 2.05675 | 40520100013- | 955 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 25 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure
Variable: RESID (Residual)

#### Moments

| N | 370 | Sum Weights | 370 |
|-----------------|------------|------------------|------------|
| Mean | -0.4073769 | Sum Observations | -150.72947 |
| Std Deviation | 10.1669831 | Variance | 103.367545 |
| Skewness | -0.7010249 | Kurtosis | 0.12558616 |
| Uncorrected SS | 38204.0278 | Corrected SS | 38142.6241 |
| Coeff Variation | -2495.7189 | Std Error Mean | 0.52855628 |

## Basic Statistical Measures

Location Variability

| Mean | -0.40738 | Std Deviation | 10.16698 |
|--------|----------|---------------------|-----------|
| Median | 1.71750 | Variance | 103.36754 |
| Mode | 7.54797 | Range | 54.45127 |
| | | Interquartile Range | 14.48720 |

Note: The mode displayed is the smallest of 2 modes with a count of 2.

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| CENTANAFADINE 26 0 | OF 48 |
|--------------------|-------|
|--------------------|-------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------ Analysis Visit (N)=28 ------

The UNIVARIATE Procedure Variable: RESID (Residual)

Tests for Location: Mu0=0

| Test | -Statistic- | p Value |
|-------------|-------------|--------------------|
| Student's t | t -0.77074 | Pr > t 0.4414 |
| Sign | M 25 | Pr >= M 0.0108 |
| Signed Rank | S 1007.5 | Pr >= S = 0.6252 |

#### Tests for Normality

| Test | Sta | tistic | p V | alue |
|--------------------|------|----------|----------|-----------|
| Shapiro-Wilk | W | 0.959992 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.090634 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.856785 | Pr > W-S | q <0.0050 |
| Anderson-Darling | A-Sq | 4.871079 | Pr > A-S | q <0.0050 |

------

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| CENTANAFADINE | 27 OF 48 |
|------------------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------ Analysis Visit (N)=28 -------

The UNIVARIATE Procedure Variable: RESID (Residual)

Quantiles (Definition 5)

| Level | Quantile |
|------------|-----------|
| 100% Max | 20.54164 |
| 99% | 18.23384 |
| 95% | 12.28388 |
| 90% | 10.47477 |
| 75% Q3 | 7.54797 |
| 50% Median | 1.71750 |
| 25% Q1 | -6.93923 |
| 10% | -14.81352 |
| 5% | -20.55486 |
| 1% | -29.58661 |
| 0% Min | -33.90962 |

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC STAT/normality.sas

OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-6.1.2

CENTANAFADINE 28 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_\_

------ Analysis Visit (N)=28 ------

The UNIVARIATE Procedure Variable: RESID (Residual)

Extreme Observations

Highogt

| Dowest | | | | n. | ignest |
|----------|--------------|------|---------|--------------|--------|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -33.9096 | 40520100013- | 1498 | 18.2304 | 40520100013- | 1344 |
| -31.7656 | 40520100013- | 1517 | 18.2338 | 40520100013- | 1519 |
| -31.3573 | 40520100013- | 1478 | 19.0985 | 40520100013- | 1518 |
| -29.5866 | 40520100013- | 1372 | 20.0136 | 40520100013- | 1589 |
| -28.0541 | 40520100013- | 1504 | 20.5416 | 40520100013- | 1341 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 29 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Moments

| N | 370 | Sum Weights | 370 |
|-----------------|------------|------------------|------------|
| Mean | -0.040986 | Sum Observations | -15.164837 |
| Std Deviation | 1.01442638 | Variance | 1.02906089 |
| Skewness | -0.6955724 | Kurtosis | 0.11422617 |
| Uncorrected SS | 380.345015 | Corrected SS | 379.723468 |
| Coeff Variation | -2475.053 | Std Error Mean | 0.05273752 |

Basic Statistical Measures

Location Variability

| Mean | -0.04099 | Std Deviation | 1.01443 |
|--------|----------|---------------------|---------|
| Median | 0.16987 | Variance | 1.02906 |
| Mode | 0.74219 | Range | 5.47903 |
| | | Interquartile Range | 1 45931 |

Note: The mode displayed is the smallest of 2 modes with a count of 2.

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| CENTANAFADINE | 30 OF 48 |
|---------------|----------|
|---------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------ Analysis Visit (N)=28 ------

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Tests for Location: Mu0=0

| Test | -Statistic- | p Value |
|-------------|-------------|------------------|
| Student's t | t -0.77717 | Pr > t 0.4376 |
| Sign | M 25 | Pr >= M 0.0108 |
| Signed Rank | S 976.5 | Pr >= S 0.6359 |

#### Tests for Normality

| Test | Sta | tistic | p Va | alue |
|--------------------|------|----------|-----------|-----------|
| Shapiro-Wilk | W | 0.96038 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.09143 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.859455 | Pr > W-So | q <0.0050 |
| Anderson-Darling | A-Sq | 4.871 | Pr > A-So | q <0.0050 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| CENTANAFADINE | 31 OF 48 |
|---------------|----------|
|---------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

## The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Quantiles (Definition 5)

| Level | Quantile |
|-----------------|------------------------|
| 100% Max<br>99% | 2.070287 |
| 95% | 1.228575 |
| 90%<br>75% O3 | 1.053543 |
| 50% Median | 0.169875 |
| 25% Q1<br>10% | -0.711522<br>-1.471843 |
| 5% | -2.092184 |
| 1%<br>0% Min | -2.912932<br>-3.408746 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 32 OF 48 PROTOCOL 405-201-00013

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------

------- Analysis Visit (N)=28 ------

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Extreme Observations

| Lowest | | | | -iiigiiesc | | |
|--------|----------|--------------|------|------------|--------------|------|
| | Value | USUBJID | Obs | Value | USUBJID | Obs |
| | -3.40875 | 40520100013- | 1498 | 1.79657 | 40520100013- | 1519 |
| | -3.13286 | 40520100013- | 1517 | 1.88169 | 40520100013- | 1518 |
| | -3.10958 | 40520100013- | 1478 | 1.93934 | 40520100013- | 1344 |
| | -2.91293 | 40520100013- | 1372 | 1.97622 | 40520100013- | 1589 |
| | -2.80668 | 40520100013- | 1504 | 2.07029 | 40520100013- | 1341 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 33 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

The UNIVARIATE Procedure Variable: RESID (Residual)

#### Moments

| N | 349 | Sum Weights | 349 |
|-----------------|------------|------------------|------------|
| Mean | -0.4303981 | Sum Observations | -150.20894 |
| Std Deviation | 10.4068682 | Variance | 108.302907 |
| Skewness | -0.5781918 | Kurtosis | -0.263225 |
| Uncorrected SS | 37754.0612 | Corrected SS | 37689.4115 |
| Coeff Variation | -2417.9632 | Std Error Mean | 0.55706689 |

## Basic Statistical Measures

Location Variability

| Mean | -0.43040 | Std Deviation | 10.40687 |
|--------|----------|---------------------|-----------|
| Median | 1.66772 | Variance | 108.30291 |
| Mode | -6.91304 | Range | 55.34813 |
| | | Interquartile Range | 14.82125 |

Note: The mode displayed is the smallest of 5 modes with a count of 2.

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| CENTANAFADINE | 34 OF 48 |
|---------------|----------|
|---------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

Tests for Location: Mu0=0

| Test | -Sta | tistic- | p Val | .ue |
|-------------|------|---------|----------|--------|
| Student's t | t - | 0.77261 | Pr > t | 0.4403 |
| Sign | M | 15.5 | Pr >= M | 0.1082 |
| Signed Rank | S | 345.5 | Pr >= S | 0.8550 |

#### Tests for Normality

| Test | Stat | istic | p Val | ue |
|--------------------|------|----------|-----------|---------|
| Shapiro-Wilk | W | 0.964262 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.092832 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.74979 | Pr > W-Sq | <0.0050 |
| Anderson-Darling | A-Sq | 4.328771 | Pr > A-Sq | <0.0050 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| CENTANAFADINE | 35 OF 48 |
|------------------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_\_

The UNIVARIATE Procedure Variable: RESID (Residual)

Quantiles (Definition 5)

| Level | Quantile |
|------------|-----------|
| 100% Max | 22.75938 |
| 99% | 17.91271 |
| 95% | 12.68687 |
| 90% | 10.84392 |
| 75% Q3 | 7.40753 |
| 50% Median | 1.66772 |
| 25% Q1 | -7.41372 |
| 10% | -15.22456 |
| 5% | -20.06777 |
| 1% | -26.48683 |
| 0% Min | -32.58874 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 36 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------

------ Analysis Visit (N)=35 ------

The UNIVARIATE Procedure Variable: RESID (Residual)

Extreme Observations

Highogt

| | | | nighest- | | |
|----------|--------------|------|----------|--------------|------|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -32.5887 | 40520100013- | 1852 | 17.4072 | 40520100013- | 1877 |
| -31.9099 | 40520100013- | 1833 | 17.9127 | 40520100013- | 1872 |
| -26.7640 | 40520100013- | 1731 | 17.9954 | 40520100013- | 1891 |
| -26.4868 | 40520100013- | 1694 | 18.6219 | 40520100013- | 1938 |
| -26.1038 | 40520100013- | 1857 | 22.7594 | 40520100013- | 1702 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 37 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Moments

| N | 349 | Sum Weights | 349 |
|-----------------|------------|------------------|------------|
| Mean | -0.0428873 | Sum Observations | -14.967661 |
| Std Deviation | 1.0147428 | Variance | 1.02970295 |
| Skewness | -0.5766127 | Kurtosis | -0.2605306 |
| Uncorrected SS | 358.978549 | Corrected SS | 358.336627 |
| Coeff Variation | -2366.0694 | Std Error Mean | 0.05431794 |

Basic Statistical Measures

Location Variability

| Mean | -0.04289 | Std Deviation | 1.01474 |
|--------|----------|---------------------|---------|
| Median | 0.16924 | Variance | 1.02970 |
| Mode | -0.67533 | Range | 5.44081 |
| | | Interquartile Range | 1.43320 |

Note: The mode displayed is the smallest of 5 modes with a count of 2.

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| CENTANAFADINE | 38 OF 4 | 18 |
|---------------|---------|----|
|---------------|---------|----|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------ Analysis Visit (N)=35 ------

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Tests for Location: Mu0=0

| Test | -St | tatistic- | p Valı | 1e |
|-------------|-----|-----------|----------|--------|
| Student's t | t | -0.78956 | Pr > t | 0.4303 |
| Sign | M | 15.5 | Pr >= M | 0.1082 |
| Signed Rank | S | 313.5 | Pr >= S | 0.8683 |

#### Tests for Normality

| Test | Sta | tistic | p Va | alue |
|--------------------|------|----------|-----------|-----------|
| Shapiro-Wilk | W | 0.964473 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.092875 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.750058 | Pr > W-Sc | <0.0050 |
| Anderson-Darling | A-Sq | 4.316386 | Pr > A-Sc | q <0.0050 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| CENTANAFADINE | 39 OF 48 |
|------------------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

## The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Quantiles (Definition 5)

| Level | Quantile |
|------------|-----------|
| 100% Max | 2.240482 |
| 99% | 1.731891 |
| 95% | 1.229753 |
| 90% | 1.062172 |
| 75% Q3 | 0.718334 |
| 50% Median | 0.169236 |
| 25% Q1 | -0.714868 |
| 10% | -1.501925 |
| 5% | -1.944037 |
| 1% | -2.576562 |
| 0% Min | -3.200330 |

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100013/STAT/Program.dev/DOC STAT/normality.sas

OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-6.1.2

CENTANAFADINE 40 OF 48 PROTOCOL 405-201-00013

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------ Analysis Visit (N)=35 ------

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Extreme Observations

Highogt

| | Lowest- | | | | Hignest |
|----------|--------------|------|---------|-------------|---------|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -3.20033 | 40520100013- | 1852 | 1.72589 | 40520100013 | 1872 |
| -3.09371 | 40520100013- | 1833 | 1.73189 | 40520100013 | 1891 |
| -2.60303 | 40520100013- | 1694 | 1.74498 | 40520100013 | 1705 |
| -2.57656 | 40520100013- | 1731 | 1.79761 | 40520100013 | 1938 |
| -2.55159 | 40520100013- | 1857 | 2.24048 | 40520100013 | 1702 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 41 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

The UNIVARIATE Procedure
Variable: RESID (Residual)

#### Moments

| N | 347 | Sum Weights | 347 |
|-----------------|------------|------------------|------------|
| Mean | -0.3635827 | Sum Observations | -126.16319 |
| Std Deviation | 10.8189753 | Variance | 117.050226 |
| Skewness | -0.8029258 | Kurtosis | 0.15184193 |
| Uncorrected SS | 40545.2491 | Corrected SS | 40499.3783 |
| Coeff Variation | -2975.6575 | Std Error Mean | 0.58079302 |

## Basic Statistical Measures

Location Variability

| Mean | -0.36358 | Std Deviation | 10.81898 |
|--------|----------|---------------------|-----------|
| Median | 1.86002 | Variance | 117.05023 |
| Mode | 0.60473 | Range | 53.83629 |
| | | Interquartile Range | 14.88131 |

Note: The mode displayed is the smallest of 4 modes with a count of 2.

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| F 48 |
|------|
| )F |

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

Tests for Location: Mu0=0

| Test | -St | atistic- | p Va | lue |
|-------------|-----|----------|----------|--------|
| Student's t | t | -0.62601 | Pr > t | 0.5317 |
| Sign | M | 28.5 | Pr >= M | 0.0026 |
| Signed Rank | S | 1596 | Pr >= S | 0.3942 |

#### Tests for Normality

| Test | Sta | tistic | p Val | ue |
|--------------------|------|----------|-----------|---------|
| Shapiro-Wilk | W | 0.946801 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.099018 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 1.011224 | Pr > W-Sq | <0.0050 |
| Anderson-Darling | A-Sq | 5.883925 | Pr > A-Sq | <0.0050 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| CENTANAFADINE | 43 OF 48 |
|---------------|----------|
|---------------|----------|

PROTOCOL 405-201-00013 STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

Quantiles (Definition 5)

| Level | Quantile |
|------------|-----------|
| 100% Max | 19.94892 |
| 99% | 17.59826 |
| 95% | 13.42180 |
| 90% | 11.14587 |
| 75% Q3 | 7.91676 |
| 50% Median | 1.86002 |
| 25% Q1 | -6.96455 |
| 10% | -15.95262 |
| 5% | -21.57855 |
| 1% | -31.78702 |
| 0% Min | -33.88736 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 44 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------

------ Analysis Visit (N)=42 ------

The UNIVARIATE Procedure Variable: RESID (Residual)

Extreme Observations

Highogt

| | | | nighes | L | |
|----------|-------------|------|---------|--------------|------|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -33.8874 | 40520100013 | 2201 | 16.6970 | 40520100013- | 2053 |
| -33.3787 | 40520100013 | 2183 | 17.5983 | 40520100013- | 2144 |
| -33.1571 | 40520100013 | 2007 | 18.8332 | 40520100013- | 2278 |
| -31.7870 | 40520100013 | 2218 | 19.4803 | 40520100013- | 2284 |
| -28.1267 | 40520100013 | 2160 | 19.9489 | 40520100013- | 2153 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 45 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Moments

| N | 347 | Sum Weights | 347 |
|-----------------|------------|------------------|------------|
| Mean | -0.0353861 | Sum Observations | -12.278976 |
| Std Deviation | 1.02339086 | Variance | 1.04732886 |
| Skewness | -0.8014075 | Kurtosis | 0.14366209 |
| Uncorrected SS | 362.810289 | Corrected SS | 362.375784 |
| Coeff Variation | -2892.0705 | Std Error Mean | 0.0549385 |

Basic Statistical Measures

Location Variability

| Mean | -0.03539 | Std Deviation | 1.02339 |
|--------|----------|---------------------|---------|
| Median | 0.17390 | Variance | 1.04733 |
| Mode | 0.05664 | Range | 5.12952 |
| | | Interquartile Range | 1 41016 |

Note: The mode displayed is the smallest of 4 modes with a count of 2.

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| OF 48 |
|-------|
|-------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------ Analysis Visit (N)=42 ------

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Tests for Location: Mu0=0

| Test | -St | atistic- | p Valı | ıe |
|-------------|-----|----------|----------|--------|
| Student's t | t | -0.6441 | Pr > t | 0.5199 |
| Sign | M | 28.5 | Pr >= M | 0.0026 |
| Signed Rank | S | 1567 | Pr >= S | 0.4028 |

#### Tests for Normality

| Test | Sta | tistic | p Val | ue |
|--------------------|------|----------|-----------|---------|
| Shapiro-Wilk | W | 0.946825 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.099802 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 1.019493 | Pr > W-Sq | <0.0050 |
| Anderson-Darling | A-Sq | 5.928715 | Pr > A-Sq | <0.0050 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

| CENTANAFADINE | 47 OF 48 |
|---------------|----------|
|---------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_

## The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Quantiles (Definition 5)

| Level | Quantile |
|----------------------|-----------|
| 100% Max<br>99% | 1.902521 |
| 95% | 1.269575 |
| 90% | 1.049981 |
| 75% O3 | 0.749161 |
| 50% Median<br>25% O1 | 0.173896 |
| 10% | -1.496158 |
| 5% | -2.066916 |
| 1% | -2.976287 |
| 0% Min | -3.227003 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00

CENTANAFADINE 48 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------

------ Analysis Visit (N)=42 ------

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Extreme Observations

Highogt

| Lowest | | | Hignest | | |
|----------|-------------|------|---------|--------------|------|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -3.22700 | 40520100013 | 2201 | 1.65677 | 40520100013- | 2144 |
| -3.14078 | 40520100013 | 2183 | 1.67196 | 40520100013- | 2053 |
| -3.10521 | 40520100013 | 2007 | 1.76566 | 40520100013- | 2278 |
| -2.97629 | 40520100013 | 2218 | 1.82508 | 40520100013- | 2284 |
| -2.70089 | 40520100013 | 2160 | 1.90252 | 40520100013- | 2153 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 18JUN2020 10:00



# This page is a manifestation of an electronically captured signature

# SIGNATURE PAGE

Document Name: P40520100013\_DOC\_STAT

Document Number: 1000084975

**Document Version: 2.0** 

| Signed by | Meaning of Signature | Server Date<br>(dd-MMM-<br>yyyy hh:min) -<br>UTC timezone |
|---|---|---|
| | Safety Approval | 04-Aug-2020<br>14:03:59 |
| | Biostatistics Approval | 28-Jul-2020<br>15:44:56 |
| | Clinical Programming<br>Approval | 28-Jul-2020<br>14:13:56 |
| | Clinical Approval | 03-Aug-2020<br>18:34:55 |